## **PROTOCOL MG0002**

A MULTICENTER, RANDOMIZED, INVESTIGATOR- AND SUBJECT-BLIND, PLACEBO-CONTROLLED, TREATMENT SEQUENCE STUDY EVALUATING THE SAFETY, TOLERABILITY, AND EFFICACY OF UCB7665 IN SUBJECTS WITH MODERATE TO SEVERE MYASTHENIA GRAVIS

UCB Biopharma SPRL

Allée de la Recherche 60

1070 Brussels

BELGIUM

| Protocol/Amendment number | Date | Type of amendment |
|---------------------------|-------------|-------------------|
| Final Protocol | 21 Oct 2016 | Not applicable |
| Protocol Amendment 1 | 07 Feb 2017 | Substantial |
| Protocol Amendment 2 | 15 Sep 2017 | Substantial |

### **Confidential Material**

### **Confidential**

This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.


## STUDY CONTACT INFORMATION

## **Sponsor**

UCB Biopharma SPRL

Allée de la Recherche 60

1070 Brussels

**BELGIUM** 

## **Principal/Coordinating Investigator**

| Name: | Dr. Vera Bril | ans |
|---|---|---|
| Affiliation: | - | alaid |
| Address: | Toronto General Hospital<br>200 Elizabeth St.<br>Toronto, ON<br>Canada | on and any other |
| Phone: | | ot licatile |
| Fax: | | COX 350 |

## **Sponsor Study Physician**

| Name: | L'DA itholi |
|----------|---------------------------|
| Address: | UCB Biosciences, Inc. |
| | 8010 Arco Corporate Drive |
| | Raleigh, NC 27617 |
| | UNITED STATES |
| Phone: | |
| Fax: | - 1/1/80 |

# Clinical Project Manager

| Name: | |
|----------|----------------------------------|
| Address: | GCSO Clinical Project Management |
| call! | UCB Biosciences, Inc. |
| Ment | 8010 Arco Corporate Drive |
| clime | Raleigh, NC 27617 |
| | UNITED STATES |
| Phone: | |
| Fax: | - |


## **Clinical Trial Biostatistician**

| Name: | |
|----------|-------------------------|
| Address: | UCB BIOSCIENCES GmbH |
| | Alfred-Nobel-Strasse 10 |
| | 40789 Monheim |
| | GERMANY |
| Phone: | lali <sup>2</sup> |
| Fax: | COL |

# **Clinical Monitoring Contract Research Organization**

| | Name: | PAREXEL International (IRL) Limited |
|---|---|---|
| | Address: | 70 Sir John Rogerson's Quay Dublin 2 IRELAND |
| | Phone: | +353 1 473 9500 |
| | Fax: | +353 1 477 3390 |
| This d | ocument cannot be us | PAREXEL International (IRL) Limited 70 Sir John Rogerson's Quay Dublin 2 IRELAND +353 1 473 9500 +353 1 477 3390 AREA AND AN |


## **SERIOUS ADVERSE EVENT REPORTING**

| | Serious adverse event reporting (24h) |
|---|---|
| Fax | Europe and Rest of the World: +32 2 386 6561 |
| | <b>USA and Canada:</b> 011 32 2 386 65 61 |
| Email | Global: safetyreportingUCB7665@ucb.com |
| nis document canno | Europe and Rest of the World: +32 2 386 6561 USA and Canada: 011 32 2 386 65 61 Global: safetyreportingUCB7665@ucb.com Global: safetyreportingUCB7665@ucb.com |


# **TABLE OF CONTENTS**

| LIST OF | ABBREVIATIONS | 11 |
|---|---|---|
| 1 SUM | IMARY | 14 |
| 2 INTI | RODUCTION | 15 |
| 3 STU | DY OBJECTIVES | 18 |
| 3.1 Prim | ary objective | 18 |
| 3.2 Seco | ndary objectives | 18 |
| 3.3 Expl | oratory objectives | 18 |
| 4 STU | DY VARIABLES | 9 |
| 4.1 Effic | acy variables | 19 |
| 4.1.1 | Primary efficacy variable | 19 |
| 4.1.2 | Secondary efficacy variable | 19 |
| 4.1.3 | Other efficacy variables | 19 |
| 4.2 Othe | r and exploratory variables | 20 |
| 4.2.1 | Safety variables | 20 |
| 4.2.2 | Pharmacokinetic variable | 20 |
| 4.2.3 | Pharmacodynamic variables | 20 |
| 4.2.4 | Immunological variables | 21 |
| 5 STU | DY VARIABLES acy variables Primary efficacy variable Secondary efficacy variable Other efficacy variables r and exploratory variables Safety variables Pharmacokinetic variable Pharmacodynamic variables Immunological variables DY DESIGN y description Exploratory genomic analyses Study duration per subject | 21 |
| 5.1 Stud | y description | 21 |
| 5.1.1 | Exploratory genomic analyses | 23 |
| 5.1.2 | Study duration per subject | 23 |
| 5.1.3 | Planned number of subjects and sites | |
| 5.1.4 | Anticipated regions and countries | 23 |
| 5.2 Sche | dule of study assessments. | 24 |
| 5.3 Sche | matic diagram | 31 |
| | onale for study design and selection of dose | 31 |
| 5.4.1 | Choice of study design and endpoints | 31 |
| 5.4.2 | Rationale for dose selection | 32 |
| 5.4.3 | Justification for additional genomic analyses | 33 |
| 6 SEL | ECTION AND WITHDRAWAL OF SUBJECTS | 34 |
| 6.1 Inclu | sion criteria | 34 |
| 6.2 Excl | usion criteria | 35 |
| 6.2.1 | Exclusion criteria related to health status | 35 |
| 6.2.2 | Exclusion criteria related to concomitant medications/procedures | 37 |
| 6.2.3 | Exclusion criteria related to other risks | 38 |
| 6.3 Resc | reening and Rechecking | 38 |
| | drawal criteria | 39 |

| 6.4.1 Potential drug-induced liver injury IMP discontinuation criteria | 40 |
|---|---|
| 7 STUDY TREATMENT | 41 |
| 7.1 Description of investigational medicinal product | 41 |
| 7.2 Treatments to be administered | 41 |
| 7.3 Packaging | 42 |
| 7.4 Labeling | 42 |
| 7.5 Handling and storage requirements | 42 |
| 7.6 Drug accountability | -/ |
| 7.7 Procedures for monitoring subject compliance | |
| 7.8 Concomitant medication/treatment | |
| 7.8.1 Permitted concomitant medication 7.8.2 Prohibited concomitant treatments (medications and therapies) 7.8.3 Rescue medication | 43 |
| 7.8.2 Prohibited concomitant treatments (medications and therapies) | 44 |
| 7.8.3 Rescue medication 7.9 Blinding. | 44 |
| 7.9 Blinding. | 45 |
| 7.9.1 Procedures for maintaining and breaking the treatment blind | 45 |
| 7.9.1.1 Maintenance of study treatment blind | 45 |
| 7.9.1.2 Breaking the treatment blind in an emergency situation | 45 |
| 7.10 Randomization and numbering of subjects | 46 |
| 8 STUDY PROCEDURES BY VISIT | 46 |
| 8.1 Screening Period 8.1.1 Visit 1 (Day -28 to -1) Screening Visit 8.2 Dosing Period 1 8.2.1 Visit 2 (Day 1, Baseline) 8.2.2 Visit 3 (Day 2) 8.2.3 Visit 4 (Day 8) 8.2.4 Visit 5 (Day 9) | 46 |
| 8.1.1 Visit 1 (Day -28 to -1) Screening Visit | 46 |
| 8.2 Dosing Period 1 | 4/ |
| 8.2.1 Visit 2 (Day 1, Baseline) | 48 |
| 8.2.2 Visit 3 (Day 2) | 49 |
| 8.2.3 Visit 4 (Day 8) | 49 |
| | 31 |
| 8.2.5 Visit 6 (Day 15) | |
| 8.2.7 Visit 8 (Day 22) | |
| 8.3 Dosing Period 2 | |
| 8.3.1 Visit 9 (Day 29) | |
| 8.3.2 Visit 10 (Day 30) | |
| 8.3.3 Visit 11 (Day 36) | |
| 8.3.4 Visit 12 (Day 37) | |
| 8.3.5 Visit 13 (Day 43) | |
| 8.3.6 Visit 14 (Day 44) | |
| 8.4 Observation Period | |
| 9.4.1 Vigit 15 (Day 50) | 50 |

| 8.4.2 Visit 16 (Day 57) | 59 |
|---|---|
| 8.4.3 Visit 17 (Day 64) | 60 |
| 8.4.4 Visit 18 (Day 78) | 61 |
| 8.4.5 Visit 19 (Day 92) | |
| 8.4.6 Visit 20 (Day 99, Final Visit) and | Premature End of Treatment Visit |
| 8.5 Premature End of Treatment Visit | 64 |
| | 64 |
| 9 ASSESSMENT OF EFFICACY | |
| 9.1 Quantitative Myasthenia Gravis scale | |
| 9.2 MG-Composite scale | 65 |
| 9.3 Patient-reported outcomes | 65 ility 65 |
| 9.3.1 MG muscle weakness and fatigab | ility |
| 9.3.2 Fatigue | 66 |
| 9.3.3 MG-Activities of Daily Living | 66 dex 66 do 67 |
| 9.3.4 Myasthenia Gravis Impairment Ir | dex 66 |
| 9.4 MGFA classification | 66 |
| 9.5 Jitter (Single Fiber Electromyography) | $\sim$ 67 |
| 9.6 Subject exit interview | 67 |
| 10 ASSESSMENT OF PHARMACOKINE | |
| | GENOMIC VARIABLES67 |
| 10.1 Pharmacokinetic variable | 67 |
| 10.2 Pharmacodynamic variables | . 67 |
| | ES |
| | bles |
| | 69 |
| 12.1 Adverse events | 69 |
| 12.1.1 Definitions | 69 |
| 12.1.1.1 Adverse event | 69 |
| | 69 |
| 12.1.1.3 Adverse events of special i | nterest70 |
| 12.1.1.4 Adverse events of interest | 70 |
| | rerse events |
| 12.1.2 Procedures for reporting and reco | rding adverse events71 |
| Description of adverse ever | nts71 |
| 12.1.2.2 Rule for repetition of an ad | verse event71 |
| 12.1.2.3 Additional procedures for i | reporting serious adverse events71 |
| 12.1.3 Follow up of adverse events | 72 |
| 12.1.4 Pregnancy | 72 |

| 12.1.5 | Suspected transmission of an infectious agent via a medicinal product | 73 |
|---|---|---|
| 12.1.6 | Suicidality | 73 |
| 12.1.7 | Overdose of investigational medicinal product | 74 |
| 12.1.8 | Safety signal detection | 74 |
| 12.1.9 | Hypersensitivity and adverse reactions | 74 |
| 12.1.10 | Management of severe headache | 75 |
| 12.1.11 | Management of moderate or severe diarrhea. | 75 |
| 12.2 Labor | ratory measurements | 75 |
| 12.2.1 | Evaluation of PDILI | 37 |
| 12.2 | 1.1 Consultation with medical monitor and local hepatologist | |
| 12.2 | .1.2 Immediate action: determination of IMP discontinuation | ž81 |
| 12.2. | .1.3 Testing: identification/exclusion of alternative etiology | 82 |
| 12.2 | .1.4 Follow-up evaluation | 83 |
| 12.3 Other | safety measurements | 84 |
| 12.3.1 | Assessment and management of TB and TB risk factors | 84 |
| 12.3.2 | Pregnancy testing. | 85 |
| 12.3.3 | Vital signs | 86 |
| 12.3.4 | Body weight and height | 86 |
| 12.3.5 | Physical examination | 86 |
| 12.3 | 1.3 Testing: identification/exclusion of alternative etiology 1.4 Follow-up evaluation safety measurements Assessment and management of TB and TB risk factors Pregnancy testing Vital signs Body weight and height Physical examination 5.1 Full physical examination Neurological examination 12-lead ECG DY MANAGEMENT AND ADMINISTRATION | 86 |
| 12.3 | .5.2 Brief physical examination | 87 |
| 12.3.6 | Neurological examination | 87 |
| 12.3.7 | 12-lead ECG | 87 |
| 13 STUD | OY MANAGEMENT AND ADMINISTRATION | 88 |
| 13.1 Adher | rence to protocol | 88 |
| 13.2 Monit | rence to protocoltoring | 88 |
| 13.2.1 | Definition of source data | 88 |
| 13.2.2 | Source data verification | 89 |
| 13.3 Data l | handling | |
| 13.3.1 | Case Report Form completion | 89 |
| 13.3.2 | Database entry and reconciliation | 89 |
| | Subject Screening and Enrollment log/Subject Identification Code list | |
| L | ination of the study | |
| ~~ | ving and data retention | |
| 1 1 | and inspection | |
| | Clinical Practice | |
| | TISTICS | 91 |
| 14 1 Defini | ition of analysis sets | 91 |

| 14.2 Gener | ral statistical considerations | 92 |
|---|---|---|
| 14.3 Plann | ed efficacy analyses | 92 |
| 14.3.1 | Analysis of the primary efficacy variable | 92 |
| 14.3.2 | Other efficacy analyses | 93 |
| 14.4 Plann | ed other and exploratory analyses | 94 |
| 14.4.1 | Safety analyses | 94 |
| 14.4.2 | Pharmacokinetic analysis | 94 |
| 14.4.3 | Pharmacodynamic analysis | 95 |
| 14.4.4 | Immunalaciaal variables | 05 |
| 14.4.5 | Subject exit interview | 95 |
| 14.5 Hand | ling of protocol deviations | 95 |
| 14.6 Hand | ling of dropouts or missing data | 95 |
| 14.7 Plann | ed interim analysis and data monitoring | 96 |
| 14.8 Deter | mination of sample size | 96 |
| 15 ETHI | CS AND REGULATORY REQUIREMENTS | 97 |
| 15.1 Inform | ned consent | 97 |
| 15.2 Subje | ct identification cards | 97 |
| 15.3 Institu | Subject exit interview ling of protocol deviations ling of dropouts or missing data ed interim analysis and data monitoring mination of sample size CS AND REGULATORY REQUIREMENTS med consent ct identification cards ational Review Boards and Independent Ethics Committees | 97 |
| 15.4 Subje | ct privacycol amendments | 98 |
| 15.5 Protoc | col amendments | 98 |
| 16 FINA | NCE, INSURANCE, AND PUBLICATION | 99 |
| 17 REFE | RENCES | 99 |
| 18 APPE | ERENCES ENDICES | 101 |
| 18.1 Quant | titative Myasthenia Gravis Testing form | 101 |
| 18.2 MG-C | Composite score | 105 |
| 18.3 MG n | nuscle weakness PRO, Version 1 | 106 |
| | ue PRO, Version 1 | |
| | Activities of Daily Living | |
| | mpairment Index - Patient Questionnaire and Manual | |
| | A classification | |
| | ested management guidelines for infusion reactions | |
| | osis of anaphylactic reactions | |
| 18.10 | Headache Questionnaire | |
| | Tuberculosis Questionnaire | |
| 18.12 | Protocol Amendment 1 | |
| 18.13 | Protocol Amendment 2 | |
| | LARATION AND SIGNATURE OF INVESTIGATOR | |
| 20 SPON | ISOR DECLARATION | 193 |

## **LIST OF TABLES**

| Table 5.1: | Schedule of assessments | 25 |
|---|---|---|
| Table 6.1: | No-treatment periods for exclusionary immunosuppressants, biologics, and other therapies | 37 |
| Table 7.1: | Permitted concomitant treatments. | 43 |
| Table 12.2: | Safety laboratory measurements | 76 |
| Table 12.3: | Required investigations and follow up for PDILI. | 39 |
| Table 12.4: | PDILI laboratory measurements | <u></u> 82 |
| Table 12.5: | PDILI information to be collected | 83 |
| Table 18.1: | Suggested management guidelines for infusion reactions | 122 |
| Table 18.2: | Headache Questionnaire | 123 |
| | PDILI laboratory measurements PDILI information to be collected Suggested management guidelines for infusion reactions Headache Questionnaire LIST OF FIGURES Schematic diagram Quantitative Myasthenia Gravis Testing form | |
| Figure 5.1: | Schematic diagram | 31 |
| Figure 18.1: | | |
| Figure 18.2: | MG-Composite score | 105 |
| Figure 18.3: | | |
| Figure 18.4: | Fatigue PRO, Version 1 | 109 |
| Figure 18.5: | MG-Activities of Daily Living | 112 |
| Figure 18–6: | MG Impairment Index Patient Questionnaire | 113 |
| Figure 18–7: | MG Impairment Index – Examination Manual | 118 |
| Figure 18–8: | MG Impairment Index – Scoring Manual and Sheet | 119 |
| Figure 18.9: | MGFA classification | 121 |

. AGFA co

### LIST OF ABBREVIATIONS

ADL activities of daily living

AE adverse event

**ALP** alkaline phosphatase ALT alanine aminotransferase

analysis of covariance ANCOVA

**AST** aspartate aminotransferase

**BAFF** B-cell activating factor

BP blood pressure

tion application and any extensions of variations thereof. clinical data management system **CDMS** 

confidence interval CI

**CPM** Clinical Project Manager

Contract Research Organization **CRO** 

Columbia Suicide Severity Rating Scale C-SSRS

Common Terminology Criteria for Adverse Events **CTCAE** 

Data Cleaning Plan **DCP** 

**Data Monitoring Committee DMC** 

deoxyribonucleic acid **DNA ECG** electrocardiogram

electronic Case Report Form **eCRF** 

**Enrolled Set** ES

FAS Full Analysis Set

Fc crystalizable fragment

neonatal Fc receptor for IgG FcRnx

Final Visit

forced vital capacity Good Clinical Practice

GI gastrointestinal

**GMP** Good Manufacturing Practice HIV human immunodeficiency virus

application and any extensions of variations thereof. International Council for Harmonisation **ICH** 

**Independent Ethics Committee IEC** 

Ig immunoglobulin immunoglobulin A **IgA** IgE immunoglobulin E immunoglobulin G IgG

**IGRA** interferon-gamma release assay

immunoglobulin M **IgM** 

**IMP** investigational medicinal product

IPI interpotential interval

**IRB** Institutional Review Board

**IRT** interactive response technology

ITP immune thrombocytopenic purpura

iv

intravenous immunoglobulin IVIg LLOQ last observation carried forward LOCF

LS least squares

**LTBI** Latent tuberculosis infection mean consecutive difference **MCD** 

MG myasthenia gravis

myasthenia gravis-Activities of Daily Living **MGADL MGFA** Myasthenia Gravis Foundation of America

**MGII** Myasthenia Gravis Impairment Index

**MMRM** mixed model repeated measures

micro ribonucleic acid miRNA

mRNA messenger ribonucleic acid

**NMJ** neuromuscular junction NTMBI non-tuberculosis mycobacterium infection

PD pharmacodynamic(s)

an Jauthorization application and any extensions of variations thereof. **PDILI** potential drug-induced liver injury

**PEOT** premature end of treatment

PK pharmacokinetic(s) **PLEX** plasma exchange Per-Protocol Set **PPS** 

**PRO** patient-reported outcome

PS Patient Safety

QMG quantitative myasthenia gravis

corrected QT interval QTc

RNA ribonucleic acid RS Randomized Set

serious adverse event SAE

Statistical Analysis Plan SAP

subcutaneous sc

SD standard deviation

single fiber electromyography **SFEMG** Standard Operating Procedure **SOP** 

Safety Set SS tuberculosis TB

Treatment-emergent adverse event **TEAE** 

TNIP1 TNFAIP3-interacting protein 1

**TST** Tuberculin skin test This document cannot upper limit of normal United States of America

### 1 SUMMARY

The MG0002 study is a Phase 2a, multicenter, randomized, investigator- and subject-blind, placebo-controlled, 2-arm, repeat dose, treatment sequence study which will evaluate the efficacy, safety, and tolerability of chronic-intermittent treatment with UCB7665 in subjects with moderate to severe generalized myasthenia gravis (MG). UCB7665 will be administered as subcutaneous (sc) doses of 4mg/kg or 7mg/kg, in subjects ≥18 years of age.

The study is planned to be conducted at approximately 30 sites in United States of America (USA), Canada, and Europe, with possible extension to other regions and countries. A total of 42 subjects are planned to enter the Treatment Period in the study. The maximum study duration for an individual subject is approximately 18 weeks.

The study will consist of 3 Periods: Screening, Treatment, and Observation. After Screening, subjects will enter the Treatment Period, which will consist of Dosing Period 1 followed by Dosing Period 2. Subjects will receive 3 doses of investigational medicinal product (IMP) at weekly intervals during each dosing period as follows:

- Dosing Period 1 will be 4 weeks, with 2 parallel arms (UCB7665 7mg/kg or placebo).
- Dosing Period 2 will be 2 weeks, with 2 parallel treatment arms (UCB7665 7mg/kg or UCB7665 4mg/kg).

The Observation Period will span 8 weeks after the final dose of UCB7665, with a Final Visit (FV) being scheduled at Visit 20. The sc infusions will last approximately 30 minutes, and subjects will be required to remain in the hospital/clinic at least 4 hours for safety monitoring after each infusion.

A Data Monitoring Committee (DMC) will be implemented as described in Section 14.7.

The primary efficacy variable will be the change from Baseline in Quantitative MG (QMG) score to Visit 9 (Day 29). The secondary efficacy variables will be the change from Baseline in MG-Composite score to Visit 9 (Day 29) and the change from Baseline in MG-Activities of Daily Living (MGADL) score to Visit 9 (Day 29). Other efficacy variables will be the following: value and change from Baseline in QMG at each scheduled assessment during Treatment and Observation Periods; QMG responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MG-Composite score at each scheduled assessment during Treatment and Observation Periods; MG-Composite responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MGADL at each scheduled assessment during Treatment and Observation Periods; MGADL responder (>3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods: Myasthenia Gravis Foundation of America (MGFA) classification at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MG muscle weakness severity, fatigue scales and Myasthenia Gravis Impairment Index (MGII) scores at each scheduled assessment during Treatment and Observation Periods; and change in mean consecutive difference (MCD) in jitter (single fiber electromyography [SFEMG]) studies from Baseline to Visit 9 for the subjects consenting to this measurement at participating sites.

15 Sep 2017 UCB7665 MG0002

Other and exploratory variables include: safety and tolerability variables, pharmacokinetic (PK), pharmacodynamic (PD), and immunologic variables.

Safety and tolerability variables include the following: occurrence of treatment-emergent adverse in subjects experiencing severe headache and/or moderate to severe gastrointestinal furbance; and TEAEs leading to withdrawal of IMP.

concentration of UCB7665 over time will be assessed as the DTZ will be the maximum decrease from Baseline in ation; value and change for a lassesser. events (TEAEs); vital sign values and changes from Baseline (systolic and diastolic blood pressure [BP], temperature, pulse rate, respiratory rate, and body weight); 12-lead electrocardiogram (ECG) values and change from Baseline; laboratory values (hematology, clinical chemistry, and urinalysis) and changes from Baseline; change from Baseline in exploratory safety biomarkers (may include but not limited to

(GI) disturbance; and TEAEs leading to withdrawal of IMP.

Plasma concentration of UCB7665 over time will be assessed as the PK variable. The main PD variables will be the maximum decrease from Baseline in serum total immunoglobulin G (IgG) concentration; value and change from Baseline in total serum IgG concentrations at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in serum IgG subclass concentrations at each scheduled assessment during Treatment and Observation Periods; and change in MG-specific autoantibody levels in serum from Baseline at each scheduled assessment during Treatment and Observation Periods. Additionally, change from Baseline in other immunological variables and other exploratory biomarkers during the Treatment and Observational Periods will be assessed.

During this study, subjects will also have the option of providing additional informed consent for exploratory deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) (ie, messenger RNA [mRNA] and micro RNA [miRNA]) analyses (see Section 5.1.1) to understand the cause, progression, and appropriate treatment of MG. Participation in this additional portion of the study is optional and does not preclude subject's eligibility for participation in the main study. The additional genomic samples must not be collected if the subject has not consented to participate in this exploratory genomic substudy.

### INTRODUCTION 2

UCB7665 is a humanized anti-neonatal Fc receptor for IgG (FcRn) monoclonal antibody that has been specifically designed to inhibit IgG binding to FcRn without inhibiting albumin binding to FcRn. UCB7665 is being developed as an inhibitor of FcRn activity with the aim to reduce the concentration of pathogenic IgG in patients with IgG autoantibody mediated diseases.

The neonatal Major histocompatibility complex-class FcRn recycles IgG and albumin from most cells and transports it bi-directionally across epithelial barriers to affect systemic and mucosal immunity. It was shown that FcRn rescues both IgG and albumin from intracellular lysosomal degradation by recycling it from the sorting endosome to the cell surface (Anderson et al, 2006). With respect to IgG, this is achieved by interaction of IgG with the receptor, FcRn. Thus in effect FcRn salvages IgG, and blockade of FcRn accelerates removal of endogenous IgG.

As individual disease entities, IgG autoantibody mediated conditions are relatively rare. Treatment of these disorders remains a difficult clinical problem, requiring in many of these conditions the long-term use of high-dose corticosteroids alone or combined with cytotoxic agents. These therapeutic approaches are not effective in all patients and conditions and have broad immunosuppressive effects causing considerable toxicity and treatment-related morbidity.


UCB 15 Sep 2017 Clinical Study Protocol UCB7665 MG0002

Treatments aimed at reducing the quantity of circulating IgG autoantibody, including plasmapheresis, immunoadsorption, or high-dose intravenous immunoglobulin (IVIg), are being used for primary and secondary therapy of autoimmune disease, particularly where corticosteroid-based immune suppression is not or no longer effective (eg, immune thrombocytopenic purpura [ITP], MG, and chronic inflammatory demyelinating polyradiculoneuropathy). The therapeutic approach of these treatments is thought to be based on lowering levels of pathogenic autoantibodies, which represents rational and effective treatment modalities of autoimmune diseases.

Myasthenia gravis is a rare autoimmune disorder of the peripheral motor system in which autoimmune antibodies most commonly form at the neuromuscular junction (NMJ). The autoantibody impairs the ability of to bind to receptors, and leads to the destruction of receptors, either by inducing the muscle cell to eliminate the receptors through endocytosis or by complement fixation. A second category of MG is due to autoantibodies against the which is required for the formation of the NMJ. Antibodies inhibit signaling, resulting in a decrease in patency of the NMI, and the consequent symptoms of MG. In both categories, this results in a characteristic pattern of progressively reduced muscle strength with repeated muscle use and muscle strength recovery following a period of rest. Additional antibodies have been found to be associated with MG but less is yet known about them and they appear less common than the main two. The essential role of the autoimmune antibodies in mediating this pathology is supported by the improvement seen after plasma exchange (PLEX). Plasma Exchange which reduces IgG levels including pathogenic IgG autoantibody is used both in patients non-responsive to inhibitors or immunosuppressive treatments and in patients experiencing myasthenic crisis (Gilhus and Verschuuren, 2015).

Although the prognosis of MG has markedly improved over the last decades, with new therapies dramatically improving survival, significant mortality and even morbidity remains an issue. Treatment of MG remains a difficult clinical problem, requiring the long-term use of high-dose corticosteroids alone or combined with cytotoxic agents. Many of the therapies thought to be effective in MG have insufficient data to clearly support their use, are not effective in all patients and conditions, and have broad immunosuppressive effects causing considerable toxicity and treatment-related morbidity. Moreover, due to the natural fluctuations in the course of the disease, many patients need an effective treatment for acute situations requiring urgent treatment. Both PLEX and IVIg currently are used as the standard of care to improve symptoms in situations requiring chronic-intermittent treatment; however, neither treatment is approved in the US for MG, and the procedures often are burdensome for the patients. Thus a significant unmet medical need exists in this patient population for an effective chronic-intermittent treatment with increased convenience for patients with generalized MG.

UCB 7665 is being developed as an inhibitor of FcRn activity with the aim to reduce the concentration of pathogenic IgG in patients with IgG autoantibody mediated diseases. UCB7665 was derived from a rat antibody with specificity for human FcRn.

Both preclinical studies in nonhuman primates and clinical studies suggest that treatment with UCB7665 may reduce the concentration of pathogenic IgG. The relationship between UCB7665 exposure and the primary PD effect on plasma IgG levels was studied in Cynomolgus monkeys

following single- and repeat dose administrations by both intravenous (iv) and sc routes. UCB7665 mediated a clear dose- and exposure-related decrease in plasma IgG concentrations, achieving 45% to ≥70% decreased IgG concentrations at dose levels ranging from 5 to 30mg/kg in the absence of adverse effects. No consistent or dose-related effects of UCB7665 on albumin levels were observed in these studies.

To date, UCB7665 has been administered to human subjects in 2 clinical studies, UP0018 and TP0001. UP0018 is a completed first-in-human study in 49 healthy subjects. The study evaluated the safety, tolerability, PK, and the PD effect on total IgG levels of single ascending doses of iv and sc administered UCB7665. Doses of UCB7665 1, 4, and 7mg/kg were administered by both iv and sc routes in 3 cohorts, respectively, as an 1 hour infusion. The information from the study is summarized below.

Dose-dependent statistically significant reductions in levels of serum total IgG and dose-dependent reductions in levels of IgG subclasses (IgG 1 to 4) were observed after UCB7665 was administered by iv or sc routes. There were no deaths or serious adverse events (SAEs) reported during the study, and no subjects discontinued the study due to TEAEs. UCB7665 was tolerated with an acceptable safety profile after the single administration of up to 4mg/kg iv and up to 7mg/kg sc doses. For iv administration of UCB7665, the most frequently reported TEAEs were headache (10 subjects [55.6%]) and nasopharyngitis, nausea, pyrexia, and vomiting (each reported by 7 subjects [38.9%]). Four TEAEs with a maximum intensity of severe were reported in this study: headache (3 subjects [50.0%]) and back pain (1 subject [16.7%]); all of which were reported in the UCB7665 7mg/kg iv group. For sc administration of UCB7665, the most frequently reported TEAEs were headache (5 subjects [27.8%]) and back pain and diarrhea (each reported by 3 subjects [16.7%]). Importantly, there were fewer incidences of headaches and GI disturbances following sc administration of UCB7665 compared with iv administration. The safety profile of the sc route of administration, up to 7mg/kg of UCB7665, was considered to be manageable, and all subject reported TEAEs had a maximum intensity of mild or moderate. The peak and total exposure of UCB7665 showed nonlinear increases consistent with target-mediated disposition. Based on the preliminary results, a minimal level of immunogenicity and minimal effects on antibodies were observed.

An ongoing study, TP0001, is a multicenter, open-label, single- and multiple-dose, multiple-arm Phase 2a study to evaluate the safety, tolerability, and efficacy of UCB7665 administered as sc doses in adult subjects with primary ITP. This ongoing study is the first study to evaluate multiple doses of UCB7665 and will evaluate multiple Treatment Groups of UCB7665. The dose arms are as follows:

- Dose Arm 1 (15 subjects): UCB7665 4mg/kg sc (5 doses at an interval of 1 week)
- Dose Arm 2 (15 subjects): UCB7665 7mg/kg sc (3 doses at an interval of 1 week)
- Dose Arm 3 (6 to 12 subjects): UCB7665 10mg/kg sc (2 doses at an interval of 1 week)
  - Dose Arm 4 (6 to 12 subjects): UCB7665 15mg/kg sc (1 dose)
- Dose Arm 5 (6 to 12 subjects): UCB7665 20mg/kg sc (1 dose)

To date, 15 subjects in Dose Arm 1 (5x4mg/kg) and 13 subjects in Dose Arm 2 (3x7mg/kg) have safely completed his/her treatment period.

MG0002 will be the first study of the use of UCB7665 in MG. The aim of the study is to evaluate the efficacy, safety, and immunological effect of UCB7665, and to gather data for future study planning to fully evaluate the use of UCB7665 in MG.

For more detailed information, refer to the current version of the UCB7665 Investigator's Brochure.

### 3 STUDY OBJECTIVES

### 3.1 Primary objective

The primary objective of the study is:

• To evaluate the clinical efficacy of UCB7665 as an chronic-intermittent treatment in subjects with generalized MG who are classified as moderate to severe

### 3.2 Secondary objectives

The secondary objectives of the study are:

- To gather data for future study planning, whether for chronic-intermittent treatment or a longer therapy option by evaluating the general concept that UCB7665 has a clinical effect in patients with generalized MG
- To evaluate the safety and tolerability of UCB7665 administered by sc infusion in subjects with MG
- To assess the effect of UCB7665 as measured by total IgG concentrations in serum

## 3.3 Exploratory objectives

The exploratory objectives are:

| • | To assess the effect of UCB7665 on MG-specific autoantibodies ( |
|---|-----------------------------------------------------------------|
| | levels in serum |

- To evaluate the effects of UCB7665 on the concentration of IgG subclasses, immunoglobulin M (IgM), immunoglobulin A (IgA), and immunoglobulin E (IgE), and serum and plasma complement levels
- To evaluate the effect of UCB7665 on B-cell activating factor (BAFF) and on cytokines (in all subjects)
- To evaluate the effect of UCB7665 on cytokines in subjects experiencing infusion reactions
- To evaluate the emergence of PK/PD with respect to immunogenicity and
- To evaluate the effect of UCB7665 on clinical electrophysiological parameters of neuromuscular transmission in a subset of subjects
- To assess the plasma concentrations of UCB7665 administered by sc infusion
- To evaluate the effects of UCB7665 on blood biomarkers for safety (including, but not limited to

only in subjects with severe headache and/or moderate to severe GI disturbance

The effects of UCB7665 on

antibodies

- To evaluate peripheral blood biomarkers in relation to disease etiology, progression and treatment outcome
- ication and any extensions of variations thereof. To evaluate the genomic components of MG to understand the molecular etiology, progression, and treatment of the disease, applicable only for subjects consenting to participate in the optional genomic analyses substudy

#### 4 STUDY VARIABLES

#### 4.1 **Efficacy variables**

#### 4.1.1 Primary efficacy variable

The primary efficacy variable is:

Change from Baseline in QMG score to Visit 9 (Day 29)

#### 4.1.2 Secondary efficacy variable

The secondary efficacy variables are:

- Change from Baseline in MG-Composite score to Visit 9 (Day 29)
- Change from Baseline in MGADL score to Visit 9 (Day 29)

### Other efficacy variables 4.1.3

The other efficacy variables are:

- Value and change from Baseline in QMG at each scheduled assessment during Treatment and Observation Periods
- QMG responder ( $\geq$ 3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
- Value and change from Baseline in MG-Composite score at each scheduled assessment during Treatment and Observation Periods
- MG-Composite responder (>3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
- Value and change from Baseline in MGADL at each scheduled assessment during Treatment and Observation Periods
- MGADL responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
- MGFA classification at each scheduled assessment during Treatment and Observation Periods
- Value and change from Baseline in MG muscle weakness and fatigability at each scheduled assessment during Treatment and Observation Periods

- Value and change from Baseline in fatigue at each scheduled assessment during Treatment and Observation Periods
- Value and change from Baseline in MGII scores at each scheduled assessment during Treatment and Observation Periods
- Change in the percentage of normal fiber pairs in jitter (SFEMG) studies from Baseline to Visit 9 for the subjects consenting to this measurement at the participating sites
- Change in MCD of the interpotential interval (IPI) in jitter (SFEMG) studies from Baseline to Visit 9 for the subjects consenting to this measurement at the participating sites
- A reduction in MCD of ≥9µs in jitter (SFEMG) studies will define clinical improvement

### 4.2 Other and exploratory variables

### 4.2.1 Safety variables

The safety variables are the following:

- Occurrence of TEAEs
- Vital sign values and changes from Baseline (systolic and diastolic BP, temperature, pulse rate, respiratory rate, and body weight) at each scheduled assessment during Treatment and Observation Periods
- 12-lead ECG values and change from Baseline at each scheduled assessment during Treatment and Observation Periods
- Laboratory values and changes from Baseline at each scheduled assessment during Treatment and Observation Periods (hematology, clinical chemistry, and urinalysis)
- Change from Baseline in exploratory safety biomarkers (may include but not limited to

in subjects with severe headache and/or moderate to severe GI disturbance

TEAEs leading to withdrawal of IMP

The clinical safety laboratory tests are detailed in Table 12.2.

### 4.2.2 Pharmacokinetic variable

The PK variable is the following:

 Plasma concentration of UCB7665 at each scheduled assessment during Treatment and Observation Periods

### 4.2.3 Pharmacodynamic variables

The PD variables are the following:

- Minimum value and maximum (absolute and percentage) decrease from Baseline in serum total IgG concentration during the study
- Value and change (absolute and percentage) from Baseline in total serum IgG concentrations at each scheduled assessment during Treatment and Observation Periods

- Value and change (absolute and percentage) from Baseline in serum IgG subclass concentrations at each scheduled assessment during Treatment and Observation Periods
- Change in MG-specific autoantibody levels in serum from Baseline valiations thereof at each scheduled assessment during Treatment and Observation Periods

#### 4.2.4 Immunological variables

The other immunological variables are the following:

- Change from Baseline in serum immunoglobulin (Ig) concentrations (total IgA, IgE, and IgM) at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in serum complement levels (C3 and C4) and plasma complement levels (C3a and C5a) predose at Visit 2 and 4 hours postdose at each scheduled assessment during Treatment and Observation Periods
- status (negative or confirmed positive) and either change from Baseline in relative mass units at each scheduled assessment during Treatment and Observation Periods or titre for those confirmed positive.
- Change from Baseline in serum BAFF levels
- Change from Baseline in cytokines predose and postdose (postdose in subjects experiencing infusion reactions) at assessments during Treatment and Observation Periods
- antibodies Change from Baseline in
- Change from Baseline in exploratory biomarkers relating to mechanism of action, disease activity, treatment response, and clinical outcome

#### STUDY DESIGN 5

#### Study description 5.1

This is a Phase 2a, multicenter, randomized, investigator- and subject-blind, placebo-controlled, 2-arm, repeat dose, treatment sequence study evaluating the safety and efficacy of UCB7665 as an chronic-intermittent treatment for subjects with moderate to severe generalized MG.

Approximately 42 randomized subjects will be enrolled at approximately 30 sites from USA, Canada, and Europe to achieve the targeted number of 40 evaluable subjects.

The maximum duration of the study per subject is approximately 18 weeks, consisting of a Screening Period (1 to 28 days), Treatment Period (6 weeks), and an Observation Period (8 Weeks).

**Screening Period:** The purpose of the Screening Period is to evaluate and confirm the subject's eligibility. During the Screening Visit (Visit 1), subjects will sign a written Informed Consent form prior to the conduct of any study-related procedures. The use of concomitant medication while in the study will be discussed and subjects' eligibility will be determined on the basis of the inclusion/exclusion criteria. The Screening Period should not exceed 28 days in total.

**Treatment Period:** The Treatment Period will consist of Dosing Period 1 followed by Dosing Period 2. Subjects will receive 3 doses of IMP at weekly intervals during each dosing period as follows

- Dosing Period 1 will be 4 weeks, with 2 parallel Treatment Groups (UCB7665 7mg/kg or placebo).
- Dosing Period 2 will be 2 weeks, with 2 parallel Treatment Groups (UCB7665 7mg/kg or UCB7665 4mg/kg).

Prior to receiving an infusion with IMP, subjects will be assessed for efficacy measurements at each visit in the Treatment Period. For all safety and efficacy measurements, the order specified in the Study Procedures Manual is recommended to be used as a guide.

Valiations thereof Dosing Period 1: Dosing Period 1 will last for approximately 4 weeks (Day 1 to Day 28) and includes Visits 2, 3, 4, 5, 6, 7, and 8. Following completion of the Screening Period, eligible subjects will check-in at the clinic/hospital for the Randomization Visit (Visit 2). Subjects who continue to meet eligibility requirements will be randomized 1:1 to receive 7mg/kg of UCB7665 or placebo, administered by an approximately 30 minute sc infusion at weekly intervals for 3 weeks (Visits 2, 4, and 6) followed by an assessment visit at Week 4 (Visit 8). At Visits 2, 4, and 6 in Dosing Period 1, subjects will be required to remain in the clinic/hospital for at least 4 hours for safety monitoring after the infusion. Subjects may leave the clinic/hospital once the safety monitoring postdose period is over and the investigator or designee has no safety concerns. A follow-up telephone call will be conducted 24 hours postdose to assess the status of the subject (Visits 3, 5, and 7). Subjects will return to the clinic/hospital at Visit 8 for safety and efficacy assessments (see Section 5.2, Schedule of Study Assessments). The primary efficacy endpoint, change from Baseline in the QMG score, will be assessed at the beginning of Dosing Period 2 at Visit 9 (Day 29) prior to rerandomization. The efficacy assessments that are performed at Visit 9 will therefore occur 2 weeks after the final dose of study drug in Dosing Period 1.

Dosing Period 2: Dosing Period 2 will last for approximately 2 weeks (Day 29 to Day 43) and includes Visit 9, 10, 11, 12, 13, and 14. Subjects will return to the clinic for Visit 9, 11, and 13 for safety and efficacy assessments (see Section 5.2, Schedule of Assessments) in the order specified in Section 8. At Visit 9, following the administration of safety and efficacy assessments, subjects initially randomized at Baseline to placebo or to 7mg/kg of UCB7665 will be rerandomized 1:1 to receive either 3 doses of 7mg/kg or 3 doses of 4mg/kg administered by a 30 minute sc infusion at weekly intervals (Visit 9, 11, and 13). The interactive response technology (IRT) will stratify the rerandomization based on the treatment received in Dosing Period 1 (see Section 7.10 for further details regarding randomization). At each weekly clinic visit in Dosing Period 2 (Visits 9, 11, and 13), subjects will be required to remain in the clinic/hospital for at least 4 hours safety monitoring postdose period as determined. Subjects may leave the clinic/hospital once the safety monitoring postdose period is over and the investigator or designee has no safety concerns. A follow-up telephone call will be conducted 24 hours postdose to assess the status of the subject (Visits 10, 12, and 14).

**Observation Period:** All subjects must be followed for 8 weeks after the final dose of IMP is administered. Subjects will return to the clinic for Visits 15, 16, 18, and 20 for efficacy and for safety assessments (see Section 5.2, Schedule of Assessments). Subjects will either return to the clinic/hospital, or, if possible and agreed by both investigator and subject, have home visits conducted by certified healthcare professionals, for Visits 17 and 19. The Observation Period begins the day after the final dose of IMP (ie, Visit 13, Day 43); Visit 15 (Day 50) is the first visit in the Observation Period.

#### 5.1.1 **Exploratory genomic analyses**

During this study, subjects will also have the option of providing additional informed consent for exploratory genomic (DNA and RNA) analyses. Participation in this additional portion of the For RNA: Blood samples will be collected at Baseline (Visit 2), at Visit 8, and prior to the last dose of IMP (Visit 13).

For each DNA blood

For each DNA blood study is optional and does not preclude subject's eligibility for participation in the main study.

a volume of 2.5mL whole blood is needed.

Any exploratory biomarker or genomic analysis will only ever be related to the exploration of the underlying causes of MG in patients, related biology, and drug response. Justification for additional genomic analyses is detailed in Section 5.4.3.

Details on the collection, storage, preparation, and shipping of samples will be presented in the Laboratory Manual provided separately.

Any results from this analysis will be reported separately and will not form a part of the main clinical study report.

#### Study duration per subject 5.1.2

The maximum duration of the study per subject will be approximately 18 weeks, consisting of the following 3 periods:

Screening Period: 1 to 28 days

Treatment Period: 6 weeks

Observation Period: 8 weeks

The end of the study is defined as the date of the final clinic/hospital or home visit of the final subject in the study.

#### 5.1.3 Planned number of subjects and sites

To ensure that at least 40 subjects are evaluable for the primary efficacy variables, a sample size of approximately 42 randomized subjects is planned at approximately 30 sites to achieve the targeted number of 40 evaluable subjects.

#### 5.1.4 **Anticipated regions and countries**

It is planned to recruit subjects in USA, Canada, and Europe in this study, with possible extension to other regions and countries.

15 Sep 2017 MG0002

RELEASE TO THE BELLIAR TO THE LEASE OF THE BEAUTY OF THE BEAUTY.


Table 5.1: Schedule of assessments

| Assessments | Screen | ning | Trea | atment I | Period | l | | | | | | | | | | Obs | serva | tion I | Perio | d <sup>a</sup> | <del>)</del> | UV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ing Peri | od 1 | | | | | Dos | ing Pe | riod 2 | | | | | | | O | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | P | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> | 9 | 15 <sup>d</sup> | 16 | 22 <sup>d</sup> | 29 <sup>d</sup> | 30 | 36 <sup>d</sup> | 37 | 43 <sup>d</sup> | 44 | 50 | 57 | 64 | 78 | 92 | 99 | |
| | | | | | (± 2<br>days) | | (± 2<br>days) | ı | (± 2 days) | (± 2<br>days) | | (± 2<br>days) | | (± 2 days) | 79.8 | | (± 2 | days) | | | (± 2 days) | |
| Written informed | consent | X | | | | | | | | | | | | ion | 0 | | | | | | | |
| Written informed for genomic subst | | X | | | | | | | | c. | RY | á | 20lice | | | | | | | | | |
| Demographic data | ı | X | | | | | | | | | •.( | 20 | | | | | | | | | | |
| Verification of inc/exclusion criteria | | X | X | | | | | | OPC/V | | 1120 | | | | | | | | | | | |
| Call or enter IRT register the visit | to | X | | | X | | X | 4 | | Jill | | X | | X | | | | | | | X | |
| Call or enter IRT/<br>Randomization | r | | X | | | | | | Kejins | X | | | | | | | | | | | | |
| Withdrawal criter | ia | | X | X | X | X | X | Xζ | X | X | X | X | X | X | X | X | X | X | X | X | | |
| General medical/<br>procedures history | y | X | | | | | z os | 3 | | | | | | | | | | | | | | |
| Prior and concom<br>medication | itant | X | X | X | X | 7:56<br>X6 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant med procedures | ical | | X | | Ø | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Vital signs <sup>f</sup> | | X | X | 272 | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Body weight, heig | ght <sup>g</sup> | X | O'L'C | | | | | | | X | | | | | | | | | | | X | |
| Recording of AEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Table 5.1: Schedule of assessments

| | Protocol | | | | | | | | | | | | | | | | | | | | | MG000 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | Sche | edule of | ass | essm | ents | <b>S</b> | | | | | | | | | | | | | | , | ionsiti | |
| Assessments | Screen | ning | Treatment Period | | | | | | | | | | | | Obs | UV | | | | | | |
| | | | Dosi | ing Peri | od 1 | | | | | Dos | ing Per | riod 2 | | | | o's | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | <b>14</b> <sup>b</sup> | 15 | 16 | B | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> (± 2 days) | 9 | 15 <sup>d</sup><br>(± 2<br>days) | 16 | | 29 <sup>d</sup><br>(± 2<br>days) | 30 | 36 <sup>d</sup><br>(± 2<br>days) | | 43 <sup>d</sup><br>(± 2<br>days) | 44 | 560 | 57<br>(± 2 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| Full physical examination | | X | | | | | | | | | | | × | 1017 | 9 | | | | | | X | |
| Brief physical examination | | | X | | | | | | | X | RT | ~ | 3Plico | | | | | | | | | |
| Full neurological examination h | | X | | | | | | | 4 | | ii | 20,0 | | | | | | | | | X | |
| Brief neurologica examination | ıl | | X | | | | | < | DRC, | X | Sille | | | | | | | | | | | |
| Query for suicida | ılity <sup>i</sup> | X | X | | X | | X | 4 | X | X | | X | | X | | X | X | X | X | X | X | X |
| 12-lead ECG <sup>j</sup> | | X | X | | X | | X | | Xeims | X | | X | | X | | X | | | X | | X | |
| Laboratory tests (hematology, che urinalysis) | mistry, | X | X | | X | | X | 74 | òΧ | X | | X | | X | | X | X | | X | | X | |
| Serology testing the Hepatitis B, and I | for HIV,<br>Hepatitis | X | | | | 7166 <sub>0</sub> | 35.0 | | | | | | | | | | | | | | | |
| IGRA tuberculos | is test <sup>k</sup> | X | | | 10 | | | | | | | | | | | | | | | | | |
| Tuberculosis Sign<br>Symptoms questi | | X | | USE | ) | | | | | | | | | | | | | | | | X | |
| Blood sampling f<br>of UCB7665 <sup>l</sup> | or PK | | X/C | | X | | X | | X | X | | X | | X | | X | | | | | | |

Table 5.1: Schedule of assessments

| UCB<br>Clinical Study P | rotocol | | | | | | | | UCF | 3766 | 5 | | | | | | | | | | "VOLG | Sep 201<br>MG000 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | Sche | dule of | ass | essm | ents | 8 | | | | | | | | | | | | | | | ijons | |
| Assessments | Screen | ing | Trea | tment I | Period | ı | | | | | | | | | | Obs | Observation Period <sup>a</sup> | | | | | |
| | | | Dosi | ing Perio | od 1 | | | | | Dos | ing Per | riod 2 | | | | | | | , oʻ | | | |
| | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 150 | 18 | 19 | 20<br>FV/PEOT | | |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup> (± 2 | 9 | 15 <sup>d</sup> (± 2 | 16 | 22 <sup>d</sup><br>(± 2 days) | | | 36 <sup>d</sup> (± 2 | 37 | 43 <sup>d</sup><br>(± 2 | 44 | 500 | 57 | 64 | 78 | 92 | 99<br>(± 2 days) | |
| Blood sampling fo | | | X | | days) | | days) | | X | days) | | days) | ×. | days) | 200 | | (± 2 | uays) | | | | |
| Blood sampling fo<br>analysis sub-study | | | X | | X | | | | X | | RT | ~ | Splice | X | | | | | | | X | |
| Serum pregnancy | test | X | | | | | | | | ) | 3.0 | 50 | | | | | | | | | | |
| Urine pregnancy t | est <sup>n</sup> | | X | | X | | X | | X | X | :130 | X | | X | | X | X | X | X | X | X | |
| Administration of | IMP | | X | | X | | X | < | Ö | X | ), | X | | X | | | | | | | | |
| | | | X | | X | | X | √ | X | X | | X | | X | | X | X | X | X | X | X | |
| Serum complement<br>(C3,C4) and plasm<br>complement level<br>and C5a) <sup>o</sup> | na | | X | | X | | X | 40 | aixec | X | | X | | X | | | | | | | X | |
| Immunoglobulins<br>IgG and IgG subc | | X | X | | X | .08 | X | | X | X | | X | | X | | X | X | X | X | X | X | |
| IgA, IgM, IgE | | | X | | Ç. | 7.7 | | | X | X | | X | | X | | X | X | | | | X | |
| MG-specific autoantibodies | | | X | sed | X | | | | | X | | X | | | | X | | | | | X | |

Table 5.1: Schedule of assessments

| UCB<br>Clinical Study Pr | rotocol | | | | | | | | UCE | 3766 | 5 | | | | | | | | | | "Veig | Sep 201'<br>MG0002 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | Sche | edule of | ass | essm | ents | 6 | | | | | | | | | | | | | | | ijon <sup>s</sup> iti | |
| Assessments | Screen | ing | Treatment Period | | | | | | | | | | | | | | Observation Period <sup>a</sup> | | | | | |
| | | | Dosi | ing Peri | od 1 | | | | | Dos | ing Per | riod 2 | | | | | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | 5 <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 100 | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup> | 9 | 15 <sup>d</sup> | 16 | 22 <sup>d</sup> | 29 <sup>d</sup> | 30 | 36 <sup>d</sup> | 37 | 43 <sup>d</sup> | 44 | 50 | 57 | 64 | 78 | 92 | 99 | |
| | | | | | (± 2<br>days) | | (± 2<br>days) | | (± 2 days) | (± 2<br>days) | | (± 2<br>days) | | (± 2<br>days) | 90 | | (± 2 | days) | | | (± 2 days) | |
| Blood sampling fo<br>exploratory bioma<br>analysis | | | X | | X | | X | | Х | X | | Х | . ~ ? | X | <i>5</i> * | | | X | | X | | |
| Blood sampling for<br>safety biomarker<br>analysis: may include but<br>not limited to | | | X | | Х | | Х | 2 | X | XC | sila <sup>il</sup> | X | | X | | X | х | Х | X | Х | Х | |
| BAFF analysis | | | X | | X | | X | | X | X | | X | | X | | | | X | | X | | |
| Cytokines <sup>q</sup> | | | X | | | | X | | di | X | | | | X | | | | | | | X | X |
| Vaccination-special antibody titers | fic | X | | | | | K of | 4 | | | | | | | | | | | | | X | |
| MG-composite sca | ale <sup>r</sup> | X | X | | X | 166 | X | | X | X | | X | | X | | Х | Х | X | X | X | X | |
| QMG scale <sup>s</sup> | | X | X | | X | | X | | X | X | | X | | X | | X | Х | | X | | X | |
| Muscle weakness<br>severity and fatiga<br>scale | bility | | X | e Jisel | Х | | X | | X | X | | X | | X | | Х | Х | Х | X | X | X | |
| Fatigue scale | | | X. | | X | | X | | X | X | | Х | | X | | х | Х | X | X | X | X | |
| MGADL scale | | 25 | X | | | | | | | X | | | | | | Х | | X | | | X | |

### Table 5.1: Schedule of assessments

| Assessments | Screen | ning | Trea | tment P | eriod | | | | | | | | | | | Obs | serva | <del>)</del> | UV | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ng Perio | od 1 | | | | | Dos | ing Per | riod 2 | | | | | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 150 | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> | 9 | 15 <sup>d</sup> | 16 | 22 <sup>d</sup> | 29 <sup>d</sup> | 30 | 36 <sup>d</sup> | 37 | 43 <sup>d</sup> | 44 | 500 | 57 | 64 | 78 | 92 | 99 | |
| | | | | | (± 2<br>days) | | (± 2<br>days) | | (± 2 days) | (± 2<br>days) | | (± 2<br>days) | ) | (± 2<br>days) | 793 | | (± 2 | days) | | | (± 2 days) | |
| MGII | | | X | | | | X | | | X | | | | X | <i>D</i> . | | X | | X | | X | |
| MGFA classificati | ion | X | X | | | | | | | X | -1 | | S. | 10 | | | | | | | X | |
| Jitter (SFEMG)<br>measurement <sup>t</sup> | | | X | | | | | | | X | R | Ó | Ship | | | | | | | | | |
| Headache question | nnaire <sup>u</sup> | | X | X | X | X | X | X | X | $\mathcal{I}_{\mathbf{X}}$ | X | X | X | X | X | X | X | X | X | X | X | X |
| Stool sample asses | ssment | | X | | X | | X | | X,C | X | NI CO | X | | X | | X | X | X | X | X | X | X |
| Subject exit interv | riew | | | | | | | 2 | | Jil. | | | | | | | | | | | X | |

AE=adverse event; BAFF=B-cell activating factor; BL=Baseline; BP=blood pressure; CSF=cerebrospinal fluid; CT=computed tomography; DNA=deoxyribonucleic acid; ECG=electrocardiogram; FV=Final Visit; GI=gastrointestinal; HIV=human immunodeficiency virus; IgA=immunoglobulin A; IgE=immunoglobulin E; IgG=immunoglobulin G; IGRA= interferon-gamma release assay; IgM=immunoglobulin M; IMP=investigational medicinal product; IRT=interactive response technology; LP=lumbar puncture; MG=myasthenia gravis; MGADL=myasthenia gravis-Activities of Daily Living; MGFA=Myasthenia Gravis Foundation of America; MRI=magnetic resonance imaging; PEOT=premature end of treatment; PK=pharmacokinetics; PR=pulse rate; RNA=ribonucleic acid; QMG=Quantitative Myasthenia Gravis; B; SFEMG=single fiber electromyogram; TB=tuberculosis; UV=Unscheduled Visit


<sup>&</sup>lt;sup>a</sup> Subjects will return to the clinic/hospital for Visits 15, 16, 18, and 20; for Visits 17 and 19 subjects will either return to the clinic/hospital, or, if possible and agreed by both the investigator and subject, have home visits conducted by certified healthcare professionals.

<sup>&</sup>lt;sup>b</sup> This visit is a telephone contact 24 hours post-IMP dose start.

<sup>&</sup>lt;sup>c</sup> Subjects who withdraw early will be encouraged to complete the PEOT Visit plus the FV (approximately 8 weeks after the final study drug administration).

d A visit window of ±2 days is allowed for the dosing visits. The visit window of ±2 days is relative to the first dosing visit date. However, there should be a minimum interval of 5 days and maximum interval of 9 days as compared to the previous dose.

<sup>&</sup>lt;sup>e</sup> Includes consent for jitter (SFEMG) for the subjects consenting to this measurement at the participating sites. Additional informed consent is needed for participation in the exploratory genomic substudy.

Systolic and diastolic BP, pulse rate, temperature, and respiratory rate. On dosing days, vital signs will be measured prior to IMP administration, 15 minutes after the start of the infusion, at the end of the infusion, 2 hours after the end of infusion and 4 hours after the end of the infusion. At nondosing visits, vital signs need only be taken once during the visit.

- <sup>g</sup> Body weight at Screening and at Visit 9 will be used for calculation of dose; height will be assessed only at Screening.
- h In addition to Screening and the FV, a full neurological examination should be performed for any subject who experiences severe headache.
- A query for suicidal ideation will be asked by Investigator at each clinical visit (including Visit 17 or Visit 19 when it is conducted at the clinic). A full Columbia Suicide Severity Rating Scale (C-SSRS) assessment will be performed only when subject has a positive response to the suicidal ideation query. If a subject has active suicidal ideation as confirmed by the answer 'Yes' to Question 4 or Question 5 of the C-SSRS assessments, the subject will be excluded or withdrawn from the study and immediately referred to a Mental Healthcare Professional.
- j ECGs will be read by a central reader.
- <sup>k</sup> The IGRA test will be performed in a central laboratory. Subject should not be dosed until IGRA result is available and negative.
- Pre- and postdose at Visits 2, 4, 6, 9, 11, and 13; postdose samples are to be taken 4 hours after the infusion has ended
- <sup>m</sup> Blood sample to be taken prior to dosing of IMP.
- <sup>n</sup> Urine pregnancy test will be performed using a dipstick test; a positive urine pregnancy test must be confirmed using a serum pregnancy test.
- <sup>o</sup> Sampling will be performed predose at Visit 2 and 4 hours postdose at Visits 2, 4, 6, 9, 11 and 13. A sample will be obtained at Visit 20.
- <sup>p</sup> Sampling for exploratory safety biomarkers at Baseline (Visit 2) and 4 hours post dosing (Visit 2) for all subjects. During follow up only in subjects with severe headache and/or moderate to severe GI disturbances.
- <sup>q</sup> Sampling will be performed pre- and 4 hours postdose at Visits 2, 6, 9 and 13. A sample will be obtained at Visit 20. Samples will be obtained at Visits 4 and 11 for subjects with an infusion reaction.
- This assessment will be performed at the clinic/hospital. If the subject has a home visit with certified health professionals at Visit 17 and Visit 19, this assessment will not be performed.
- Subjects should not take pyridostigmine (or any inhibitor medication) from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last any inhibitor dosing for each evaluation during the study.
- <sup>u</sup> This assessment is applicable only to subjects experiencing severe headaches and will be performed daily until resolution (ie, if headache becomes moderate or mild, normal collection of AEs should apply); this assessment will be followed by a neurological assessment (including fundoscopy). Additionally, other diagnostic procedures including but not limited to CT scan, MRI and/or LP for CSF collection to be performed if indicated at the discretion of the investigator.
- V Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally.

#### 5.3 Schematic diagram

Figure 5.1 presents a schematic diagram of the study design.

Figure 5.1: Schematic diagram



#### Rationale for study design and selection of dose 5.4

### Choice of study design and endpoints 5.4.1

The primary objective of the study is to evaluate the clinical efficacy of UCB7665 as a chronic-intermittent treatment for subjects with moderate to severe generalized MG. Additionally, this study will provide data for future study planning, whether for chronicintermittent treatment or a longer therapy option by evaluating the general concept that UCB7665 has a clinical effect in patients with generalized MG.

During the first Treatment Period, a 2-arm parallel design study will allow comparison of the change from Baseline in QMG score to Visit 9 (Day 29) between UCB7665 7mg/kg and placebo.

The choice of the primary efficacy outcome measures and the timing of approximately 4 weeks after the first dose of study drug are predicted to be the optimal approach to measure improvements based on effect seen in other therapies and recommendations of the Scientific Advisory Board of the MGFA (Barth 2013; Benatar 2012; Howard 2013). Then the second Dosing Period with a rerandomization allows for additional supportive data to be evaluated as well as offering the placebo subjects a chance to receive UCB7665.

Each subject will be asked to participate up to a maximum of approximately 18 weeks. consisting of a Screening Period (14 to 28 days), Treatment Period (6 weeks) and an Observation Period (8 weeks). The Treatment Period will consist of Dosing Period 1 followed by Dosing Joseph Period 2.

Joseph Period 2.

Joseph Period 2.

Joseph Period 2.

Joseph Period 2.

Joseph Period 2.

Joseph Period 2.

Joseph Period 2.

Joseph Period 3.

Joseph Period 2.

Joseph Period 4.

Joseph Period 5.

Joseph Period 5.

Joseph Period 6.

Joseph Period 6.

Joseph Period 7.

Joseph Period 7.

Joseph Period 8.

Joseph Period 9.

Joseph Period 1.

Joseph Perio Period 2. Dosing Period 1 will have 2 parallel Treatment Groups (UCB7665 7mg/kg or placebo)

change from Baseline in QMG score compared to placebo at Visit 9, will be assessed for subjects treated with 7mg/kg UCB7665 vs subjects treated with placebo in Dosing Period 1. The comparison of the change from Baseline in QMG score at Visit 16 in Group 3 will strengthen analyses of the results of the primary outcome measure in Group 1. Because subjects in both Group 1 and 2 will be dosed for 6 times over 6 weeks, the data from these subjects will inform safety and the development of ADAs with extended dosing durations. Data regarding dose response and the time to clinical and PD response from Group 3 (7mg/kg) vs. Group 4 (4mg/kg) in the second Dosing Period will be able to be compared. Furthermore, safety and efficacy data from Group 2 in particular will provide information addressing the concept of treating subjects with a higher "loading" dose and then maintaining them on a lower dose regimen.

#### 5.4.2 Rationale for dose selection

The dose and regimen of IMP to be used in the current study (UCB7665 7mg/kg sc) was selected based on the results from the first-in-human study UP0018. UP00018, a single ascending dose study in healthy subjects, explored the dose range of UCB7665 (between 1 and 7mg/kg) and characterized the PK and PD effect on total IgG. Data indicate that mean absolute decreases in IgG and mean percent change from Baseline IgG were greater in the active dose groups (n=6 each) compared to the pooled iv and sc placebo group (n=12) with maximum decreases of 49.3% (range: 44.6% to 55.9%) observed on Day 6 for a UCB7665 7mg/kg iv dose and 42.8% (range: 39.6% to 48.6%) on Day 9 for a UCB7665 7mg/kg sc dose. UCB7665 was tolerated with an acceptable safety profile after the single administration of a 7mg/kg sc dose, and all subject reported TEAEs had a maximum intensity of mild or moderate.

The dose-exposure-response relationship, with serum total IgG as primary endpoint, was determined using nonlinear mixed effects modeling. The derived population PK-PD (structural PK-PD model based on that of Lowe [Lowe et al, 2010]) was then used to guide, through simulation, the selection of appropriate repeat-dose regimens that would mimic decreases achieved by plasmapheresis paradigms and result in an IgG reduction of 70% or greater. The

model based simulations demonstrate that weekly doses of UCB7665 7mg/kg for 3 consecutive weeks are expected to produce maximum mean IgG reductions of >70%. Thus, exploratory comparisons of the 4mg/kg and 7mg/kg dosing regimens for treating adult subjects with moderate to severe generalized MG will be evaluated in the current study, MG0002.

### 5.4.3 Justification for additional genomic analyses

### **DNA** analysis

Monozygotic MG twin concordance is estimated to be about 35% supporting the central role of environmental factors in MG etiology. MicroRNAs provide a mechanistic link between environmental and genetic risk factors in disease development, and are providing support for specific epigenetic mechanisms associated with MG. Genetic studies have mainly pointed at specific human leukocyte antigen alleles implicated in MG susceptibility, however recently both and

were indicated to be associated with MG in a genome wide association study.

Direct genetic and environmental/epigenetic influences are complex and require further elucidation to understand the cause, progression and potential treatment of MG. Through the collection of whole blood DNA from consenting subjects, this substudy will help enable further investigation of this complex disease, facilitate identification and characterization of genetic and/or epigenetic components of MG and will lead to important clues into the pathogenesis of MG and possibly advance understanding of drug response phenotypes.

### RNA analysis

Gene expression (mRNA) analyses have identified distinct gene transcription signatures from whole blood associated with many autoimmune diseases including rheumatoid arthritis, systemic lupus erythematosus, ITP, and MG. Such signatures have provided molecular insight into disease biology and activity and can facilitate patient stratification via gene expression panels predictive of therapeutic response and clinical outcomes.

MicroRNAs are short (19-25 nucleotides) evolutionarily conserved single-stranded RNA molecules that regulate the expression of genes involved in diverse biological processes. The effect of miRNA on mRNA is mediated through the binding of the miRNA to the target mRNA ribonucleoprotein complex resulting in altered expression and decreased protein translation.

Collection of blood for RNA analysis will facilitate insight into the molecular etiology of MG at the genomic level and may enable identification of candidate markers for treatment effect and safety, and assessment of the feasibility of patient stratification.

In summary, the genetic, epigenetic, and genomic elements of MG require further elucidation to understand the cause, progression, and appropriate treatment of MG. Through the voluntary collection of blood DNA and RNA samples from consenting subjects, this substudy will help enable further investigation of this complex disease.

### 6 SELECTION AND WITHDRAWAL OF SUBJECTS

### 6.1 Inclusion criteria

To be eligible to participate in this study, all of the following criteria must be met:

- 1. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject.
- 2. Subject is  $\geq 18$  years of age at Visit 1 (Screening).
- 3. Subject has a well-documented diagnosis of MG at Visit 1 (Screening), based on subject history and supported by previous evaluations.
- 4. Subject would currently be considered for treatment with immunological therapy (eg IVIG/PLEX) by the investigator.
- 5. Subject has a well-documented record of autoantibodies against Visit 1 (Screening).
- 6. Female subjects of child bearing potential must have a negative serum pregnancy test at the Screening Visit, which is confirmed to be negative by urine testing prior to the first dose of study drug at Week 1 (Visit 2) and prior to further dosing at each study visit thereafter.
  - Female subjects of childbearing potential must agree to use a highly effective method of birth control, during the study and for a period 2 months after their final dose of study drug. According to the International Council for Harmonisation (ICH) M3 (R2), highly effective forms of birth control are methods which achieve a failure rate of less than 1% per year when used consistently and correctly. Highly effective methods of birth control include:
  - Combined (estrogen- and progesterone-containing) hormonal contraception (oral, implant, injectable) associated with inhibition of ovulation, (which must be stable for at least 1 full month prior to Screening [Visit 1], and should remain stable during the study).
  - Progesterone-only hormonal contraceptives (oral, implant, injectable) associated with inhibition of ovulation (which must be stable for at least 1 full month prior to Screening [Visit 1], and should remain stable during the study).
  - Progesterone-releasing intrauterine systems or the TCu 380A intrauterine device.
  - Vasectomized partner (provided sole partner and partner has medical proof of surgical success).
  - True heterosexual sexual abstinence is an acceptable form of contraception when this is
    in line with the preferred and usual lifestyle of the person. Periodic abstinence (eg,
    calendar, ovulation, symptothermal, postovulation methods), declaration of abstinence for
    the duration of the study, and withdrawal are not acceptable methods of contraception.

Women not agreeing to use birth control must be of nonchildbearing potential, defined as being:

- Postmenopausal (for at least 2 years before the Screening Visit), verified by serum follicle stimulating hormone level >40mIU/mL at the Screening Visit, or
- Permanently sterilized (eg, bilateral tubal occlusion, hysterectomy, bilateral salpingectomy), or

- Congenitally sterile
- 7. Contraception methods for male subjects and their female partners:
  - Male subject with a partner of childbearing potential must be willing to use a condom when sexually active during the study and for 3 months after the final administration of IMP.
  - In addition the female partner of childbearing potential of a male subject must be willing to use a highly effective method of contraception (as above), during the study period and

- Subjects are not permitted to enroll in the study if any of the following criteria are metals.

  1. Subject has previously received treatment in this study or subject to UCB7665
- 2. Subject has participated in another study of an IMP (or a medical device) within the previous 30 days of Screening or is currently participating in another study of an IMP (or a medical device).
- 3. Subject has a known hypersensitivity to any components of the IMP.
- 4. Subject has a history of hyperprolinemia, since L-proline is a constituent of the UCB7665 IMP.

#### 6.2.1 Exclusion criteria related to health status

- 5. Subjects with MG only affecting the ocular muscles.
- 6. Subjects with severe weakness affecting or opharyngeal or respiratory muscles, or who have myasthenic crisis at Screening or impending crisis.
- 7. Subject has QMG score of <11 at Baseline.
- 8. Subject has a serum total IgG level ≤6g/L at Screening.
- 9. Absolute neutrophil count \$1500 cells/mm<sup>3</sup>.
- 10. Subject has any medical condition (acute or chronic illness) or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study.
- 11. Subject has any laboratory abnormality that, in the opinion of the investigator, is clinically significant, has not resolved at randomization, and could jeopardize or would compromise the subject's ability to participate in this study.
- 12. Subject has 12-lead ECG with changes considered to be clinically significant upon medical review. The ECG contains findings that may represent a significant abnormality. The clinical significance of the findings needs to be assessed by the investigator to determine eligibility. and any queries regarding continuation of the subject must be addressed with the medical monitor.

- 13. A screening glycosylated hemoglobin HbA1c value >8%, for subjects with known history of diabetes mellitus.
- 14. Subject has renal impairment, defined as:
  - Serum creatinine level of ≥1.4mg/dL for females and ≥1.5mg/dL for males at Screening Visit
- 15. Subject has >2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%).

For randomized subjects with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin but <1.5xULN, a Baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report Form (eCRF).

If subject has >ULN, ALT, AST, or ALP that does not meet the exclusion limit at Screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the subject must be discussed with the medical monitor.

Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit (>2xULN) may be repeated once for confirmation. This includes rescreening.

- 16. Female subject who is pregnant or lactating.
- 17. Subject has planned an elective surgical procedure in the coming 6 months.
- 18. The subject is not considered reliable and capable of adhering to the protocol visit schedule, or medication intake according to the judgment of the investigator.
- 19. Subject has a history of chronic alcohol or drug abuse within the previous 12 months.
- 20. Subject has a clinically relevant active infection (eg, sepsis, pneumonia, or abscess) or has had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to the first dose of IMP.
- 21. Subject has a history of clinically relevant ongoing chronic infections including but not limited to human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C, or who tests positive for HIV, Hepatitis B, or Hepatitis C at the Screening Visit.
- 22. Subject has a family history (immediate family member) of primary immunodeficiency.
- 23. Subject has active neoplastic disease or history of neoplastic disease within 5 years of study entry (except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix which has been definitively treated with standard of care approaches).
- 24. Subject has a history of a major organ transplant or hematopoietic stem cell/marrow transplant.
# 6.2.2 Exclusion criteria related to concomitant medications/procedures

- 25. Subject has received a live vaccination within 8 weeks prior to the Baseline Visit; or intends to have a live vaccination during the course of the study or within 7 weeks following the final dose of IMP.
- 26. Subject has received any experimental biological agent within or outside of a clinical study in the past 3 months or within 5 half-lives prior to Baseline (whichever is longer).
- 27. Subject has had prior treatment with rituximab in the 6 months prior to the Baseline Visit or subject has had prior treatment with rituximab in the 12 months prior to Baseline and B cells monitoring has shown they did not return to normal range.
- 28. Subject has been treated with immunosuppressants, biologics, and other therapies as detailed in the recent timeframe as detailed in Table 6.1 OR has not been on stable dosing regimens of the medications as detailed in Table 7.1.
- 29. Exclusion Criterion 29 was deleted per Protocol Amendment 1.
- 30. Subject had a thymectomy in the past 6 month or a thymoma at any time that required chemotherapy and/or radiotherapy.

Table 6.1: No-treatment periods for exclusionary immunosuppressants, biologics, and other therapies

| Generic name (commercial/trade names) | Period relative to Baseline Visit (regardless of |
|---|---|
| | route) |
| Immunosuppressants | orile |
| Cyclophosphamide (Cytoxan®) | |
| Pimecrolimus (Elidel®) | |
| Vinca alkaloids (vincristine, vinblastine) | |
| Biologics (mabs and fusion proteins) | |
| Abatacept (CTLA 4-Ig) (Orencia®) | |
| Belimumab (Benlysta <sup>TM</sup> ) | |
| Golimumab (Simponi <sup>TM</sup> ) | |
| Natalizumab (Tysabri®) | |
| Ofatumumab (Arzerra) | |
| Rituximab (Rituxan®) and ocrelizumab | |
| TACI-Ig (Atacicept) | |
| Veltuzumab | |
| Other biologics | |
| Others | |
| Intravenous or subcutaneous immunoglobulin | |

| Generic name (commercial/trade names) | Period relative to Baseline Visit (regardless of route) |
|---|---|
| IPP-201101 (Lupuzor <sup>TM</sup> ) | |
| PLEX (plasma exchange) | |
| Immunoabsorption | |

#### 6.2.3 Exclusion criteria related to other risks

- y of suicide attempt (including an or has suicidal ideation in the past 6 months as indicated by a ther Question 4 or Question 5 of the Columbia-Suicide Severitreening.

  losis (TB) infection, at high LTBI), or com-31. Subject has a lifetime history of suicide attempt (including an positive response (Yes) to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening.
- 32. Subjects with known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent tuberculosis infection (LTBI), or current/history of nontuberculous mycobacterial infection (NTMBI) are excluded.
  - a. Known TB infection whether present or past is defined as:
  - Active TB infection or clinical signs and symptoms suggestive of TB (pulmonary or extrapulmonary).
  - History of active TB infection involving any organ system or findings in other organ systems consistent with TB infection.
  - Any historical evidence by radiography or other imaging modalities consistent with previously active TB infection.
  - b. High risk of acquiring TB infection is defined as:
  - Known exposure to another person with active TB infection within the 3 months prior to Screening.
  - Time spent in a healthcare delivery setting or institution where individuals infected with TB are housed and where the risk of transmission of infection is high.
  - c. LTBI (see Section 12.3) for further details and instructions).
  - d. NTMBI is defined as a group of lung infections caused by mycobacteria different from mycobacterium tuberculosis infections.

### 6.3 Rescreening and Rechecking

Subjects with isolated results that are outside the specified ranges and that are deemed potentially clinically significant will be allowed to rescreen at the discretion of the investigator, following discussion with the sponsor's medical monitor/study physician, if appropriate.

If a subject has 1 isolated test result outside the specific range which is deemed clinically nonsignificant, the abnormal value may be rechecked at the discretion of the investigator, following discussion with the sponsor's medical monitor/study physician. If the normalization of the test result occurs within the Screening Period, then no other Screening procedures need to be repeated.

### 6.4 Withdrawal criteria

Subjects are free to withdraw from the study at any time, without prejudice to their continued care.

Subjects MUST be withdrawn from the study if any of the following events occur:

- 1. Subject withdraws his/her consent.
- 2. Subject becomes pregnant during the study, as confirmed by a positive pregnancy test.

Subjects MUST discontinue IMP if any of the following events occur:

- 1. Subject develops an illness or has a change in health status that would interfere with his/her continued participation, including but not limited to:
  - Subject has a serious infective episode requiring hospitalization or iv antibiotic therapy (including but not limited to bacteremia or sepsis, bacterial meningitis, osteomyelitis or septic arthritis, bacterial pneumonia, or visceral abscess).
  - Subject experiences a severe adverse event (AE) of GI disturbance or severe headache which is considered related to the IMP in the opinion of the investigator (Section 12.1.10).
  - Subject has an AE of infusion reaction of severe intensity requiring corticosteroid and/or epinephrine therapy.
  - Subject has an AE of anaphylactic reaction requiring corticosteroid and/or epinephrine therapy.
  - Subject has a TB test that is confirmed positive or any further evidence suggestive of potential TB infection (eg. exposure) and further examinations result in a diagnosis of active TB or LTBI (refer to Section 12.3.1) for further details and instructions.
  - If an NTMBI is identified during a study, the same withdrawal procedures as those used for an active TB infection identified during the study should be followed.
- 2. The sponsor or a regulatory agency requests withdrawal of the subject.
- 3. Subject is treated with rescue therapy (refer to Section 7.8.3).
- 4. Subject received rituximab during the Treatment Period.
- 5. Subject received prohibited concomitant medications (as defined in Section 7.8.2 of this protocol) during the Treatment Period.
- 6. According to the investigator's judgment this is in the best interest of the patient.
- 7. Meets criteria for liver injury (Section 6.4.1).
- 8. Subject has active suicidal ideation as indicated by a positive response (Yes) to either Question 4 or Question 5 of the "Since Last Visit" version of the C-SSRS. The subject should be referred immediately to a Mental Healthcare Professional.

Subjects MAY be withdrawn from the study at the discretion of investigator, medical monitor, and study physician if any of the following events occur:

Subject is noncompliant with the study procedures or medications in the opinion of the investigator.

Subjects who withdraw from the study or discontinue IMP should complete the assessments outlined for the Premature End Of Treatment (PEOT) Visit (see Table 5.1 and Section 8.5). Subjects will be encouraged to return to the clinic/hospital to complete the Observation Period Visits and the FV (approximately 8 weeks after the final study drug administration).

Investigators should attempt to obtain information on subjects in the case of withdrawal.

For subjects considered as lost to follow up, the investigator should make an effort (at least 1 phone call and 1 written message to the subject), and document his/her effort (date and summary of the phone call and copy of the written message in the source documents), to complete the final evaluation. All results of these evaluations and observations, together with a narrative description of the reason(s) for IMP discontinuation and subject withdrawal, must be recorded in the source documents. The eCRF must document the primary reason for withdrawal or discontinuation, plus whether or not the blind was broken, with the reason and date for this.

Investigators should contact the medical monitor, whenever possible, to discuss the withdrawal of a subject in advance. Subjects who are withdrawn will not be replaced.

# 6.4.1 Potential drug-induced liver injury IMP discontinuation criteria

Subjects with potential drug-induced liver injury (PDILI) must be assessed to determine if IMP must be discontinued. In addition, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued.

The PDILI criteria below require immediate and permanent discontinuation of study drug:

- Subjects with either of the following:
  - ALT or AST ≥5xULN
  - ALT or AST ≥3xULN and coexisting total bilirubin ≥2xULN

The PDILI criterion below requires immediate discontinuation of study drug:

• Subjects with ALT or AST ≥3xULN who exhibit temporally associated symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, right upper quadrant pain or tenderness. Hypersensitivity symptoms include fever (without clear alternative cause), rash, or eosinophilia (ie, >5%).

If a nondrug-related cause for the symptoms can be confirmed, these subjects may resume study drug administration after discussion with the responsible UCB physician, but only when the requirements for rechallenge with study drug as provided in Section 12.2.1.2.1 are followed.

The PDILI criterion below allows for subjects to continue on study drug at the discretion of the investigator.

Subjects with ALT or AST  $\ge 3x$ ULN (and  $\ge 2x$  Baseline) and < 5xULN, total bilirubin < 2xULN, and no eosinophilia (ie,  $\le 5\%$ ), with no fever, rash, or symptoms of hepatitis (eg, fatigue, nausea, vomiting, right upper quadrant pain or tenderness).

Evaluation of PDILI must be initiated as described in Section 12.2.1. If subjects are unable to comply with the applicable monitoring schedule, IMP must be discontinued immediately.

Investigators should attempt to obtain information on subjects in the case of IMP discontinuation to complete the final evaluation. Subjects with PDILI should not be withdrawn from the study until investigation and monitoring are complete. All results of these evaluations and observations, as well as the reason(s) for IMP discontinuation and subject withdrawal (if applicable), must be recorded in the source documents. The eCRF must document the primary reason for IMP discontinuation.

### 7 STUDY TREATMENT

# 7.1 Description of investigational medicinal product



or sc administration, is supplied with a commercial source.

# 7.2 Treatments to be administered

Dosing Period 1: Subjects will be randomized in a O1 manner to receive either:

• 3 sc doses of UCB7665 7mg/kg at 1 week intervals

OR

3 sc doses of placebo
 at 1 week intervals

After completing Dosing Period 1, subjects will enter Dosing Period 2.

Dosing Period 2: Subjects will be rerandomized in a 1:1 manner to receive either:

- 3 sc doses of UCB7665 7mg/kg at 1 week intervals
   OR
- 3 sc doses of UCB7665 4mg/kg at 1 week intervals

The IMP will be administered as a sc infusion using an infusion pump.

The perfusor will be programmed at a constant flow rate of for all subjects. In the case of any blockage of the infusion, a suitable flush (eg, infusion time will be set to for all subjects.

The subject's body weight at the Screening Visit and Visit 9 will be used for the dose calculation. Screening Visit is for dosing in Period 1 and Visit 9 is for dosing in Period 2.

The exact procedure for dose preparation according to Treatment Group and body weight will be provided in an IMP Handling Manual.

The infusion rate may be reduced at any time at the discretion of the investigator. If an infusion is interrupted, it can be restarted if the investigator considers it appropriate to do so. The


chronology of these events (infusion start and stop time) should be recorded accurately in the source data and eCRF, along with the volume infused, and the location of the infusion.

# 7.3 Packaging

The IMP will be manufactured, packaged, and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. The IMP will be suitably packaged in such a way as to protect it from deterioration during transport and storage.

# 7.4 Labeling

Clinical drug supplies will be labeled in accordance with the current ICH guidelines on Good Clinical Practice (GCP) and GMP and will include any locally required statements. If necessary, labels will be translated into the local language.

# 7.5 Handling and storage requirements

The investigator (or designee) is responsible for the safe and proper storage of IMP at the site. Investigational medicinal product stored by the investigator is to be kept in a secured area with limited access according to the storage conditions mentioned on the label.

Appropriate storage conditions must be ensured either by controlling the temperature (eg, room, refrigeration unit) or by completion of a temperature log in accordance with local requirements on a regular basis (ie, every workday), showing actual and minimum/maximum temperatures reached over the time interval.

In case an out-of-range temperature is noted, it must be immediately reported as per instructions contained in the IMP Handling Manual.

# 7.6 Drug accountability

A Drug Accountability form will be used to record IMP dispensing and return information on a by-subject basis and will serve as source documentation during the course of the study. Details of any IMP lost, damaged (due to breakage or wastage), not used, partially used, disposed of at the study site, or returned to the sponsor or designee must also be recorded on the appropriate forms. All supplies and pharmacy documentation must be made available throughout the study for UCB (or designee) to review.

The investigator (or designee) is responsible for retaining all used, unused, and partially used containers of IMP until returned or destroyed.

The investigator may assign some of the investigator's duties for drug accountability at the study site to an appropriate pharmacist/designee.

The investigator must ensure that the IMP is used only in accordance with the protocol.

Periodically, and/or after completion of the clinical phase of the study, all used (including empty containers), partially used, unused, damaged, and/or expired IMP must be reconciled and either destroyed at the site according to local laws, regulations, and UCB Standard Operating Procedure (SOPs), or returned to UCB (or designee). Investigational medicinal product intended for the study cannot be used for any other purpose than that described in this protocol.

### 7.7 Procedures for monitoring subject compliance

Drug accountability is ensured by administering the IMP as sc infusion by designated personnel. Drug accountability must be recorded on the Drug Accountability form.

#### 7.8 Concomitant medication/treatment

#### 7.8.1 Permitted concomitant medication

ons or variations thereof Table 7.1 lists the concomitant medications that are permitted during the course of the study at a stable dose.

**Table 7.1:** Permitted concomitant treatments

| Permitted<br>Medications | Dose | Comment |
|---|---|---|
| Oral Corticosteroids (eg, prednisolone) | - | |
| Methotrexate | ≤30mg/week | |
| Mycophenolate mofetil | ≤3g/day | |
| Cyclosporin <sup>a</sup> | ≤5mg/kg/day for<br>unmodified<br>≤4mg/kg/day for modified<br>(microemulsion) | |
| Azathioprine | ≤3mg/kg/day | |
| Cholinesterase inhibitors | ≤600mg<br>Pyridostigmine/day | |
| Tacrolimus <sup>b</sup> | ≤5mg/day | |

<sup>&</sup>lt;sup>a</sup> Doses higher than listed are permissible if trough level is ≤300ng/L.

Subjects should not take pyridostigmine (or any midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post any last medication inhibitor dosing for each evaluation during the study.

<sup>&</sup>lt;sup>b</sup> If the total daily weight-based dose is >5mg, then a plasma trough level should be checked to ensure subject is not above the recommended therapeutic range.

In the event of a subject developing an infection during the course of the study, samples for culture will be taken prior to commencing antimicrobial treatment. Antimicrobial treatment may be modified accordingly when the identity of the infective organism is known.

#### 7.8.2 Prohibited concomitant treatments (medications and therapies)

The following concomitant medications and therapies are prohibited during the study:

- IVIg
- All biologics including rituximab
- Cyclophosphamide
- **Pimecrolimus**
- IPP-201101 (Lupuzor<sup>TM</sup>)
- **PLEX**
- Immunoadsorption
- 3 any extensions or variations thereof. Medications which could interfere with the function of the NMJ (and which therefore could impair subjects with MG), such as, but not limited to, the following medications. For a more ed stind authorization detailed list please refer to the MGFA medication list (http://www.myasthenia.org/LivingwithMG/DrugstoAvoid.aspx).
  - botulinum toxin
  - aminoglycoside antibiotics
  - tetracycline antibiotics
  - penicillamine

If a subject needs or takes any prohibited medication or therapy (except IVIg, PLEX, or rituximab), the investigator will (where possible) discuss with the sponsor study physician and a decision will be made whether the subject can continue in the study or must be withdrawn. If the subject is treated with IVIg, rituximab, or PLEX, the subject must be withdrawn from the IMP, but should be encouraged to continue with Observation Period Visits.

For subjects who require a medical or surgical procedure that requires the use of general anesthesia, discussion must occur prior to the procedure with the medical monitor or study physician. In an emergency situation, discussion should occur as soon as possible after the procedure, such that a decision on the subject's continued participation in the study can be made.

#### Rescue medication 7.8.3

In the case of prolonged hypogammaglobulinemia the subject will be considered for treatment with prophylactic antimicrobial therapy. Subjects will be followed up until Ig levels return to within the normal range.

If, during the Treatment and Observation Period, in the opinion of the investigator, a subject has a significant deterioration in clinical condition, then rescue therapy such as IVIg or PLEX should be considered.

#### 7.9 Blinding

#### 7.9.1 Procedures for maintaining and breaking the treatment blind

#### 7.9.1.1 Maintenance of study treatment blind

All subject treatment details, ie, UCB7665 4mg/kg, 7mg/kg sc, or placebo, will be allocated and maintained by the IRT system.

The following individuals will receive the randomization and the system. and variensions of variors of var

- Sponsor and designated bioanalytical staff analyzing PK samples
- Sponsor clinical trial supply staff
- IRT provider

Study site pharmacists or other suitably qualified site personnel who are responsible for preparation of IMP treatments and any necessary assistants will have access to treatment allocations for individual subjects via the IRT. The unblinded pharmacy monitors from the Contract Research Organization (CRO), the Clinical Supply Manager, and the unblinded Clinical Project Manager (CPM) (or designee) will also have access to the treatment allocations and to the drug accountability records, if applicable.

The following individuals may, as necessary, have access to the randomization code as indicated:

- Sponsor Patient Safety (PS) staff as needed for reporting SAEs to regulatory authorities.
- On request, members of the DMC who participate in unblinded sessions will be given information about the IMP allocation for those subjects for whom data are provided at these sessions.
- Sponsor and/or CRO staff supporting preparation of the data outputs for the DMC review and/or any interim analyses.
- A Quantitative Clinical Pharmacologist/Modeling and Simulation Scientist may have access to the randomization code if PK data are requested for review by the DMC.

All subject treatment details will be allocated and maintained by the IRT system.

### Breaking the treatment blind in an emergency situation 7.9.1.2

In the event of an emergency, it will be possible to determine to which Treatment Group and dose the subject has been allocated by contacting the IRT. All sites will be provided with details of how to contact the system for code breaking at the start of the study. The medical monitor or equivalent should be consulted prior to unblinding, whenever possible. The study blind should not be broken except in a medical emergency, where knowledge of the study drug received would affect the treatment of the emergency.

The CPM and medical monitor will be informed immediately via the IRT when a code is broken, but will remain blinded to specific treatment information. Any unblinding of the IMP performed

 by the investigator must be recorded in the source documents and on the Study Termination eCRF page.

Inadvertent unblinding has to be listed as a major protocol deviation.

# 7.10 Randomization and numbering of subjects

An IRT will be used for assigning eligible subjects to the different treatment regimens (as applicable) based on a predetermined production randomization and/or packaging schedule. The 1:1 randomization schedules will be produced by the IRT vendor. The IRT vendor will also generate lists of IMP, as appropriate, according to the visit schedule, the Treatment Group and the subject's weight.

To enroll a subject (Visit 1), the investigator or designee will contact the IRT and provide brief details about the subject to be screened. Each subject will receive a 5-digit number assigned at Screening that serves as the subject identifier throughout the study. The subject number will be required in all communication between the investigator or designee and the IRT regarding a particular subject. Subject numbers and kit numbers will be tracked via the IRT.

To enroll a subject in Dosing Period 1, the investigator or designee will contact the IRT and provide brief details about the subject to be randomized. The IRT will allocate kit numbers to the subject based on the randomization number.

To enroll a subject in Dosing Period 2, the investigator or designee will again contact the IRT and provide the subject's screening number and weight at Visit 9. The subject will be rerandomized in a 1:1 ratio to receive one of the two doses of UCB7665. The IRT will stratify the rerandomization based on the treatment received in Dosing Period 1. At this rerandomization, the subject will receive a second randomization number which, as in Dosing Period 1, will be used by the IRT to allocate appropriate kit numbers.

# 8 STUDY PROCEDURES BY VISIT

A detailed schedule of study procedures is provided in Table 5.1.

For details of the standard safety hematology, clinical chemistry, and urinalysis, see Table 12.2.

# 8.1 Screening Period

# 8.1.1 Visit 1 (Day -28 to -1) Screening Visit

At Visit 1, subjects will be evaluated for their suitability for enrollment. Prior to the conduct of any study-related procedures, a complete explanation (both verbal and written) of the nature and purpose of the study will be given to the subject by the investigator (or designee). The subject is required to sign and date the IRB/IEC-approved Informed Consent form if he/she decides to participate in the study.

Subjects will also have the option of providing additional voluntary informed consent for collection of whole blood samples for exploratory genomic (DNA and RNA) analyses.

The subject's eligibility for the study will be determined on the basis of the inclusion/exclusion criteria and signature of an informed consent prior to any study-related procedures or evaluations.

The following assessments and procedures will be performed during Visit 1 of MG0002:

- UCB7665
- Obtain written informed consent
- Obtain optional informed consent for genomic substudy
- Demographic data (includes date of birth, gender, and race/ethnicity)
- Verification of inclusion/exclusion criteria
- Cyrate) corveitation and any extensions of variations thereof.

  S will be r General medical history and medical procedures history (including history of tetanus immunization)
- Prior and concomitant medications
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Body weight and height
- Recording of AEs
- Physical examination (Full)
- Neurological examination (Full)
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - MGFA classification
- Query for suicidality (Screening)

- 12-lead ECG
- Blood samples:
  - Standard safety laboratory tests: hematology and clinical chemistry, plus serology testing for HIV, Hepatitis B, and Hepatitis C
  - Immunoglobulins (Total IgG and subclasses)
  - Vaccination-specific antibody titers (
  - Serum pregnancy test for women of childbearing potential
- Tuberculosis assessments:
  - **IGRA**
  - Tuberculosis Sign and Symptoms questionnaire
- Standard safety urinalysis
- Call or enter IRT to register the visit

### 8.2 **Dosing Period 1**

In Dosing Period 1, visits will be performed at weekly intervals.

# 8.2.1 Visit 2 (Day 1, Baseline)

Visit 2 can occur at any time after Visit 1, but no later than 28 days after Visit 1. Eligible subjects will be randomized at Visit 2 and the first dose of IMP (UCB7665 7mg/kg sc infusion) or placebo will be administered as per the subject's randomization.

The following assessments and procedures will be performed at this visit:

### Predose:

- Verification of inclusion/exclusion criteria
- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Physical examination (brief)
- Neurological examination (brief)
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
  - MGADL scale
  - MGII
  - MGFA classification
- Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

- 12-lead ECG
- Blood samples:
  - Standard safety laboratories: hematology and clinical chemistry
  - PK of UCB7665
  - Serum complement (C3,C4) and plasma complement levels (C3a and C5a)
  - Ig (total IgG and subclasses)
  - IgA, IgM, and IgE

- MG-specific autoantibodies
- Exploratory biomarker analysis
- Exploratory safety biomarkers: may include but not limited to
- BAFF
- Cytokines
- Collection of whole blood for exploratory genomic (DNA and RNA) analyses
- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential
- Call or enter to IRT/Randomization
- Jitter (SFEMG) measurement

During dosing of IMP:

- IMP administration
- ation and any extensions or variations thereof. Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs

Postdose:

- Vital signs (systolic and diastolic BP pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Stool sample assessment (if required)
  Blood samples:
- - PK of UCB7665
  - Cytokines

#### 8.2.2 Visit 3 (Day 2)

The subject will be contacted by telephone for collection of prior and concomitant medications, AEs, and withdrawal criteria data. Headache questionnaire will be completed if required. This visit should occur 24 hours after the IMP dose started.

# Visit 4 (Day 8)

The following assessments and procedures will be performed at this visit:

Predose:

- Withdrawal criteria
- Prior and concomitant medications

- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Assessment of MG status:

  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
- Query for suicidality (since last visit):

- 12-lead ECG
- Blood samples

  - Ig (total IgG and subclasses)
  - MG-specific autoantibodies
  - Exploratory biomarker analysis
  - Exploratory safety biomarkers: may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

- **BAFF**
- Collection of whole blood for exploratory RNA analysis
- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential
- Call or enterIRT to register the visit

During dosing of IMP:

- IMP administration
- Wital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs

### Postdose:

Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)

cook samples

Standard safety laboratories: hematology and clinical chemistry

PK of UCB7665

(total IgG and subclasses)

G-specific autoantibodies

bloratory

- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Blood samples
  - Serum complement (C3,C4) and plasma complement levels (C3a and C5a)
  - PK of UCB7665
  - Cytokines should be collected if infusion reaction occurs

#### 8.2.4 Visit 5 (Day 9)

Ins of variations thereof The subject will be contacted by telephone for collection of prior and concomitant medications, AEs, and withdrawal criteria data. Headache questionnaire will be completed if required. This visit should occur 24 hours after the IMP dose started.

The following assessments and procedures will be performed at this visit:

Predose:

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Assessment of MG status:
  - MG-composite scale
  - OMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
  - **MGII**
- Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

- 12-lead ECG
- Blood samples:
  - Standard safety laboratories: hematology and clinical chemistry
  - PK of UCB7665

- Ig (total IgG and subclasses)
- Exploratory biomarker analysis
- Exploratory safety biomarkers: may include but not limited to

with severe headache and/or moderate to severe GI disturbance

- BAFF
- Cytokines
- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential
- Call or enter IRT to register the visit

During dosing of IMP:

- IMP administration
- and any extensions or variations thereof. Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs

### Postdose:

- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Blood samples
  - Serum complement (C3,C4) and plasma complement levels (C3a and C5a)
  - PK of UCB7665
  - Cytokines

#### 8.2.6 Visit 7 (Day 16)

The subject will be contacted by telephone for collection of prior and concomitant medications, AEs, and withdrawal criteria data. Headache questionnaire will be completed if required. This visit should occur 24 hours after the IMP dose started.

# **Visit 8 (Day 22)**

This is a nondosing visit. The following assessments and procedures will be performed at this visit?

- Assessment of withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures

- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
- Query for suicidality (since last visit):

- 12-lead ECG
- Blood samples:
- and elimical c. Standard safety laboratories: hematology and clinical chemistry
  - PK of UCB7665
  - Ig (total IgG and subclasses)
  - IgA, IgM, and IgE
  - Exploratory biomarker analysis
  - Exploratory safety biomarkers; may include but not limited to with severe headache and/or moderate to severe GI disturbance

only in subjects

**BAFF** 

- Collection of whole blood for exploratory genomic (DNA and RNA) analyses
- Standard safety orinalysis
- Urine pregnancy test for women of childbearing potential

### **Dosing Period 2** 8.3

In Dosing Period 2, visits will be performed at weekly intervals.

#### 8,39 Visit 9 (Day 29)

Subjects will be rerandomized at Visit 9 and the IMP (UCB7665 7mg/kg or 4mg/kg sc infusion) will be administered as per the subject's randomization. The QMG and safety and efficacy assessments will be performed before rerandomization.

The following assessments and procedures will be performed at this visit:

ation and any extensions or variations thereof, strong and any extensions or variations thereof.

### Predose:

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- scale

  ACTED COPT

  Will. Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Body weight
- Recording of AEs
- Physical examination (brief)
- Neurological examination (brief)
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
  - MGADL scale
  - MGII
  - MGFA classification
- Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

- 12-lead ECG
- Blood samples:
  - Standard safety laboratories: hematology and clinical chemistry
  - PK of UCB7665
  - Ig (total IgG and subclasses)
  - IgA, IgM, and IgE
  - MG-specific autoantibodies

Exploratory biomarker analysis

Exploratory safety biomarkers: may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

**BAFF** 

- Cytokines
- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential
- Call or enter to IRT/Rerandomization
- Jitter (SFEMG) measurement

### During dosing of IMP:

- IMP administration
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs

### Postdose:

- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Blood samples
  - Serum complement (C3,C4) and plasma complement levels (C3a and C5a)
  - PK of UCB7665
  - Cytokines

### 8.3.2 Visit 10 (Day 30)

The subject will be contacted by telephone for collection of prior and concomitant medications, AEs, and withdrawal criteria data. Headache questionnaire will be completed if required. This visit should occur 24 hours after the IMP dose started.

# 8.3.3 Visit 11 (Day 36)

The following assessments and procedures will be performed at this visit:

### Predose:

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Assessment of MG status:
  - MG-composite scale
  - QMG scale

- Muscle weakness severity and fatigability scale
- Fatigue scale
- Query for suicidality (since last visit):

- 12-lead ECG
- Blood samples:
  - Standard safety laboratories: hematology and clinical chemistry
  - PK of UCB766

  - Ig (total IgG and subclasses)
  - IgA, IgM, and IgE
  - MG-specific autoantibodies
  - Exploratory biomarker analysis
- tion and any extensions of variations thereof. Exploratory safety biomarkers: may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

- BAFF
- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential
- Call or enter IRT to register the visit

During dosing of IMP:

- **IMP** administration
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs

### Postdose:

- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- - Serum complement (C3,C4) and plasma complement levels (C3a and C5a)
  - PK of UCB7665
  - Cytokines should be collected if infusion reaction occurs

Blood samples

#### 8.3.4 Visit 12 (Day 37)

The subject will be contacted by telephone for collection of prior and concomitant medications, AEs, and withdrawal criteria data. Headache questionnaire will be completed if required. This visit should occur 24 hours after the IMP dose started.

#### 8.3.5 Visit 13 (Day 43)

The following assessments and procedures will be performed at this visit:

### Predose:

UCB

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
  - MGII
- Query for suicidality (since last visit):

Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

- 12-lead ECG
- Blood samples:
  - Standard safety laboratories: hematology and clinical chemistry
  - PK of UCB7665
  - Ig (total IgG and subclasses)
  - IgA, IgM, and IgE
  - Exploratory biomarker analysis

Exploratory safety biomarkers: may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

- **BAFF**
- Cytokines

- Collection of whole blood for exploratory genomic (DNA and RNA) analyses
- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential
- Call or enter IRT to register the visit
- Administration of IMP

### During dosing of IMP:

- IMP administration
- (e) ication and any extensions of variations thereof. Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs

### Postdose:

- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Blood samples
  - Serum complement (C3,C4) and plasma complement levels (C3a and C5a)
  - PK of UCB7665
  - Cytokines

#### 8.3.6 Visit 14 (Day 44)

The subject will be contacted by telephone for collection of prior and concomitant medications, AEs, and withdrawal criteria data. Headache questionnaire will be completed if required. This visit should occur 24 hours after the IMP dose started.

#### **Observation Period** 8.4

During the Observation Period, visits will be performed at weekly intervals, apart from between Visits 17, 18, and 19, when visits will be performed at 2 weekly intervals. Subjects will return to the clinic for Visits 15, 96, 18, and 20 for efficacy and for safety assessments. Subjects will either return to the clinic, or, if possible and agreed by both the investigator and the subject, have home visits conducted by certified healthcare professionals, for Visits 17 and 19. No IMP will be administered in the Observation Period.

### Visit 15 (Day 50) 8.4.1

The following assessments and procedures will be performed at this visit:

- Assessment of withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)

- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
  - MGADL scale
- Query for suicidality (since last visit):

- 12-lead ECG
- Blood samples:
- ation and any extensions or variations thereof Standard safety laboratories: hematology and clinical chemistry
  - PK of UCB7665
  - Ig (total IgG and subclasses)
  - IgA, IgM, and IgE
  - MG-specific autoantibodies
  - Exploratory safety biomarkers, may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential

### 8.4.2 Visit 16 (Day 57)

The following assessments and procedures will be performed at this visit:

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Headache questionnaire if required

and elimical c.

- Stool sample assessment if required
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
  - **MGII**
- Query for suicidality (since last visit):

- Blood samples:
- ication and any extensions or variations thereof. Standard safety laboratories: hematology and clinical chemistry

  - Ig (total IgG and subclasses)
  - IgA, IgM, and IgE
  - Exploratory safety biomarkers: may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential

#### 8.4.3 Visit 17 (Day 64)

The following assessments and procedures will be performed at this visit:

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Assessment of MG status:
  - MG-composite scale (this assessment will be performed at the clinic/hospital. If the subject has a home visit with certified health professionals, this assessment will not be performed)
  - Muscle weakness severity and fatigability scale

- Fatigue scale
- MGADL scale
- Query for suicidality (since last visit):

- Blood samples:
  - \_
  - Ig (total IgG and subclasses)
  - Exploratory biomarker analysis
  - Exploratory safety biomarkers: may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

**BAFF** 

· Urine pregnancy test for women of childbearing potential

### 8.4.4 Visit 18 (Day 78)

The following assessments and procedures will be performed at this visit:

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- · Headache questionnaire if required
- Stool sample assessment if required
- Assessment of MG status:
  - MG-composite scale
  - QMG scale
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
  - MGII
- Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

• 12-lead ECG

- Blood samples:
  - Standard safety laboratories: hematology and clinical chemistry

  - Ig (total IgG and subclasses)
  - Exploratory safety biomarkers: may include but not limited to

with severe headache and/or moderate to severe GI disturbance

- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential

#### 8.4.5 Visit 19 (Day 92)

The following assessments and procedures will be performed at this visit:

- Withdrawal criteria
- Prior and concomitant medications
- Concomitant medical procedures
- ication and any extensions of variations thereof. Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Assessment of MG status:
  - MG-composite scale (this assessment will be performed at the clinic/hospital. If the subject has a home visit with certified health professionals, this assessment will not be performed)
  - Muscle weakness severity and fatigability scale
  - Fatigue scale
- Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

Blood samples:

Ig (total IgG and subclasses)

- Exploratory biomarker analysis
- Exploratory safety biomarkers: may include but not limited to

only in subjects

with severe headache and/or moderate to severe GI disturbance

- **BAFF**
- Urine pregnancy test for women of childbearing potential

#### 8.4.6 Visit 20 (Day 99, Final Visit) and Premature End of Treatment Visit

Concomitant medications

Concomitant medications

Concomitant medical procedures

Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)

Body weight

Recording of AEs

Headache questionnaire if required

Tuberculosis Sign and Symptoms questionnaire

Itool sample assessment if required

hysical examination (full)

eurological examination (full)

seessment of MG status:

MG-composite scale

QMG scale

Muscle weakness severity and fatigability scale

Fatigue scale

MGAEY Subjects who withdraw from the study drug will be encouraged to return to the clinic to complete a PEOT Visit and an FV approximately 8 weeks after the final dose of study drug. The following assessments and procedures will be performed at the FV (and PEOT Visit if applicable):

- - MGADL scale
  - MGII
  - MGFA classification
- Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

- 12-lead ECG
- Blood samples:

Standard safety laboratories: hematology and clinical chemistry

- Serum complement (C3,C4) and plasma complement levels (C3a and C5a)
- Ig (total IgG and subclasses)



- IgA, IgM, and IgE
- MG-specific autoantibodies
- and any extensions or variations thereof. Exploratory safety biomarkers: may include but not limited to with severe headache and/or moderate to severe GI disturbance
- Vaccination-specific antibody titers (
- Cytokines
- Collection of whole blood for exploratory RNA analyses
- Standard safety urinalysis
- Urine pregnancy test for women of childbearing potential
- Call or enter IRT to register the visit
- Subject Exit Interview

#### 8.5 Premature End of Treatment Visit

All subjects who withdraw early from the study treatment should attend a PEOT Visit which will be scheduled as close as possible to the date of the decision for the study or treatment withdrawal. Subjects are encouraged to return to the clinic for all visits of the Observation Period following the PEOT Visit. An FV will be scheduled 8 weeks after the subject's final dose. In case a subject is not willing to attend the visits in the Observation Period, the subjects should still be strongly encouraged to attend at least the PEOT Visit and FV.

The assessments to be done at the PEOT Visit are the same as those at the FV (Visit 20).

#### 8.6 **Unscheduled Visit**

Unscheduled visits may include the following assessments or other assessments deemed necessary by the investigator:

- Prior and concomitant medication
- Concomitant medical procedures
- Recording of AEs
- Headache questionnaire if required
- Stool sample assessment if required
- Vital signs (systolic and diastolic BP, pulse rate, temperature, and respiratory rate)
- Cytokines
- Query for suicidality (since last visit):

If positive response (Yes), a full C-SSRS will be performed.

Other safety assessments (eg, physical examination, 12-lead ECG, laboratory assessments) may be performed at the discretion of the investigator.

In the event of a subject developing an infection during the course of the study, samples for culture will be taken prior to commencing antimicrobial treatment.

#### 9 ASSESSMENT OF EFFICACY

#### 9.1 **Quantitative Myasthenia Gravis scale**

For assessment of the QMG scale, investigators will follow the MGFA's QMG Manual instructions (see Section 18.1). Clinical personnel must complete mandatory training and be certified to assess subjects' OMG score (details are provided in the Study Procedures Manual). Subjects should not take pyridostigmine (or any inhibitor medication) from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. The scale tests 13 items, including ocular and facial involvement, swallowing speech, limb strength, and forced vital capacity (FVC). For the assessment of FVC, the same spirometer should be used each time a subject is tested, and if possible, the same person should carry out the assessment. Parameters and normal values for FVC will be decided between the study sites, such that all sites are using the same information. The QMG is a validated assessment (Barnett et al, 2012), with a higher score indicating more severe disease. Scoring for each item ranges from no weakness (0) to severe weakness (3), with an overall score range from 0 to 39. A 3 point change in the total score is considered clinically relevant. The test takes approximately 30 minutes to perform.

### MG-Composite scale 9.2

For assessment of the MG-Composite scale, the investigator will examine the subject to score all items, except for talking, chewing, and swallowing for which the subject will self-assess. The MG-Composite scale is a validated assessment (Burns et al. 2010), with a higher score indicating more severe disease (see Section 18.2) and a 3-point change being of clinical relevance. The scale tests 10 items, with individual items being weighted differently. The overall score ranges from 0 to 50. Clinical personnel must complete mandatory training and be certified to assess subjects' MG-Composite score (details are provided in the Study Procedures Manual).

### 9.3 Patient-reported outcomes

Subjects will complete 4 patient-reported outcomes (PROs) and participate in 1 subject exit interview as per time points mentioned in the schedule of study assessments in Section 5.2. Study personnel other than the treating physician should administer the PROs. The PROs should be completed by the subject themselves in a quiet place.

The PROs and the subject exit interview should be completed in the following order: MG muscle weakness and fatigability, Fatigue, MGADL and MGII, followed by the subject exit interview (which will be performed only at the FV). The PROs should only be checked for completeness. On dosing days, the PROs will be completed prior to dosing.

# 9.3.1 MG muscle weakness and fatigability

The MG muscle weakness and fatigability instrument (Appendix 18.3) consists of 27 items across 2 domains: 18 muscle weakness severity items and 9 symptom fatigability items. The subject will be asked to choose the response option that best describes the severity of muscle

weakness symptoms over the past 7 days using a 6-point Likert scale ("none" to "very severe") and how frequently they experienced symptom fatigability over the past 7 days using a 5-point Likert scale ("none of the time" to "all of the time"), respectively. The muscle weakness score ranges from 0 to 90; the fatigability score ranges from 0 to 36. The overall score ranges from 0 to 126, with a higher result indicating more severe muscle weakness and fatigability.

### 9.3.2 Fatigue

The fatigue instrument (Appendix 18.4) consists of 55 items across 3 domains: 16 physical domain items (with a scale of 16 to 80), 18 mental domain items (with a scale of 18 to 90), and 21 fatigability domain items (with a scale of 21 to 105). The subject will be asked to score each item based on how frequently she/he experienced the item during the past 7 days using a 5-point Likert scale ("none of the time" to "all of the time"). The overall score ranges from 55 to 275, with a higher result indicating more severe fatigue.

### 9.3.3 MG-Activities of Daily Living

The MGADL is an 8-item PRO instrument developed on the basis of the QMG (Wolfe et al, 1999) (Appendix 18.5). The MGADL targets symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. In a recent study, reliability, validity, and responsiveness of the MGADL were further assessed. The questionnaire showed strong construct validity when evaluated against the MG-Composite as well as against the MG-QOL15, high test retest reliability in a 1 week interval, and it was demonstrated that a 2-point improvement indicates clinical improvement (Muppidi, 2012; Muppidi et al, 2011). The total MGADL score ranges from 0 to 24, with a higher score indicating more disability. Subjects will complete the MGADL by themselves as described in the standardized administration of PROs.

# 9.3.4 Myasthenia Gravis Impairment Index

The MGII is a measure of disease severity based on the signs and symptoms of Myasthenia Gravis patients (Appendix 18.6). It was developed using a patient-centered approach and following current guidelines for outcome measure development, incorporating patient input throughout the different development phases (Barnett et al, 2014, Barnett et al, 2016). The MGII has 22 patient-reported and 6 examination items, and scores are presented as a sum of all items for a total score but also as an ocular and generalized sub-score.

The MGII has shown construct validity and reliability in an outpatient setting. It has less floor effect compared to other commonly used outcome measures, and it can effectively discriminate among patients with different degrees of severity (Barnett et al, 2016). Finally, the MGII is sensitive to detect clinical change after interventions, and most importantly it can detect patient-meaningful change. Additionally, the MGII showed more relative efficiency than the QMGS, MGC and MG-ADL to detect change in short-term interventions for Myasthenia. Estimates for the minimal important difference were developed.

### 9.4 MGFA classification

The investigator will classify the subject's MG using the MGFA Clinical Classification (Section 18.6) (Jaretzki et al, 2000). This is a 5 stage classification (I to V), with a higher class indicating more severe disease.

# 9.5 Jitter (Single Fiber Electromyography)

At participating sites, subjects consenting to jitter (SFEMG) measurement should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. If pyridostigmine is taken, the time must be documented. This measurement will be performed by adequately trained and equipped investigators. Jitter measurements may be performed with a single-fiber EMG (SFEMG) electrode having a side-ported recording surface with a 25µm diameter, or a disposable concentric needle electrode. This enables the measurement of fiber density and neuromuscular jitter (SFEMG) (which is a sensitive measurement of transmission across the NMJ) (Sanders, 2014). Jitter (SFEMG) can assist in demonstrating MG-associated abnormalities. In well treated MG, the jitter (SFEMG) displays a more normal profile.

Details of the jitter (SFEMG) performance will be described in the jitter (SFEMG) measurement manual.

# 9.6 Subject exit interview

At the FV, qualitative interviews will be conducted by a study nurse/study personnel using a semi-structured interview guide. The aim of the interview is to collect the subject's experience with MG in terms of symptoms and impact on daily activities, and the perceived changes during the course of the study. The extent to which the exploratory PRO items and scales used fully captured their experience will also be assessed. The interviews will be audio-recorded. If a subject leaves the study prematurely, he/she will also be invited to participate in an exit interview at the PEOT Visit.

# 10 ASSESSMENT OF PHARMACOKINETIC/ PHARMACODYNAMIC/PHARMACOGENOMIC VARIABLES

### 10.1 Pharmacokinetic variable

The plasma concentration of UCB7665 will be characterized. Blood samples will be drawn according to the schedule of study assessments (Section 5.2).

Blood samples will be collected pre- and post- UCB7665 dosing. Additional blood will be drawn at the predose sampling for standard clinical laboratory tests. Postdose samples will be taken 4 hours after the infusion has ended. At Visits 8 and 15, when no IMP is administered, blood for PK analysis will also be taken. The time and date of collection will be recorded in the eCRF.

Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the Laboratory Manual for this study.

# 10.2 Pharmacodynamic variables

For all PD assessments, blood samples will be collected by qualified site personnel at the same time that samples are collected for standard clinical laboratory assessments. At dosing visits, these samples will be collected predose. Blood samples for PD analysis will be drawn according to the schedule of study assessments (Section 5.2). The time and date of collection will be recorded in the eCRF.

Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the Laboratory Manual for this study.

The following will be measured:

- Serum total IgG concentrations
- Serum IgG subclass concentrations
- Serum MG-specific autoantibody ( ) levels

#### 11 ASSESSMENT OF OTHER VARIABLES

#### 11.1 Assessment of other immunological variables

, or variations thereof. At levels

At levels

At levels For all immunological assessments, blood samples will be collected by qualified site personnel at the same time that samples are collected for standard clinical laboratory assessments. At dosing visits, these samples will be collected predose. The time and date of the blood draws will be recorded in the eCRF. The following immunological assessments will be performed according to the schedule of study assessments (Section 5.2):

- Serum Ig concentrations
  - **IgA**
  - **IgE**
  - IgM
- Serum complement levels
  - C3
  - C4
- Plasma complement levels
  - C3a
  - C5a
- Serum BAFF levels
- status (negative or confirmed positive) and changes Plasma in relative mass units for all scheduled assessments or titre for those confirmed positive
- Cytokines

### 12 ASSESSMENT OF SAFETY

### 12.1 Adverse events

### 12.1.1 Definitions

### 12.1.1.1 Adverse event

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

In order to ensure complete safety data collection, all AEs occurring during the study (ie, after the signing of the Informed Consent form), including any pretreatment and posttreatment periods required by the protocol, must be reported in the eCRF even if no IMP was taken but specific study procedures were conducted. This includes all AEs not present prior to the initial visit and all AEs that recurred or worsened after the initial visit.

Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a clinically significant manner as compared to the clinical profile known to the investigator from the subject's history or the Baseline Period.

Treatment-emergent AEs are defined as AEs starting after the time of first IMP administration up to and including 8 weeks after the final dose.

### 12.1.1.2 Serious adverse event

Once it is determined that a subject experienced an AE, the seriousness of the AE must be determined. An SAE must meet 1 or more of the following criteria:

- Death
- Life-threatening

(Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form)

- Significant or persistent disability/incapacity
- Congenital anomaly/birth defect (including that occurring in a fetus)
- Important medical event that, based upon appropriate medical judgment, may jeopardize the
  patient or subject and may require medical or surgical intervention to prevent 1 of the other
  outcomes listed in the definition of serious

(Important medical events may include, but are not limited to, potential Hy's Law [see Section 12.1.1.3], allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.)

• Initial inpatient hospitalization or prolongation of hospitalization

(A patient admitted to a clinic/hospital, even if he/she is released on the same day, meets the criteria for the initial inpatient hospitalization. An emergency room visit that results in admission to the clinic/hospital would also qualify for the initial inpatient hospitalization criteria. However, emergency room visits that do not result in admission to the clinic/hospital would not qualify for this criteria and, instead, should be evaluated for 1 of the other criteria in the definition of serious [eg, life-threatening adverse experience, important medical event]).

Hospitalizations for reasons not associated with the occurrence of an AE [eg, preplanned surgery or elective surgery for a pre-existing condition that has not worsened or manifested in an unusual or uncharacteristic manner] do not qualify for reporting. For example, if a subject has a condition recorded on his/her medical history and later has a preplanned surgery for this condition, it is not appropriate to record the surgery or hospitalization as an SAE, since there is no AE upon which to assess the serious criteria. Please note that, if the pre-existing condition has worsened or manifested in an unusual or uncharacteristic manner, this would then qualify as an AE and, if necessary, the seriousness of the event would need to be determined.)

# 12.1.1.2.1 Anticipated serious adverse events

Myasthenic crisis is anticipated to occur in the population studied in this protocol at some frequency that is independent of drug exposure.

This information does not change the investigator's obligation to report all SAEs (including Anticipated SAEs) as detailed in Section 12.1.2.3.

### 12.1.1.3 Adverse events of special interest

An AE of special interest is any AE that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a UCB product/compound.

Potential Hy's Law, defined as  $\ge 3x$ ULN ALT or AST with coexisting  $\ge 2x$ ULN total bilirubin in the absence of  $\ge 2x$ ULN ALP, with no alternative explanation for the biochemical abnormality, must ALWAYS be reported to UCB as an AE of special interest (ie, without waiting for any additional etiologic investigations to have been concluded). Follow-up information should then be reported if an alternative etiology is identified during investigation and monitoring of the subject.

### 12.1.1.4 Adverse events of interest

For UCB7665, AEs of interest that require immediate reporting to UCB are:

- Severe headache
- Moderate to severe diarrhea
- Moderate to severe abdominal pain
- Moderate to severe vomiting

### 12.1.1.5 Immediate reporting of adverse events

The following AEs must be reported immediately using the SAE Report Form according to the procedure in Section 12.1.2.3:

- SAE: AE that the investigator classifies as serious by the above definitions regardless of causality
- Suspected transmission of an infectious agent via a medicinal product
- AE of special interest (see Section 12.1.1.3)
- AE of interest (see Section 12.1.1.4)
- Confirmed LTBI, active TB, and NTMBI (see Section 12.3.1)

#### 12.1.2 Procedures for reporting and recording adverse events

valiations the reof The subject will be given the opportunity to report AEs spontaneously. A general prompt will "Did you notice anything unusual about your health (since your last visit)?"

Description of adverse and a second and adverse and a second a second and a second a second and a second a second and a second a second a second and a second a sec also be given at each study visit to detect AEs. For example:

### 12.1.2.1

When recording an AE, the investigator should use the overall diagnosis or syndrome using standard medical terminology, rather than recording individual symptoms or signs. The eCRF and source documents should be consistent. Any discrepancies between the subject's own words and the corresponding medical terminology should be clarified in the source documentation.

For recording an AE, Common Terminology Criteria for Adverse Events (CTCAE) will be used, and only if it is impossible to assess severity using CTCAE, then AE intensity will be used, using a scale of mild, moderate, or severe.

Details for completion of the AE eCRF (including judgment of relationship to IMP) are described in the eCRF Completion Guidelines.

#### Rule for repetition of an adverse event 12.1.2.2

An increase in the intensity of an AE should lead to the repetition of the AE being reported with:

- The outcome date of the first AE that is not related to the natural course of the disease being the same as the start date of the repeated AE, and the outcome of "worsening"
- The AE verbatim term being the same for the first and repeated AE, so that the repeated AE can be easily identified as the worsening of the first one

### Additional procedures for reporting serious adverse events 12.1.2.3

If an SAE is reported, UCB must be informed within 24 hours of receipt of this information by the site (see contact information for SAE reporting listed in the Serious Adverse Event Reporting section at the front of the protocol). The investigator must forward to UCB (or its representative) a duly completed "Investigator SAE Report Form for Development Drug" (SAE Report Form) provided by UCB, even if the data are incomplete, or if it is obvious that more data will be needed in order to draw any conclusions. Information recorded on this form will be entered into the global safety database.

An Investigator SAE Report Form will be provided to the investigator. The Investigator SAE Report Form must be completed in English.

It is important for the investigator, when completing the SAE Report Form, to include the assessment as to a causal relationship between the SAE and the IMP administration. This insight from the investigator is very important for UCB to consider in assessing the safety of the IMP and in determining whether the SAE requires reporting to the regulatory authorities in an expedited manner.

Additional information (eg, autopsy or laboratory reports) received by the investigator must be provided within 24 hours. All documents in the local language must be accompanied by a translation in English, or the relevant information included in the same document must be summarized in the Investigator SAE Report Form.

The investigator is specifically requested to collect and report to UCB (or its representative) any SAEs (even if the investigator is certain that they are in no way associated with the IMP), up to 30 days from the end of the study for each subject, and to also inform participating subjects of the need to inform the investigator of any SAE within this period. Serious AEs that the investigator thinks may be associated with the IMP must be reported to UCB regardless of the time between the event and the end of the study.

Upon receipt of the SAE Report Form, UCB will perform an assessment of expectedness of the reported SAE. The assessment of the expectedness of the SAE is based on the Investigator's Brochure.

# 12.1.3 Follow up of adverse events

An AE should be followed until it has resolved, has a stable sequelae, the investigator determines that it is no longer clinically significant, or the subject is lost to follow up. This follow-up requirement applies to AEs, SAEs, and AEs of special interest; further details regarding follow up of PDILI events is provided in Section 12.2.1.4.

If an AE is ongoing at the end of the study for a subject, follow up should be provided until resolution/stable level of sequelae is achieved, or until the investigator no longer deems that it is clinically significant, or until the subject is lost to follow up. If no follow up is provided, the investigator must provide a justification. The follow up will usually be continued for 8 weeks after the subject has discontinued his/her IMP.

Information on SAEs obtained after clinical database lock will be captured through the PS database without limitation of time.

# 12.1.4 Pregnancy

If an investigator is notified that a subject has become pregnant after the first intake of any IMP, the investigator must immediately notify UCB's PS department by providing the completed Pregnancy Report and Outcome form (for contact details see SAE reporting information at the beginning of this protocol). The subject should be withdrawn from the study as soon as pregnancy is known (by positive pregnancy test), and the following should be completed:

- The subject should return for a PEOT Visit.
- The subject should immediately stop the intake of the IMP or be down-titrated as instructed at the PEOT Visit.

The investigator must inform the subject of information currently known about potential risks and about available treatment alternatives.
The pregnancy will be documented on the Pregnancy Report and Outcome form provided to the investigator. The progression of the pregnancy and the eventual birth (if applicable) must be followed up using the Pregnancy Report and Outcome form in which the investigator has to report on the health of the mother and of the child. Every reasonable attempt should be made to follow the health of the child for 30 days after birth for any significant medical issues. In certain circumstances, UCB may request that follow up is continued for a period longer than 30 days. If the subject is lost to follow up and/or refuses to give information, written documentation of attempts to contact the subject needs to be provided by the investigator and filed at the site. UCB's PS department is the primary contact for any questions related to the data collection for the pregnancy, eventual birth, and follow up.

In cases where the partner of a male subject enrolled in a clinical study becomes preconsinvestigator or designee is asked to contact the subject to a Partner Pregnancy Consent form.

In cases where the partner of a male subject enrolled in a clinical study becomes pregnant, the investigator or designee is asked to contact the subject to request consent of the partner via the Partner Pregnancy Consent form that has been approved by the responsible IRB/IEC and should be available in the investigator site file. In case of questions about the consent process, the investigator may contact the UCB/CRO contract monitor for the study. The investigator will complete the Pregnancy Report and Outcome form and send it to UCB's PS department (for contact details see SAE reporting information at the beginning of this protocol) only after the partner has agreed that additional information can be captured and has provided the signed Partner Pregnancy Consent form. UCB's PS department is also the primary contact for any questions related to the data collection for the partner pregnancy, eventual birth, and follow up.

A pregnancy becomes an SAE in the following circumstances: miscarriage, abortion (elective or spontaneous), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report Form.

# 12.1.5 Suspected transmission of an infectious agent via a medicinal product

For the purposes of reporting, any suspected transmission of an infectious agent via a medicinal product should be considered as an SAE; such cases must be reported immediately, recorded in the AE module of the eCRF, and followed as any other SAE. Any organism, virus, or infectious particle (eg, prion protein transmitting transmissible spongiform encephalopathy), pathogenic or nonpathogenic, is considered an infectious agent.

## 12.1.6 Suicidality

At screening, the Investigator will query each subject if he/she has a lifetime history of suicide attempt (including an or suicidal ideation in the past 6 months. A full C-SSRS "Lifetime recent" assessment will be performed only when the subject has a positive response to this query. This scale will be assessed by trained study personnel. When suicide attempt or suicidal ideation is confirmed by a positive response (Yes) to either Question 4 or Question 5 of the C-SSRS, the subject must be excluded and immediately referred to a Mental Healthcare Professional.

At each clinical visit, the investigator must query the suicidal ideation since the last visit. A full C-SSRS "Since last visit" assessment will be performed only when the subject has a positive response to this query. When suicide attempt or suicidal ideation is confirmed by a positive

response (Yes) to either Ouestion 4 or Ouestion 5 of the C-SSRS, the subject must be withdrawn and immediately referred to a Mental Healthcare Professional. The details of C-SSRS will be provided in the Study Procedures Manual.

### 12.1.7 Overdose of investigational medicinal product

protocol and including overdose) should be nollowed as any other SAE or nonserious AE. These events are only considered AEs or SAEs if there are associated clinical signs and symptoms or if the act of taking the excess medicine itself is an AE or SAE (eg, suicide attempt).

12.1.8 Safety signal detection

An unblinded DMC will

which the safety of UCB7665 will be assessed. The safety variables to be used and the decision rules will be specified in the DMC charter. Further details of these interim analyses are given in Section 14.7.

Thus, selected data from this study will be reviewed periodically to detect as early as possible any safety concern(s) related to the IMP so that investigators, clinical study subjects, regulatory authorities, and IRBs/IECs will be informed appropriately and as early as possible.

The sponsor study physician or medically qualified designee/equivalent will conduct an ongoing review of SAEs and perform ongoing SAE reconciliations in collaboration with the PS representative.

As appropriate for the stage of development and accumulated experience with the IMP. medically qualified personnel at UCB may identify additional safety measures (eg. AEs, vital signs, laboratory or ECG results) for which data will be periodically reviewed during the course of the study.

### Hypersensitivity and adverse reactions 12.1.9

In the event of a severe infusion or anaphylactic reaction requiring corticosteroid and/or epinephrine therapy, the subject must permanently discontinue IMP and be managed as described in Section 18.8.

In case of occurrence of a hypersensitivity reaction (not determined by the investigator to be a minor local reaction at the infusion site, such as minimal itching) and depending upon its severity, appropriate countermeasures will immediately be taken by the investigator. The cytokine samples must be taken for infusion reactions.

If the investigator does not initially choose to discontinue the infusion of IMP and symptoms persist or escalate during continued infusion, the infusion should be stopped. In case of any severe infusion reaction(s), the infusion of IMP must be stopped immediately and appropriate treatment initiated, as necessary, at the discretion of the investigator and in accordance with the standard of care.

Moderate or severe anaphylactic reactions should be diagnosed using Sampson's Criteria (Sampson et al, 2006) as described in Section 18.9. In the event of an anaphylactic reaction the infusion must be discontinued immediately and appropriate emergency resuscitation measures implemented.

## 12.1.10 Management of severe headache

Severe headache is defined as severe pain limiting self-care activities of daily living (ADL) or new/prolonged hospitalization for management of headache or life-threatening consequences requiring urgent medical intervention. Self-care ADL refers to bathing, dressing and undressing, feeding self, using the toilet, and taking medications. Treatment of headache will be provided as clinically indicated according to the local guidelines.

Subjects experiencing severe headache will complete the Headache Questionnaire and will complete the questionnaire daily until resolution (ie, if headache becomes moderate or mild, normal collection of AEs should apply); this assessment will be followed by a neurological assessment (including fundoscopy). Further workup will be performed (if indicated) at the discretion of the investigator and may include, eg, a computed tomography scan, magnetic resonance imaging and/or a lumbar puncture for cerebral spinal fluid collection. In addition, assessment of exploratory safety biomarkers should be performed for subjects experiencing severe headache. These investigations will be performed in order to further understand the mechanism of headache in these subjects.

Details of neurological examination to be performed are provided in Section 12.3.6. The Headache Questionnaire is available in Section 18.10.

## 12.1.11 Management of moderate or severe diarrhea

Moderate or severe diarrhea is defined as an increase of  $\geq 4$  stools per day over Baseline or incontinence due to urgency of diarrhea or new/prolonged hospitalization for management of diarrhea or limiting self-care ADL or life-threatening consequences requiring urgent medical intervention.

Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally. In addition, collection of blood samples for assessment of exploratory safety biomarkers is required for subjects with moderate to severe GI disturbances including diarrhea.

Treatment of diarrhea will be provided as clinically indicated according to the local guidelines.

## 12.2 Laboratory measurements

Blood and urine specimens for routine assay of hematology, clinical chemistry, and urinalysis testing, and as well as serum and urine pregnancy testing, will be performed according to the schedule of assessments (Section 5.2) to monitor the safety of subjects. All clinical chemistry, hematology, and urinalysis parameters will be assessed by the designated central laboratory with the exception the urine pregnancy test prior to each dose. Specific details regarding the handling and processing of the serum chemistry, hematology, and urinalysis samples are provided in the study laboratory manuals.

Table 12.2 lists the laboratory parameters that will be measured.

### Table 12.2: Safety laboratory measurements

| Hematology | Chemistry | Urinalysis | Pregnancy test |
|---|---|---|---|
| Hematocrit | Electrolytes (calcium, | Albumin | Urine HCG |
| Hemoglobin | phosphate, sodium, potassium, chloride, | Protein | Serum HCG <sup>a</sup> |
| Platelet count | and magnesium) | Nitrite | |
| RBC count | ALP | Glucose | il |
| WBC count | AST | рН | or |
| (including differential) | ALT | Leukocytes | *ensions or varia |
| HbA1c <sup>b</sup> | GGT | Blood | et e |
| | Total and direct | Bilirubin | art |
| Serology <sup>c</sup> | bilirubin | Urobilinogen | 6 |
| HBsAg | LDH | Ketone | |
| HCV Ab | Total cholesterol | Creatinine | |
| HIV (anti-HIV1 or | LDL - cholesterol | 0, 286 | |
| anti-HIV2 antibodies) Tuberculosis <sup>d</sup> | HDL – cholesterol,<br>triglycerides | ortzatio. | |
| | Amylase | Jike | |
| Exploratory Safety<br>Biomarkers <sup>e</sup> | Creatine kinase | | |
| | Creatinine | | |
| | Total protein | | |
| | Albumin | | |
| | alpha- and beta–<br>globulins | | |
| | Urea-N | | |
| * C. | Procalcitonin | | |
| Well, | hsCRP | | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; GGT=gamma glutamyltransferase; HbA1c=hemoglobin A1c; HBsAG=hepatitis B surface antigen; HCG=human chorionic gonadotropin; HCV Ab=hepatitis C virus antibody; HDL=high density lipoprotein; HIV=human immunodeficiency virus; hsCRP=high-sensitivity C-reactive protein; LDH=lactate dehydrogenase; LDL=low density lipoprotein; RBC=red blood cell; B; WBC=white blood cell

- <sup>a</sup> Serum pregnancy testing is only performed at Visit 1 and, in the event of a positive pregnancy test, to confirm the results of a urine test
- b HbA1c is performed at Screening only
- <sup>c</sup> This serology performed at Screening only
- <sup>d</sup> Interferon-gamma release assay by central laboratory.
- Or variations thereof May include but not limited to the following biomarkers listed below. Samples collected for exploratory safety biomarkers at Baseline (Visit 2) and 4 hours post dosing (Visit 2) for all subjects and during follow up only in subjects with severe headache and/or moderate to severe GI disturbances. The Baseline samples will only be analysed in case the subject experienced a severe headache and/or moderate to severe GI disturbance.

### 12.2.1 **Evaluation of PDILI**

The PDILI IMP discontinuation criteria for this study are provided in Section 6.4.1, with the accompanying required follow-up investigation and monitoring detailed below. All PDILI events must be reported as an AE and reported to the study site and sponsor within 24 hours of learning of their occurrence. Any PDILI event that meets the criterion for potential Hy's Law must be reported as an AE of special interest (see Section 12.1.1.3), and, if applicable, also reported as an SAE (see Section 12.1.1.2).

Evaluation of PDILI consists of the diagnostic testing and continued monitoring included in Table 12.3 (specific tests dependent on laboratory results and corresponding symptoms) and consultation with a local hepatologist (if applicable; discussed in Section 12.2.1.1). The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist. Additional investigation and monitoring may be required and adapted based on the diagnosis after the cause of the liver injury/abnormality is confirmed (details in Section 12.2.1.4).

The results of all monitoring, including laboratory testing and other testing, should be made available to the study site and sponsor.

All initial tests resulting in abnormal hepatic laboratory values need to be repeated, but appropriate medical action must not be delayed waiting for the repeat result.

If tests are done locally for more rapid results, a concurrent sample should also be sent to the central laboratory whenever possible. Medical care decisions are to be made initially using the most rapidly available results and a conservative approach must be taken if the results from the 2 laboratory tests are significantly different. Data from the local and central laboratory are to be recorded on the applicable eCRF pages.

When IMP is discontinued, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued. In these cases, the investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative.

When IMP is stopped due to PDILI (as described in Section 6.4.1), IMP must be permanently discontinued unless a subsequent alternative diagnosis fully explains the hepatic findings. If a subsequent alternative diagnosis fully explains the hepatic findings, and the requirements provided in Section 12.2.1.2.1 are met, rechallenge with IMP may be appropriate.

RELEASE THE BOLING TO THE BOLING

Table 12.3: Required investigations and follow up for PDILI

| | • | ed investigation | ns and follow up fo | r PDILI | | idion |
|---|---|---|---|---|---|---|
| Laborator | 1 | | Immediate | T | Follow up | , Jak |
| ALT or<br>AST | Total<br>bilirubin | Symptoms <sup>a</sup> of hepatitis or hypersensitivity | Consultation requirements | Actions | Testing | Evaluation |
| ≥3xULN | ≥2xULN <sup>b</sup> | NA | Hepatology consult. <sup>c</sup> Medical monitor must be notified within 24 hours | Immediate, permanent IMP discontinuation. | Essential: Must have repeat liver chemistry values and additional | Monitoring of liver chemistry values at least twice per week until values normalize, stabilize, or return to within Baseline |
| ≥3xULN | NA | Yes | (eg, by laboratory alert) and subject discussed with medical monitor ASAP. | Immediate,<br>temporary or<br>permanent, IMP<br>discontinuation | testing completed<br>ASAP (see<br>Section 12.2.1.3);<br>recommended to<br>occur at the site<br>with HCP. | values. <sup>d</sup> |
| ≥3xULN<br>(and ≥2x<br>Baseline)<br>and<br><5xULN | <2xULN | No | Discussion with medical monitor required if the criterion that allows for IMP continuation is met. | Further investigation – immediate IMP discontinuation not required (see Section 12.2.1.2). | Not required<br>unless otherwise<br>medically<br>indicated (at<br>discretion of<br>investigator). | |
| ≥5xULN<br>(and ≥2x<br>Baseline) | <2xULN | No No | Discussion with medical monitor required. Hepatology consult required if ALT or AST ≥8xULN | Immediate, permanent IMP discontinuation. | Essential: Every attempt must be made to have repeat liver chemistry values and additional testing completed within 48 hours at the site with HCP (see Section 12.2.1.3). | Monitoring of liver chemistry values at least twice per week until values normalize, stabilize, or return to within Baseline values. <sup>d</sup> |

## Table 12.3: Required investigations and follow up for PDILI

| Laboratory | value | | Immediate | | Follow up | Marilo |
|---|---|---|---|---|---|---|
| ALT or<br>AST | Total<br>bilirubin | Symptoms <sup>a</sup> of<br>hepatitis or<br>hypersensitivity | Consultation requirements | Actions | Testing | Evaluation |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; ASAP=as soon as possible; AST=aspartate aminotransferase; HCP=healthcare practitioner; IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug-induced liver injury; ULN=upper limit of normal

<sup>&</sup>lt;sup>a</sup> Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

<sup>&</sup>lt;sup>b</sup> If the subject also has ≥2xULN ALP, the possibility of an indication of biliary obstruction should be discussed with the medical monitor.

<sup>&</sup>lt;sup>c</sup> Details provided in Section 12.2.1.1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist.

stroentere.

JCB responsible physician

responsible physician

responsible physician

Agriculture physician

responsible physician

respo d Unless an alternative monitoring schedule is agreed by the investigator and UCB responsible physician. Determination of stabilization is at the discretion of the investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

### 12.2.1.1 Consultation with medical monitor and local hepatologist

Potential drug-induced liver injury events require notification of the medical monitor within 24 hours (eg. by laboratory alert), and the subject must be discussed with the medical monitor as Ins or variations thereof soon as possible. If required, the subject must also be discussed with the local hepatologist or gastroenterologist. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist. If determined necessary, this discussion should be followed by a full hepatology assessment (see Section 12.2.1.3) and SAE report (if applicable).

### Immediate action: determination of IMP discontinuation 12.2.1.2

All PDILI events require immediate action, testing, and monitoring.

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate and permanent discontinuation (see Section 6.4.1 and Table 12.3 for details).

When IMP is discontinued, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued. The investigator should also consider dose reduction for medically necessary concomitant medication and consider changing any medically required concomitant medication known to be hepatotoxic to a suitable alternative.

### 12.2.1.2.1 IMP restart/rechallenge (if applicable)

Rechallenge with a substance potentially causing drug-induced liver injury is dangerous, may be fatal, and must not occur.

Subjects who are immediately discontinued from IMP due to having met certain criteria for PDILI (as described in Section 6.4.1 and Table 12.3), but for whom an alternative diagnosis is confirmed, can rarely restart IMP. Rechallenge with IMP can occur only if ALL of the following requirements are met:

- The results of additional testing and monitoring described in Section 12.2.1.3 and Section 12.2.1.4 confirm a nondrug-related cause for the abnormal hepatic laboratory parameters and any associated symptoms (ie, a subsequent alternative diagnosis fully explains the hepatic findings).
- No alternative treatment options are available to the subject.
- The subject has shown clear therapeutic benefit from the IMP.
- Subject's ALT or AST elevations do not exceed >3xULN.
- Subject's total bilirubin is <1.5xULN.
- Subject has no signs or symptoms of hypersensitivity.
- The rechallenge is approved by the UCB responsible physician, DMC, and a hepatologist. The hepatologist must be external to UCB but may be a member of the DMC. It is recommended that the hepatologist be a local hepatology expert or the hepatologist treating the subject.
- Subject agrees to the investigator-recommended monitoring plan.

15 Sep 2017

MG0002

### 12.2.1.3 Testing: identification/exclusion of alternative etiology

The measurements and additional information required for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP are detailed in All blood samples should be stored, if possible. If tests are done locally for more rapid results, a concurrent sample must also be sent to the central laboratory.

Table 12.4: PDILI laborate. Table 12.4 (laboratory measurements) and Table 12.5 (additional information). Results of the

| Table 12.4: | PDILI laboratory measurements |
|---|---|
| Virology- | Hepatitis A IgM antibody |
| related | HBsAg |
| | Hepatitis E IgM antibody |
| | HBcAb-IgM |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophile antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| | Anti-smooth muscle antibody (qualitative and quantitative) |
| | Type 1 anti-liver kidney microsomal antibodies (qualitative and quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen |
| Chemistry | Amylase Survey |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| Additional | Prothrombin time/INR <sup>a</sup> |
| anno | Serum pregnancy test |
| ant Co | PK sample |

ALT=alanine aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody-IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal

The following addition information listed in Table 12.5 is to be collected:

### Table 12.5: PDILI information to be collected

### New or updated information

Concomitant prescription and over-the-counter medications (eg, acetaminophen, herbal remedies, vitamins); dosages and dates should be included

Pertinent medical history, including the following:

- History of liver disease (eg, autoimmune hepatitis, nonalcoholic steatohepatitis or other "fatty liver disease")
- Adverse reactions to drugs
- Allergies
- Relevant family history or inheritable disorders (eg, Gilbert's syndrome, alpha-1 antitrypsin deficiency)
- Recent travel
- Progression of malignancy involving the liver (Note: Metastatic disease to the liver, by itself, should not be used as an explanation for significant AST and/or ALT elevations)

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity (eg, fatigue, nausea, vomiting, right upper quadrant pain or tenderness, decreased appetite, abdominal pain, jaundice, fever, or rash)

Recent clinically significant hypotension or hypoxemia with compromised cardiopulmonary function

Alcohol and illicit drug use

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

Any postmortem/pathology reports

ALT=alanine aminotransferase; AST=aspartate aminotransferase; PDILI=potential drug-induced liver injury

## 12.2.1.4 Follow-up evaluation

Potential drug-induced liver injury events require follow-up monitoring as described in Table 123. Monitoring should continue until liver chemistry values normalize, stabilize, or return to Baseline. Determination of stabilization is at the discretion of the investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

<sup>&</sup>lt;sup>a</sup> Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

### 12.3 Other safety measurements

### 12.3.1 Assessment and management of TB and TB risk factors

With the currently available data, TB is not considered as an important potential or identified risk Appropriate rigorous precautions are being taken within this protocol to monitor the risk of TB infection in this study (see Section 6.2.3 [Exclusion Criterion 32] and Section 6.4 [Withdrawall Criteria 1]). Following are the key considerations of these procedures:

TB Tests at Screening

IGRA and TB questionnaire are required as indicated in Schedule of Assessments (Table 5.1).

- TB screening is mandatory both before study entry and during the conduct of the study. The preferred screening test is IGRA performed at a Central Laboratory
  - The IGRA result must be negative for subjects to enroll in this study
  - Subjects who test positive for IGRA test should be excluded from the study and referred for appropriate medical evaluation according to the local medical practice guidelines.
  - If the result of the IGRA test is indeterminate, the particular IGRA test previously performed may be repeated once; if positive or indeterminate on retest, the subject must not be randomized to study drug and, if already randomized, must undergo appropriate study specified withdrawal procedures. The retest must be done during the protocol-defined Screening Period.
- In addition to IGRA test, subjects will be evaluated for signs and symptoms of latent or active TB infection and for risk factors of exposure to TB, using the TB questionnaire, at Screening. See the 'TB signs and symptoms questionnaire' section for further instructions on using the questionnaire. Subjects with known TB, at a high risk of acquiring TB or with LTBI should be excluded from this study as described in Exclusion Criteria.

## Monitoring for TB during the study

Subjects will be monitored for signs/symptoms of TB using routine pharmacovigilance measures for Adverse Events. Subjects reporting AEs related to signs/symptoms of TB will be evaluated for LTBI and active TB according to the local medical practice guidelines.

Subjects with confirmed LTBI or active TB or NTMBI will be immediately withdrawn from the study as described in Withdrawal Criteria. Confirmed LTBI, active TB, and NTMBI must be reported to the Sponsor immediately regardless of seriousness using the SAE Report Form. Additional information received by the Investigator should be provided to the Sponsor within 24 hours of awareness.

Once withdrawn from study treatment, subjects should return for the PEOT, complete all early withdrawal assessments, and complete the follow-up visits.

### TB tests at Final/PEOT Visit

Subjects will be evaluated for signs and symptoms of latent or active TB infection and for risk factors of exposure to TB, using the TB questionnaire, at the Final/PEOT Visit. See the 'TB signs and symptoms questionnaire' section for further instructions on using the questionnaire.

### Signs and symptoms of TB

The Investigator should consider all potential sites of infection when assessing for TB during the physical examination, and other evaluations, and based on the subject's history.

Common symptoms with which the subject may present with include cough, blood in sputum, night sweats, lymphadenitis, joint pain/swelling, spinal deformity, headache/confusion, abdominal pain mimicking inflammatory bowel disease, frequent or painful urination, scrotal mass in men and pelvic inflammatory disease in women as well as other symptoms, or nonspecific symptoms. This is not an exhaustive list and unusual presentations should always be considered.

## TB signs and symptoms questionnaire

The questionnaire "Evaluation of signs and symptoms of tuberculosis" should be used as a source document. The questionnaire will assist with the identification of subjects who may require therapy for TB. A subject who answers "Yes" to the question

at Screening is excluded. A "Yes" response to any of the other questions within the questionnaire at Screening should trigger further careful assessment to determine if subject has latent or active TB (see Section 6.2.3 [Exclusion Critetion 32]). A "Yes" response to any of the questions at the end of the study should trigger further assessments as per local medical guidelines to determine if the subject has either LTBI or active TB infection.

### LTBI, active TB or other NMTB identified during study

During the study, subjects who develop evidence of LTBI or active TB or NMTBI must immediately stop further administration of study drug and will be referred to an appropriate medical specialist for further evaluation.

Confirmed LTBI or active TB or NTMBI must be reported to the Sponsor immediately as described above.

### 12.3.2 Pregnancy testing

Pregnancy testing will consist of a serum test at Screening Visit (Visit 1) and urine tests at all other visits, as indicated in the schedule of study assessments (Table 5.1). The Screening Visit serum pregnancy test results must be negative and should be confirmed by a negative urine pregnancy test prior to first dose of IMP. The urine pregnancy test will be performed locally. A negative urine pregnancy test result should be obtained prior to each dose of IMP. A positive urine pregnancy test must be confirmed using a serum pregnancy test. Pregnancy tests should be administered to all female subjects of childbearing potential, regardless of their use of birth control.

### 12.3.3 Vital signs

Vital signs will be measured at all visits as indicated in the schedule of study assessments (Table 5.1).

Vital signs to be assessed are as follows:

- Pulse rate
- Systolic/diastolic BP
- Temperature (oral preferred, ear or axillary allowed)
- Respiratory rate

Subjects will be sitting for at least 5 minutes prior and during the measurement of BP, PR, and respiration rate. On dosing days, vital signs will be measured prior to IMP administration, once during the infusion (at the halfway time point), at the end of infusion, 2 hours after end of infusion, and 4 hours after end of infusion. At nondosing visits, vital signs need only be taken once during the visit.

## 12.3.4 Body weight and height

The subject's body weight (without shoes) will be determined at Screening (Visit 1), Visit 9, and at the FV (Visit 20). Height will be measured at Screening (Visit 1) only.

## 12.3.5 Physical examination

Physical examination (full or brief) will be performed at visits as specified in the schedule of study assessments (Table 5.1) and findings will be recorded in the eCRF.

Clinically important abnormal changes in subsequent physical examinations will be recorded as AEs. Physical examinations must be documented in source documentation.

## 12.3.5.1 Full physical examination

The following body systems will be examined as a part of the full physical examination:

- General appearance
- Ear, nose, and throat
- Eyes
- Hair and skin
- Respiratory
- Cardiovascular
- GI
- Musculoskeletal
- Hepatic
- Neurological (including limb reflexes)
- Mental status

### 12.3.5.2 Brief physical examination

The following body systems will be examined as a part of the brief physical examination at the Jextensions of variations thereof visits outlined in the schedule of assessments (Table 5.1):

- General appearance
- Ear, nose, and throat
- Eyes
- Skin
- Respiratory
- GI
- Neurological (focused assessment of sensitivity and power)

### 12.3.6 **Neurological examination**

In addition to the Screening and FV, a full neurological examination should be performed for any subject who experiences severe headache (see Section 12.1.10). Neurological examination (full or brief) will be performed at visits as specified in the schedule of study assessments (Table 5.1) and findings will be recorded in the eCRF.

A full neurological assessment will include: 1) General appearance, including posture, motor activity and meningeal signs and, if indicated, following assessments to be done; 2) Cranial nerves examination; 3) Motor system examination, including muscle tone and power and sensory system examination – light touch; 4) Reflexes, including deep tendon reflexes; 5) Coordination, gait (if possible) and; 6) Fundoscopy.

A brief neurological assessment will include a selected assessment of the following: cognition, general reflexes, muscle strength, and coordination/cerebellar function.

### 12.3.7 12-lead ECG

A standard 12-lead ECG will be performed at visits as specified in the schedule of study assessments (Table 5.1).

Care should be taken to assure proper lead placement and quality ECG recordings. Subjects should rest in a supine position in a controlled, calm environment for at least 15 minutes prior to the recording and should be motionless during the recording. The ECG will be performed in triplicate prior to blood collection for assessment of laboratory parameters.

The ECGs will be read by a central reader. The PR, RR, QRS, QT, and corrected QT (QTc) intervals and heart rate will be assessed.

For the QTc, the following correction formula will be applied:

Fridericia's correction:  $QTc = QT/RR^{0.33}$ 

The investigator may consult with the cardiologist at the central ECG laboratory to confirm the presence of a clinically significant ECG abnormality. It remains the responsibility of the investigator to decide whether an ECG finding is of clinical significance on the basis of the

complete clinical picture and whether this finding influences the subject's participation in the study.

### 13 STUDY MANAGEMENT AND ADMINISTRATION

### 13.1 Adherence to protocol

The investigator should not deviate from the protocol. However, the investigator should take any measure necessary in deviation from or not defined by the protocol in order to protect clinical study subjects from any immediate hazard to their health and safety. In this case, this action should be taken immediately, without prior notification of the regulatory authority, IRB/IEC, or sponsor.

After implementation of such measure, the investigator must notify the CPM of the sponsor within 24 hours and follow any local regulatory requirements.

## 13.2 Monitoring

UCB (or designee) will monitor the study to meet the sponsor's monitoring SOPs, ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate. Monitoring of the study may be delegated by UCB to a CRO or a contract monitor.

The investigator and his/her staff are expected to cooperate with UCB (or designee) and to be available during the monitoring visits to answer questions sufficiently and to provide any missing information. The investigator(s)/institution(s) will permit direct access to source data/documents for study-related monitoring, audits, IRB/IEC review, and regulatory inspection(s).

The investigator will allow UCB (or designee) to periodically review all eCRFs and corresponding source documents (eg, clinic/hospital and laboratory records for each study participant). Monitoring visits will provide UCB (or designee) with the opportunity to evaluate the progress of the study, verify the accuracy and completeness of eCRFs, ensure that all protocol requirements, applicable authorities' regulations, and investigator's obligations are being fulfilled, and resolve any inconsistencies in the study records.

### 13.2.1 Definition of source data

All source documents must be accurate, clear, unambiguous, permanent, and capable of being audited. They should be made using some permanent form of recording (ink, typing, printing, optical disc). They should not be obscured by correction fluid or have temporary attachments (such as removable self-stick notes). Photocopies and /or printouts of eCRFs are not considered acceptable source documents.

Source documents are original records in which raw data are first recorded. These may include clinic/hospital/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records, ECG or other printouts, completed scales, or quality of life questionnaires, for example. Source documents should be kept in a secure, limited access area.

The following data will be recorded directly in the eCRF and will not appear in a separate source document as defined above.

Source documents that are computer generated and stored electronically must be printed for review by the monitor (eg, ECG reports). Once printed, these copies should be signed and dated by the investigator and become a permanent part of the subject's source documents. The investigator will facilitate the process for enabling the monitor to compare the content of the printout and the data stored in the computer to ensure all data are consistent.

Electronic data records, such as Holter monitor records or electroencephalogram records, must be saved and stored as instructed by UCB (or designee).

### 13.2.2 Source data verification

Source data verification ensures accuracy and credibility of the data obtained. During monitoring visits, reported data are reviewed with regard to being accurate, complete, and verifiable from source documents (eg, subject files, recordings from automated instruments, tracings [ECG], x-ray films, laboratory notes). All data reported on the eCRF should be supported by source documents, unless otherwise specified in Section 13.2.1.

## 13.3 Data handling

## 13.3.1 Case Report Form completion

The investigator is responsible for prompt reporting of accurate, complete, and legible data in the eCRFs and in all required reports.

Any change or correction to the eCRF after saving must be accompanied by a reason for the change.

Corrections made after the investigator's review and approval (by means of a password/electronic signature) will be reapproved by the investigator.

The investigator should maintain a list of personnel authorized to enter data into the eCRF.

Detailed instructions will be provided in the eCRF Completion Guidelines.

### 13.3.2 Database entry and reconciliation

Case Report forms/external electronic data will be entered/loaded into a validated electronic database using a clinical data management system (CDMS). Computerized data cleaning checks will be used in addition to manual review to check for discrepancies and to ensure consistency of the data. The data are entered into the eCRFs once by the designated site personnel and are subsequently verified.

An electronic audit trail system will be maintained within the CDMS to track all data changes in the database once the data have been saved initially into the system or electronically loaded. Regular backups of the electronic data will be performed.

## 13.3.3 Subject Screening and Enrollment log/Subject Identification Code list

The subject's screening and enrollment will be recorded in the Subject Screening and Enrollment Log.

The investigator will keep a Subject Identification Code list. This list remains with the investigator and is used for unambiguous identification of each subject.

The subject's consent and enrollment in the study must be recorded in the subject's medical record. These data should identify the study and document the dates of the subject's participation.

If the study is prematurely terminated or suspended, UCB (or its representative) will inform the investigators/institutions and the regulatory authority(ies) of the termination or suspension and the requirement(s). The IRB/IEC should also be informed and applicable regulators. unused IMP and other material in accordance with UCB procedures for the study.

### 13.5 **Archiving and data retention**

The investigator will maintain adequate records for the study, including eCRFs, medical records, laboratory results, informed consent documents, drug dispensing and disposition records, safety reports, information regarding participants who discontinued, and other pertinent data.

All essential documents are to be retained by the investigator until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or at least 2 years have elapsed since the formal discontinuation of clinical development of the IMP. These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or by an agreement with UCB (CPMP/ICH/135/95.2002 [Section 4.9.5]). The investigator will contact UCB for authorization prior to the destruction of any study records or in the event of accidental loss or destruction of any study records. The investigator will also notify UCB should he/she relocate or move the study-related files to a location other than that specified in the sponsor's trial master file.

### Audit and inspection 13.6

The investigator will permit study-related audits mandated by UCB, after reasonable notice, and inspections by domestic or foreign regulatory authorities.

The main purposes of an audit or inspection are to confirm that the rights and well-being of the subjects enrolled have been protected, that enrolled subjects (ie, signing consent and undergoing study procedures) are appropriate for the study, and that all data relevant for the evaluation of the IMP have been processed and reported in compliance with the planned arrangements, the protocol, investigational site, and IRB/IEC SOPs, ICH-GCP, and applicable regulatory requirements.

The investigator will provide direct access to all study documents, source records, and source data. If an inspection by a regulatory authority is announced, the investigator will immediately inform UCB (or designee).

### **Good Clinical Practice** 13.7

Noncompliance with the protocol, ICH-GCP, or local regulatory requirements by the investigator, institution, institution staff, or designees of the sponsor will lead to prompt action Enrolled Set:

The Enrolled Set (ES) will consist of all subjects who have given informed consent.

Randomized Set:

The Randomized Set (RS) will consist of all subjects randomized:

andomization visit.

Safety Set:

The Safety Set (CS)

The Safety Set (SS) will consist of all subjects in the RS, who have received at least 1 dose of IMP.

Safety variables will be analyzed using the SS.

It is expected that subjects will receive treatment as randomized and hence safety analyses will be based on the randomized treatment group. However, if after unblinding it is determined that a subject has received the incorrect treatment based on the randomization schedule, then for safety analyses the subject will be allocated to the actual treatment they received in the respective Dosing Period.

### Full Analysis Set:

The Full Analysis Set (FAS) will consist of all subjects in the SS, who have a Baseline and least 1 post-Baseline QMG measurement during Dosing Period 1 (up to and including Visit 9, ie, Day 29).

The FAS is the primary analysis set for efficacy analyses. As for the SS, in the case of mistreatment, subjects will be primarily analyzed as treated. However, if applicable, sensitivity analysis will also be performed according to the randomized treatment group.

### Per-Protocol Set:

The Per-Protocol Set (PPS) is a subset of the FAS, consisting of those subjects who had no important protocol deviations affecting the primary efficacy variable, as confirmed during a pre-analysis data review meeting conducted prior to study unblinding. Post-Baseline deviations will not necessarily lead to total exclusion of a subject from the PPS but may lead to exclusion of specific data.

Analysis of the primary efficacy variable will be repeated using the PPS.

### Pharmacokinetic Per-Protocol Set:

The PK-PPS is a subset of the FAS, consisting of those subjects who had no important protocol deviations affecting the plasma concentration of UCB7665.

General statistical considerations

All analyses will be performed using SAS® version 9.3 or later (SAS Institute, Cary, NC, USA). Continuous variables will be summarized by visit (where applicable) with the statistics including the number of subjects (n), mean, standard deviation (SD), median, minimum Categorical variables will be summarized by visit (where applicable). The Treatment of the statistics including the summarized by visit (where applicable) with the statistics including the number of subjects (n), mean, standard deviation (SD), median, minimum Categorical variables will be summarized by visit (where applicable).

The Treatment Groups for Dosing Period 1 will be as follows:

- Placebo
- UCB7665 7mg/kg

For Dosing Period 2 and the Observation Period the following Treatment Groups will be considered for analysis:

- Placebo UCB7665 7mg/kg
- Placebo UCB7665 4mg/kg
- UCB7665 7mg/kg UCB7665 7mg/kg
- UCB7665 7mg/kg UCB7665 4mg/kg

These Treatment Groups will be used for all safety and efficacy analyses.

Unless stated otherwise, all statistical tests will be 1-sided and conducted at 0.05 alpha levels (due to the character of the study no alpha adjustment for multiplicity will be done). For Dosing Period 2, only descriptive analyses will be performed.

Data listings containing all documented data and all calculated data will be generated.

Baseline will be the last non-missing data collected prior to the first dose of IMP in Dosing Period 1, and measurement-specific Baseline values will be defined in the SAP.

### Planned efficacy analyses 14.3

For all efficacy analyses the Treatment Groups used for analysis during Dosing Period 1 and during Dosing Period 2/Observation Period will be as defined in Section 14.2. Efficacy endpoints will be analyzed using descriptive statistics for data obtained during Treatment Period 2 and Observation Period. Further details will be provided in SAP.

### **6014.3.1** Analysis of the primary efficacy variable

The primary efficacy variable is the change from Baseline in QMG score to Visit 9 (Day 29), prior to the first infusion of IMP in Dosing Period 2.

A 1-sided hypothesis test will be performed to test the primary hypothesis of superiority of UCB7665 7mg/kg vs placebo at Visit 9. The null hypothesis is that there is no difference in the change from Baseline between Treatment Groups. The alternative hypothesis is that the mean change from Baseline in QMG score is smaller in the UCB7665 7mg/kg group than the placebo group.

The primary analysis of the primary variable will be based on a mixed model repeated measures (MMRM) analysis of covariance (ANCOVA) that includes terms for treatment group, week, the Baseline QMG score, and the interaction between treatment group and week. The model will define patient as a random effect and utilize an unstructured covariance pattern.

Least Squares (LS) Means for changes from Baseline at Visit 9 for each treatment group will be presented together with LS mean differences (UCB7665 - 7mg/kg vs placebo) and 1-sided 95% confidence interval (CI).

For subjects who prematurely withdraw for any reason before Visit 9 (Day 29), data collected during the PEOT Visit will be used to impute QMG scores at the next consecutive visit.

Different sensitivity analyses to evaluate the effect of missing observations on the primary analysis findings will be done. The first sensitivity analysis will be performed in the same way as the primary analysis for the PPS. A further analysis will utilize the Last Observation Carried Forward (LOCF) approach; missing values will be replaced by the last observed post-Baseline value of the variable and the analysis will be performed on the resulting dataset.

## 14.3.2 Other efficacy analyses

The secondary variables and change from Baseline in QMG score, MG-Composite score, MGADL score, MGII score, muscle weakness severity and fatigability scale score and fatigue scale score, at each assessed post-Randomization Visit (during Dosing Period 1 including Visit 9) will also be analyzed utilizing the MMRM approach similarly to the change from Baseline in QMG for the FAS as described in Section 14.3.1.

QMG, MG-Composite, and MGADL responder rates at each assessed post-Randomization Visit (during Dosing Period 1) will be compared between the 2 Treatment Groups utilizing Fisher's exact test.

The percentage of subjects with each MGFA classification at each scheduled assessment during Treatment and Observation Periods will be calculated.

Psychometric analyses of the newly developed measures MG muscle weakness severity and fatigability and fatigue scales will be performed blinded from treatment arms. The association between PROs and clinical variables will also be explored, as well as the association between the various PROs. A psychometric analysis of the MG muscle weakness severity and fatigability scale and fatigue scale using Rasch analysis will be performed, but reported separately from the CSR.

Changes in MCD of the IPI, and normal fiber pairs in jitter (SFEMG) will be summarized using descriptive statistics, by treatment group and time point, including changes from Baseline. A reduction in MCD of  $\geq 9\mu s$  in jitter (SFEMG) studies will also be summarized using descriptive statistics, by treatment group and time point, including changes from Baseline.

## 14.4 Planned other and exploratory analyses

### 14.4.1 Safety analyses

For all safety analyses the Treatment Groups used for analysis during Dosing Period 1 and during Dosing Period 2/Observation Period will be as defined in Section 14.2 and as described in the SAP.

The absolute and relative frequencies for subjects with a given TEAE with respect to the preferred term according to the latest available version of the Medical Dictionary for Regulatory Activities, as well as the absolute frequencies of the individual TEAEs that have occurred, will be determined within each system organ class. Additional tables will summarize TEAEs by maximum intensity and causal relationship with IMP, as judged by the investigator. Adverse events will be categorized by severity according to the CTCAE Version 4.03 grading. In case the CTCAE grading is not available, the intensity (mild/moderate/severe) will be utilized. For the purpose of the tabulations CTCAE grades will be aligned with the intensity classifications (mild/moderate/severe) to enable pooling of the AEs in the summaries. The TEAEs leading to discontinuation of IMP and treatment-emergent SAEs will also be summarized. The action taken, time of onset relative to dosing, and duration of each AE will be listed only.

Adverse events will be assigned to a Dosing Period based on the start date of the event relative to the first dose of IMP received in the respective period.

For the continuous laboratory variables, the values and changes from Baseline will be summarized at each time point. For categorized values according to the reference range, shift tables from Baseline to each post-Baseline time point will be presented for selected variables to be defined in the SAP. Values outside the reference range will be flagged in the data listings.

Exploratory safety biomarkers will be summarized by treatment group and visit using descriptive statistics.

Normal vs abnormal findings with regard to the various ECG parameters and the overall ECG will be analyzed as required. The focus of the 12-lead ECG analysis will be the identification of outliers and of any trends for changes following administration of UCB7665 with respect to QT/QTc. Descriptive statistics will be presented for ECG value and changes from Baseline over time based on the mean of the triplicate assessments at each time point.

Descriptive statistics will be reported for all vital sign measurements (including pulse rate, systolic/diastolic BP, temperature, and respiratory rate). Measured values and changes from Baseline will be summarized by treatment group.

Physical and neurological examination findings and the results of any pregnancy testing will be presented in listings only.

## 14.4.2 Pharmacokinetic analysis

The PK variable is the plasma concentration of UCB7665. Pharmacokinetic parameters such as C<sub>max</sub> and area under the curve will not be derived (eg, by non-compartmental analysis) due to the limited sampling performed at each visit.

Individual concentrations of UCB7665 will be listed and summarized at each scheduled time point. Descriptive statistics of concentrations will be calculated only if at least two thirds of the individual data points are quantifiable (≥lower limit of quantification [LLOQ]). Summaries will

include the number of available observations, mean, median, SD, minimum, maximum, geometric mean, and geometric coefficient of variation (assuming log-normally distributed data). Values below the LLOQ will be reported with a clear sign indicating that they were below the LLOQ. Individual concentrations of UCB7665 will also be displayed graphically.

### 14.4.3 Pharmacodynamic analysis

For all PD variables, descriptive statistics for the change from Baseline, and percentage change from Baseline will be tabulated by treatment group and time point.

serum total intions the reconstructions aximum virized The PD variables will include MG-specific autoantibodies IgG, and IgG subclasses. In addition, for serum total IgG, the minimum value and maximum decrease from Baseline (including percentage decrease) will be evaluated and summarized.

Population PK analyses and PK/PD analyses may be conducted for the PD variables of interest. All such PK and PK/PD analyses will be described in a separate Data Analysis Plan, however, results will not be reported in the clinical study report.

### 14.4.4 Immunological variables

All immunological variables including concentrations of Igs (IgA, IgE, and IgM), serum complement levels (C3 and C4) and plasma complement levels (C3a and C5a), and serum BAFF will be listed and summarized, using descriptive statistics, by Treatment Group and visit including changes from Baseline. Concentrations of cytokines will be listed and summarized if there are sufficient data. Figures of mean values and changes from Baseline of immunological variables may be presented, and will be described in the SAP.

status (negative or confirmed positive) and either changes in relative mass units from Baseline for all scheduled assessments or titres for those confirmed positive will be listed and summarized by treatment group.

antibodies will be listed and summarized by The treatment group.

### 14.4.5 Subject exit interview

The anonymous audio-recordings will be analyzed by a third party and reported outside the clinical study report.

### Handling of protocol deviations 14.5

Important protocol deviations are identified as part of the data cleaning process in the Data Cleaning Plan (DCP). Ongoing data cleaning meetings will be held throughout the duration of the study. Objectives of these meetings include to review and update (if necessary) the important protocol deviations in the DCP and discuss exclusion of subjects from analysis populations. Furthermore, overall trends in protocol deviations will be discussed at the Data Evaluation Meeting. Through this ongoing data cleaning and evaluation process, all decisions regarding important protocol deviations and exclusions from analysis populations are made on an ongoing basis.

### 14.6 Handling of dropouts or missing data

All imputation of missing or partial dates for safety assessments, as well as handling missing efficacy data (where applicable), will be detailed in the SAP.

## 14.7 Planned interim analysis and data monitoring

At least three interim analyses will be performed. The first interim analysis for futility will be performed once approximately 20 subjects have attended Visit 9, the first visit of the second Dosing Period (ie, Day 29). Futility of UCB7665 will be assessed based on QMG score, MG-Composite score, and MGADL data. In case of futility, the study will be stopped or amended. The decision rules for futility will be described in the DMC charter. The second interim analysis will be conducted after approximately 20 subjects (receiving 6 sc infusions) have had Visit 16 (Day 57). Based on this unblinded analysis the safety of UCB7665 will be assessed by the DMC. The safety variables to be used and the potential outcomes of the analysis will be specified in the DMC charter. During this review recruitment will not be stopped. The third interim analysis will be performed once all subjects have attended Visit 9 (Day 29), the first visit of the second Dosing Period (ie, Day 29). This interim analysis will provide the results for the primary variable 'change from Baseline to Visit 9 (Day 29) in the QMG score', and 'change from Baseline to Visit 9 (Day 29) in MG-Composite score' and 'change from Baseline to Visit 9 (Day 29) in the third interim analysis the DMC will not be utilized.

The analyses will be described in a separate Interim SAP. The first interim analysis will utilize all efficacy data (as specified in the DMC charter), which will be available at the time the 20<sup>th</sup> subject attended Visit 9. The second interim analysis will utilize all safety data (as specified in the DMC charter), which will be available at the time the 20<sup>th</sup> subject attended Visit 16. For all interim analyses, the data subject to analysis should be as clean as possible; however, the database will not be locked and a snapshot will be taken.

If needed, subsequent DMC meetings will take place. The timing of further interim analyses and reviews of data by DMC will be decided by the DMC. Ad hoc DMC meetings can be held for reasons determined appropriate by the sponsor,

The deliberations and decisions of the DMC will be formally minuted/documented.

A detailed description of the DMC composition, processes, and responsibilities will be provided in a separate DMC charter.

## 14.8 Determination of sample size

The primary efficacy endpoint of this study is change in QMG score from Baseline to Visit 9 (Day 29).

The sample size calculation use a 1-sided significance level, an estimate (based on a of the SD for change in QMG of and an anticipated treatment effect of (Zinman et al, 2007).

Assuming a treatment difference of points in the mean change from Baseline in QMG at Visit 9 between the placebo and UCB7665 treatment arm with SD equal to a sample size of subjects (for each treatment group) provides >90% power to detect a treatment difference. Further it will be assumed that approximately of the randomized subjects cannot be utilized for the FAS and, hence subjects will be randomized.

## 15 ETHICS AND REGULATORY REQUIREMENTS

### 15.1 Informed consent

Subject's informed consent must be obtained and documented in accordance with local regulations, ICH-GCP requirements, and the ethical principles that have their origin in the principles of the Declaration of Helsinki.

Prior to obtaining informed consent, information should be given in a language and at a level of complexity understandable to the subject in both oral and written form by the investigator (or designee). Each subject will have the opportunity to discuss the study and its alternatives with the investigator.

Prior to participation in the study, the Informed Consent form should be signed and personally dated by the subject, or his/her legal representative, and by the person who conducted the informed consent discussion (investigator or designee). The subject or his/her legal representative must receive a copy of the signed and dated Informed Consent form. As part of the consent process, each subject must consent to direct access to his/her medical records for study-related monitoring, auditing, IRB/IEC review, and regulatory inspection.

If the Informed Consent form is amended during the study, the investigator (or the sponsor, if applicable) must follow all applicable regulatory requirements pertaining to the approval of the amended Informed Consent form by the IRB/IEC and use of the amended form.

All studies conducted at centers in the USA must include the use of a Health Insurance Portability and Accountability Act Authorization form.

The subject may withdraw his/her consent to participate in the study at any time. A subject is considered as enrolled in the study when he/she has signed the Informed Consent form. An eCRF must not be started, nor may any study specific procedure be performed for a given subject, without having obtained his/her written consent to participate in the study.

Subjects have the right to withdraw their consent for the exploratory genomic substudy at any point without any impact on their care or participation in the main study. In this case, any data already generated on the samples will be retained and used, but no further analysis will occur.

## 15.2 Subject identification cards

Upon signing the Informed Consent and Assent form (as applicable), the subject or legal representative will be provided with a subject identification card in the language of the subject. The investigator will fill in the subject identifying information and medical emergency contact information. The investigator will instruct the subject to keep the card with him/her at all times.

# 15.3 Institutional Review Boards and Independent Ethics Committees

The study will be conducted under the auspices of an IRB/IEC, as defined in local regulations, ICH-GCP, and in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

The investigator/UCB will ensure that an appropriately constituted IRB/IEC that complies with the requirements of the current ICH-GCP version or applicable country-specific regulations will be responsible for the initial and continuing review and approval of the clinical study. Prior to


initiation of the study, the investigator/UCB will forward copies of the protocol, Informed Consent form, Investigator's Brochure, investigator's curriculum vitae (if applicable), advertisement (if applicable), and all other subject-related documents to be used for the study to the IRB/IEC for its review and approval.

Ine investigator will also promptly report to the IRB/IEC all changes in the study, all unanticipated problems involving risks to human subjects or others, and any protocol deviations to eliminate immediate hazards to subjects.

The investigator will not make any changes in the study or at a approval, except where necessary approval, except where necessary approval.

minor changes to a previously approved protocol during the period covered by the original approval, it may be possible for the investigator to obtain an expedited review by the IRB/IEC as allowed.

As part of the IRB/IEC requirements for continuing review of approved studies, the investigator will be responsible for submitting periodic progress reports to the IRB/IEC (based on IRB/IEC requirements), at intervals appropriate to the degree of subject risk involved, but no less than once per year. The investigator should provide a final report to the IRB/IEC following study completion.

UCB (or its representative) will communicate safety information to the appropriate regulatory authorities and all active investigators in accordance with applicable regulatory requirements. The appropriate IRB/IEC will also be informed by the investigator or the sponsor, as specified by the applicable regulatory requirements in each concerned country. Where applicable, investigators are to provide the sponsor (or its representative) with evidence of such IRB/IEC notification.

### **Subject privacy** 15.4

UCB staff (or designee) will affirm and uphold the subject's confidentiality. Throughout this study, all data forwarded to UCB (or designee) will be identified only by the subject number assigned at Screening.

The investigator agrees that representatives of UCB, its designee, representatives of the relevant IRB/IEC, or representatives of regulatory authorities will be allowed to review that portion of the subject's primary medical records that directly concerns this study (including, but not limited to, laboratory test result reports, ECG reports, admission/discharge summaries for clinic/hospital admissions occurring during a subject's study participation, and autopsy reports for deaths occurring during the study).

### **Protocol amendments**

Protocol changes may affect the legal and ethical status of the study and may also affect the statistical evaluations of sample size and the likelihood of the study fulfilling its primary objective.

Significant changes to the protocol will only be made as an amendment to the protocol and must be approved by UCB, the IRB/IEC, and the regulatory authorities (if required), prior to being implemented.

## 16 FINANCE, INSURANCE, AND PUBLICATION

Insurance coverage will be handled according to local requirements.

Finance, insurance, and publication rights are addressed in the investigator and/or CRO agreements, as applicable.

### 17 REFERENCES

Anderson CL, Chaudhury C, Kim J, Bronson CL, Wani MA, Mohanty S. Perspective-- FcRn transports albumin: relevance to immunology and medicine. Trends Immunol. 2006;27(7):343-8.

Barnett C, Katzberg H, Nabavi M, Bril V. The quantitative myasthenia gravis score comparison with clinical, electrophysiological, and laboratory markers. J Clin Neuromuscul Dis. 2012;13(4):201-5.

Barnett C, Bril V, Kapral M, Kulkarni A, Davis AM. A conceptual framework for evaluating impairments in myasthenia gravis. PLos One. 2014;9(5).

Barnett C, Bril V, Kapral M, Kulkarni A, Davis AM Development and validation of the Myasthenia Gravis Impairment Index. Neurology. 2016; 87(9): 879–886.Barth D, Nabari MN, Ng E, Nwe P, Bril V; Comparison of IVIg and PLEX in patients with myasthenia gravis. Neurology. 2011;76(23):2017-23.

Benatar M, Sanders DB, Burns TM, Cutter GR, Guptill JT, Baggi F,; Task Force on MG Study Design of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Recommendations for myasthenia gravis clinical trials. Muscle Nerve. 2012 Jun;45(6):909-17. doi: 10.1002/mus.23330. PubMed PMID: 22581550.

Burns TM, Conaway M, Sanders DB; MG Composite and MG-QOL15 Study Group. The MG Composite: A valid and reliable outcome measure for myasthenia gravis. Neurology. 2010 May 4;74(18):1434-40.

CPMP/ICH/135/95 Note for guidance on Good Clinical Practice (EMEA) Jul 2002.

Gilhus NE, Verschuuren JP. Myasthenia gravis: subgroup classification and therapeutic strategies.Lancet Neurol. 2015;14(10):1023-36.

Howard JF Jr, Baronn RJ, Cutter GR, Freimer M, Juel VC, Mozaffar T, Mellion ML, Benatar MG, Farrugia ME, Wang JJ, Malhotra SS, Kissel JT; MG Study Group. A randomized, double-blind, placebo-controlled phase II study of eculizumab in patients with refractory generalized myasthenia gravis. Muscle Nerve. 2013 Jul;48(1):76-84. doi: 10.1002/mus.23839. Epub 2013 Apr 30. PubMed PMID: 23512355.

Johnsen J, Pathogenesis in immune thrombocytopenia: new insights. American Society of Hematology, Hematology 2012:306-312.

Lowe PJ, Tannenbaum S, Wu K, Lloyd P, Sims J. On setting the first dose in man: quantitating biotherapeutic drug-target binding through pharmacokinetic and pharmacodynamic models. Basic Clin Pharmacol Toxicol. 2010;106(3):195-209.

Muppidi S. The myasthenia gravis-specific activities of daily living profile. Ann N Y Acad Sci, 2012. 1274: p. 114-9

UCB7665

Muppidi S, Wolfe GI, Conaway M, Burns TM; MG COMPOSITE AND MG-QOL15 STUDY GROUP. MG-ADL: still a relevant outcome measure. Muscle Nerve. 2011 Nov;44(5):727-31.

Sanders, Single fiber EMG. In: Encyclopedia of the Neurological Sciences (Second Edition):
Elsevier; 2014: 169–172.

Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn PT Cactivities of daily living profile. Neurology 1900.

ents with myasther. 837-41.

Replace of the support any marketing authorization application and the used to support any marketing authorization and the used to support any marketing authorization. This document cannot be used to support any marketing authorization.

Zinman L, Ng E, Bril V. IV immunoglobulin in patients with myasthenia gravis: a randomized


| UCB<br>Clinical Stud | dy Protocol | | UCB7665 | | 15 Sep 20<br>MG00 |
|---|---|---|---|---|---|
| 18.2 | MG-C | omposite s | score | | |
| Figure 18 | 3.2: MG-C | omposite so | core | | |
| Ptosis, upward (<br>examination) | gaze (physician | >45 seconds = 0 | 11-45 seconds = 1 | 1-10 seconds = 2 | Immediate = 3 |
| Double vision or<br>left or right (phy<br>examination) | | > 45 seconds = 0 | 11-45 seconds = 1 | 1-10 seconds = 3 | Immediate = 4 |
| Eye closure (phy<br>examination) | ysician | Normal = 0 | Mild weakness (can be forced open with effort) = 0 | Moderate weakness (can be forced open easily) = 1 | Severe weakness (unable to<br>keep eyes closed) = 2 |
| Talking (patient | t history) | Normal = 0 | Intermittent slurring or nasal speech = 2 | Constant slurring or nasal but<br>can be understood = 4 | Difficult to understand<br>speech = 6 |
| Chewing (patien | nt history) | Normal = 0 | Fatigue with solid food = 2 | Fatigue with soft food = 4 | Gastric tube = 6 |
| Swallowing (pat | tient history) | Normal = 0 | Rare episode of choking or trouble swallowing = 2 | Frequent trouble swallowing,<br>e.g. necessitating changes in<br>diet = 5 | Gastric tube = 6 |
| Breathing (thou<br>caused by MG) | | Normal = 0 | Shortness of breath with exertion = 2 | Shortness of breath at rest = 4 | Ventilator dependence = 9 |
| Neck flexion or (<br>(weakest) (physics examination) | | Normal = 0 | Mild weakness = 1 | Moderate weakness (i.e., ~50% weak, ±15%) = 3* | Secrete weakness = 4 |
| Shoulder abduct examination) | ction (physician | Normal = 0 | Mild weakness = 2 | Moderate weakness (i.e., -50% weak, ±15%) = 4* | Severe weakness - 5 |
| Hip flexion (phys | rsician | Normal - 0 | Mild weakness = 2 | Moderate weakness (i.e/)<br>~50% weak, ±15% 4* | Severe weakness = 5 |
| | | × of | Inaike | | |
| | | io support | | | |
| cument can | notbelises | <b>&gt;</b> | Mild weakness = 2 e construed as weakness that has more severe than that would be a severe than that we have a severe than that we have a severe than that would be a severe than the severe than the severe than the severe that we have a severe than the severe than the severe that the s | | |
| ,,000 | | | | | |
# 18.8 Suggested management guidelines for infusion reactions

## Table 18.1: Suggested management guidelines for infusion reactions

| Type of reaction | Sponsor recommendations for management |
|---|---|
| Acute – Mild | Slow infusion rate to |
| eg, flushing, dizziness, headache, sweating, | Infuse 500-1000mL/h iv. |
| palpitations, nausea | Administer antihistamine iv/im. |
| | Administer paracetamol 1g orally. |
| | Monitor vital signs every 10 minutes until back to Baseline. |
| | as tolerated until intended dose has been given. |
| Acute – Moderate | Stop infusion. |
| eg, flushing, chest tightness, dyspnea, | Infuse 500-1000mL/h iv. |
| hypo/hypertension (change >20mmHg in systolic | Administer antihistamine iv/im. |
| blood pressure), raised temperature, palpitations, urticaria | Administer paracetamol 1g orally. |
| | Monitor vital signs every 5 minutes until back to Baseline. |
| | Wait 20 minutes. |
| Aut. Comment of the C | If there is no indication of anaphylaxis (eg, generalized urticaria and/or bronchospasm) and if clinically appropriate, consider restarting the infusion at a lower rate following this suggested |
| etine | regimen: |
| a diffe | Restart infusion at . |
| A RIV | Increase infusion rate to |
| Soft are, | as tolerated until intended dose has been given. |
| Acute – Severe | Stop infusion definitively. |
| eg, hypo/hypertension (change >40mmHg in | Alert crash team. |
| systolic blood pressure), raised temperature with | Maintain airway, ensure oxygen is available. |
| rigors, chest tightness, dyspnea with wheezing, stridor | If wheezing, give epinephrine 0.5mg im (0.5mL 1:1000 epinephrine). |
| carl. | Administer antihistamine iv/im. |
| | Administer corticosteroids iv. |
| rigors, chest tightness, dyspnea with wheezing, stridor | Monitor vital signs every 2 minutes until back to Baseline. |

im=intramuscular; iv=intravenous

### 18.9 Diagnosis of anaphylactic reactions

Anaphylaxis is highly likely when any of the following 3 criteria is fulfilled (Sampson et al, 2006):

1. Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (eg, generalized hives, pruritus or flushing, swollen lips-tongue-uvula)

#### AND AT LEAST ONE OF THE FOLLOWING

- a. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow [PEF], hypoxemia)
- b. Reduced blood pressure [BP] or associated symptoms of end-organ dysfunction (eg, hypotonia [collapse], syncope, incontinence)
- 2. Two or more of the following that occur rapidly after exposure to a likely allergen for that patient (minutes to several hours):
- a. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips tongue-uvula)
- b. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
- c. Reduced BP or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
- d. Persistent GI symptoms (eg, crampy abdominal pain, vomiting)
- 3. Reduced blood pressure after exposure to known allergen for that subject (minutes to several hours): Systolic BP of less than 90mmHg or greater than 30% decrease from the subject's Baseline systolic BP value.

#### 18.10 Headache Questionnaire

| Symptom | s & Frequency | of Severe Headac | ches | |
|---|---|---|---|---|
| 1. Date of | collection: | apolic | Time of collection: | |
| DD | MMM | XY | НН | MM |
| 2. Is the si | ubject suffering | from a severe head | lache? | |
| Yes | US | | | |
| No | o'i bo | | | |
| a. Which | of the following | best describes hov | v the subject is affected? | |
| Able to fu | nction normally | | | |
| Activity in | mpaired to some | degree | | |
| Activity s | everely impaired | I | | |
| Bed rest re | equired | | | |
| b. Rate yo | our pain on a scal | le of 0 - 10: | | |

| Symptoms & Frequency of Severe Headaches |
|---|
| 3. During the course of this headache, has the subject experienced any of the following? |
| a. Nausea: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| b. Vomiting: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| c. Dizziness: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| i. Vertigo: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| ii. Nonvertigo: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| d. Increased neck pain or stiffness: |
| 0 Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |

| Symptoms & Frequency of Severe Headaches |
|--------------------------------------------------|
| e. Increased sensitivity to light: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| f. Increased sensitivity to noise: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| g. Increased sensitivity to smell: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| h. Pain made worse by routine physical activity: |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| i. Pain on one side of head only |
| 0 = Never |
| 1 = Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| j. Pulsating/throbbing headaches: |
| 0 = Never |
| 1 Rarely |
| 2 = Less than half the time |
| 3 = Half the time or more |
| k. Weakness on one side: |

| Symptoms & Frequency of Severe | Headaches |
|---|---|
| 0 = Never | |
| 1 = Rarely | |
| 2 = Less than half the time | |
| 3 = Half the time or more | :0 |
| 1. Seeing shimmering lights, lines, de headache and lasts more than a few | ark spots, other shapes or colors before the eyes, before or during the minutes but less than an hour: |
| 0 = Never | gions |
| 1 = Rarely | tens |
| 2 = Less than half the time | 20, |
| 3 = Half the time or more | 93 |
| m. One-sided numbness of lips, tong headache becomes severe and lasts l | gue, fingers, or legs that migrates or moves and starts before the ess than an hour: |
| 0 = Never | Rt dico |
| 1 = Rarely | 00, 300, |
| 2 = Less than half the time | adiio. |
| 3 = Half the time or more | DA NORTH |
| General | The questionnaire should be administered via an interview with the subject. The recall period for the first time the questionnaire is administered is since the severe headache began. |
| A to support | The recall period for subsequent questionnaires should be since the prior administration of the questionnaire, not since the start of the severe headache. Mark an X in only 1 box for each question. Do not write in any other choices. Transcribe the subject's responses to the eCRF screen. |

DD MMM YYYY (v.2009-09-09)

The protocol has been amended to incorporate the feedback from the U.S. Food and Drug administration (FDA) received on 09 December 2016 and the new company standard in TB management.

In addition, minor administrative changes have been made.

The following shows the changes medical dated 21 Oct 2016

dated 21 Oct 2016.

#### Modifications and changes

#### Global changes

The following changes were made throughout the protocol:

- Secondary efficacy variables and other efficacy variables were updated. Statistical analyses sections were updated accordingly.
- Sections covering collection of exploratory biomatker samples and exploratory safety biomarker sample were simplified.
- Exploratory biomarker sampling was separated from exploratory safety biomarker sampling.
- Timing of the IRT to be called was updated (at Screening and on dosing visits only, not every single visit).
- Wording for home visit at Visit 20 to be conducted at home was revised throughout the protocol. Now the home visits are allowed at Visits 17 and 19.
- The C-SSRS was added to address the request of the FDA that prospective assessments for suicidality should be included in clinical trials involving all drugs for neurological indications.
- The detailed tuberculosis assessment was added to ensure the subject safety.
- The term on-demand treatment was revised into chronic-intermittent treatment.
- Editorials and revisions on abbreviations were implemented.

## Specific changes

## Change #1

SUMMARY, 3<sup>rd</sup> paragraph

The study will consist of 3 Periods: Screening, Treatment, and Observation. After Screening, subjects will enter the Treatment Period, which will consist of 2 successive Dosing Periods.

Subjects will receive 3 doses of investigational medicinal product (IMP) at weekly intervals during both Dosing Period 1 and Dosing Period 2. Dosing Period 1 will be 4 weeks, with 2 parallel arms (UCB7665 7mg/kg or placebo). Dosing Period 2 will be 2 weeks, with 2 parallel treatment arms (UCB7665 7mg/kg or UCB7665 4mg/kg).

#### Has been changed to:

Dosing Period 1 will be 4 weeks, with 2 parallel treatment arms (UCB7665 7mg/kg).

Dosing Period 2 will be 2 weeks, with 2 parallel treatment arms (UCB7665 7mg/kg).

ange #2

SUMMARY, 4<sup>rd</sup> and e<sup>th</sup> The study will consist of 3 Periods: Screening, Treatment, and Observation. After Screening, subjects will enter the Treatment Period, which will consist of Dosing Period 1 followed by Dosing Period 2. Subjects will receive 3 doses of investigational medicinal product (IMP) at weekly intervals during each dosing period as follows:

### Change #2

A Data Monitoring Committee (DMC) will oversee at least 1 interim analysis for safety and for futility during the course of the study (see Section 14.7). Details of the interim analysis will be provided in the DMC charter and interim Statistical Analysis Plan (SAP).

The primary efficacy variable will be the change from Baseline in Quantitative MG (QMG) score to Visit 9 (Day 29). Other efficacy variables will be the following: change from Baseline in MG-Composite score to Visit 9 (Day 29); value and change from Baseline in QMG at each scheduled assessment during Treatment and Observation Periods; proportion of QMG responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MG-Composite score at each scheduled assessment during Treatment and Observation Periods; proportion of MG-Composite responder ( $\geq$ 3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MG muscle weakness severity and fatigue scales at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MG-Activities of Daily Living (MGADL) at each scheduled assessment during Treatment and Observation Periods; and change in mean jitter in single fiber electromyography (SFEMG) from Baseline to Visit 9 for the subjects consenting to this measurement at participating sites.

# Has been changed to:

1 SUMMARY, 5<sup>th</sup> and 6<sup>th</sup> paragraph

A Data Monitoring Committee (DMC) will be implemented as described in Section 14.7.

The primary efficacy variable will be the change from Baseline in Quantitative MG (QMG) score to Visit 9 (Day 29). The secondary efficacy variables will be the change from Baseline in MG-Composite score to Visit 9 (Day 29) and the change from Baseline in MG-Activities of Daily Living (MGADL) score to Visit 9 (Day 29). Other efficacy variables will be the following: value and change from Baseline in QMG at each scheduled assessment during Treatment and Observation Periods; QMG responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MG-Composite score at each scheduled assessment during Treatment and Observation Periods; MG-Composite responder (≥3.0 point improvement from Baseline) at each scheduled assessment As or variations thereof during Treatment and Observation Periods; value and change from Baseline in MGADL at each scheduled assessment during Treatment and Observation Periods; MGADL responder (>3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods: Myasthenia Gravis Foundation of America (MGFA) classification at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in MG muscle weakness severity and fatigue scales at each scheduled assessment during Treatment and Observation Periods; and change in mean jitter in single fiber electromyography (SFEMG) from Baseline to Visit 9 for the subjects consenting to this measurement at participating sites.

#### Change #3

## SUMMARY, 6<sup>th</sup> to 8<sup>th</sup> paragraph

Plasma concentration of UCB7665 over time will be assessed as the pharmacokinetic (PK) variable. The main pharmacodynamic (PD) variables will be the maximum decrease from Baseline in serum total immunoglobulin G (IgG) concentration; value and change from Baseline in serum IgG subclass concentrations at each scheduled assessment during Treatment and Observation Periods; and value and change from Baseline in total serum IgG concentrations at each scheduled assessment during Treatment and Observation Periods.

Safety and tolerability variables will include occurrence of treatment-emergent adverse events (TEAEs); vital sign values and changes from Baseline (systolic and diastolic blood pressure [BP], temperature, pulse rate, respiratory rate, and body weight); 12-lead electrocardiogram (ECG) values parameters and change from Baseline; laboratory values (hematology, clinical chemistry, and urinalysis) and changes from Baseline; change from Baseline in exploratory safety biomarkers

) only in subjects experiencing severe headache and/or moderate to severe gastrointestinal (GI) disturbance; and TEAEs leading to withdrawal of

During this study, subjects will also have the option of providing additional informed consent for exploratory deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) (ie, messenger RNA [mRNA] and micro RNA [miRNA]) analyses (see Section 5.1.1). Participation in this additional portion of the study is optional and does not preclude subject's eligibility for participation in the main study. The additional genomic samples must not be collected if the subject has not consented to participate in this exploratory genomic substudy.

# Has been changed to:

1 SUMMARY, 7<sup>th</sup> to 10<sup>th</sup> paragraph

Other and exploratory variables include: safety and tolerability variables, pharmacokinetic (PK), Pharmacodynamic (PD), and immunologic variables.

Safety and tolerability variables include the following: occurrence of treatment-emergent adverse events (TEAEs); vital sign values and changes from Baseline (systolic and diastolic blood pressure [BP], temperature, pulse rate, respiratory rate, and body weight); 12-lead


electrocardiogram (ECG) values and change from Baseline; laboratory values (hematology, clinical chemistry, and urinalysis) and changes from Baseline; change from Baseline in exploratory safety biomarkers (may include but not limited to

in subjects experiencing severe headache and/or moderate to severe gastrointestinal (GI) disturbance; and TEAEs leading to withdrawal of IMP.

Plasma concentration of UCB7665 over time will be assessed as the PK variable. The main PD variables will be the maximum decrease from Baseline in serum total immunoglobulin G (IgG) concentration; value and change from Baseline in total serum IgG concentrations at each scheduled assessment during Treatment and Observation Periods; value and change from Baseline in serum IgG subclass concentrations at each scheduled assessment during Treatment and Observation Periods; and change in MG-specific autoantibody levels in serum from Baseline at each scheduled assessment during Treatment and Observation Periods. Additionally, change from Baseline in other immunological variables and other exploratory biomarkers during the Treatment and Observational Periods will be assessed.

During this study, subjects will also have the option of providing additional informed consent for exploratory deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) (ie, messenger RNA [mRNA] and micro RNA [miRNA]) analyses (see Section 5.1.1) to understand the cause, progression, and appropriate treatment of MG. Participation in this additional portion of the study is optional and does not preclude subject's eligibility for participation in the main study. The additional genomic samples must not be collected if the subject has not consented to participate in this exploratory genomic substudy.

### Change #4

2 INTRODUCTION, 11<sup>th</sup> paragraph

MG0002 will be the first study of the use of UCB7665 in MG.

## Has been changed to:

2 INTRODUCTION, 11th paragraph

MG0002 will be the first study of the use of UCB7665 in MG. The aim of the study is to evaluate the efficacy, safety, and immunological effect of UCB7665, and to gather data for future study planning to fully evaluate the use of UCB7665 in MG.

## Change #5

3.2 Secondary objectives

The following was added:

To gather data for future study planning, whether for chronic-intermittent treatment or a longer therapy option by evaluating the general concept that UCB7665 has a clinical effect in patients with generalized MG

#### Change #6

- 3.3 Exploratory objectives
- To evaluate the effect of UCB7665 on B-cell activating factor (BAFF) and on cytokines (for subjects experiencing infusion reactions)

#### Has been changed to:

- 3.3 Exploratory objectives
- To evaluate the effect of UCB7665 on B-cell activating factor (BAFF) and on cytokines (in all subjects)
- To evaluate the effects of UCB7665 on blood biomarkers for safety (including, but not limited to
   only in subjects with severe headache and/or moderate to severe GI

In addition, the following were added:

- To evaluate the effect of UCB7665 on cytokines in subjects experiencing infusion reactions
- To evaluate peripheral blood biomarkers in relation to disease etiology, progression and treatment outcome

## Change #7

disturbance

4.1.2 Secondary efficacy variable

The secondary efficacy variable is:

Change from Baseline in MG-Composite score to Visit 9 (Day 29)

## Has been changed to:

4.1.2 Secondary efficacy variable

The secondary efficacy variables are:

- Change from Baseline in MG-Composite score to Visit 9 (Day 29)
- Change from Baseline in MGADL score to Visit 9 (Day 29)

## Change #8

- 4.1.3 Other efficacy variables
- Proportion of QMG responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
- Proportion of MG-Composite responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods

#### Has been changed to:

- 4.1.3 Other efficacy variables
- QMG responder (≥3.0 point improvement from Baseline) at each scheduled assessment
- MG-Composite responder (≥3.0 point improvement from Baseline) at each scheduled

In addition, the following was added:

Income from Baseline) at each scheduled

Baseline) at each scheduled

Baseline) at each scheduled assessment with the following was added:

MGADL responder (≥3.0 point improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods

Baseline) at each scheduled assessment with the following the following the following the following the following the following was added:

MGADL responder (≥3.0 point improvement from Baseline) at each scheduled assessment during the following the following was added:

Pharmacokine: eduled assessmand and any extensions and any extensions.

25 RELDACTED COPT application application and any extensions and any extensions.

Relation application application and any extensions.

### Change #9

Sections 4.2 to 4.4 have been restructured:

- 4.2 Pharmacokinetic and pharmacodynamic variables
- 4.2.1 Pharmacokinetic variable
- 4.2.2 Pharmacodynamic variables
- 4.3 Immunological variables
- 4.4 Safety variables

#### Has been changed to:

- 4.2 Other and exploratory variables
- 4.2.1 Safety variables
- 4.2.2 Pharmacokinetic variable
- 4.2.3 Pharmacodynamic variables
- 4.2.4 Immunological variables

## Change #10

4.2 Pharmacodynamic variables (previous heading number)

The heading number was changed to the below:

4.2.3 Pharmacodynamic variables

The below was deleted:

Change from Baseline total IgG concentration pre- and post-ADA depletion at each scheduled assessment during Treatment and Observation Periods

## Change #11

4.3 Immunological variables (previous heading number)

Additional exploratory biomarkers may be investigated if needed using the samples already available.

- 4.2.4 Immunological variables (new heading number)
- Change from Baseline in exploratory biomarkers relating to mechanism of action, disease activity, treatment response, and clinical outcome

UCB7665

### Change #12

- 4.4 Safety variables (previous heading number)
- Change from Baseline in exploratory safety biomarkers (
   at each scheduled assessment during Treatment and
   Observation Periods (only in subjects with severe headache and/or moderate to severe GI disturbance)

#### Has been changed to:

- 4.2.1 Safety variables (new heading number)
- Change from Baseline in exploratory safety biomarkers (may include but not limited to

in subjects with severe headache and/or moderate to severe GI disturbance

#### Change #13

5.1 Study description

**Treatment Period:** The Treatment Period will consist of 2 successive Dosing Periods. Subjects will receive 3 doses of IMP at weekly intervals during both Dosing Period 1 and Dosing Period 2. Dosing Period 1 will be 4 weeks, with 2 parallel Treatment Groups (UCB7665 7mg/kg or placebo). Dosing Period 2 will be 2 weeks, with 2 parallel Treatment Groups (UCB7665 7mg/kg or UCB7665 4mg/kg).

## Has been changed to:

5.1 Study description

**Treatment Period:** The Treatment Period will consist of Dosing Period 1 followed by Dosing Period 2. Subjects will receive 3 doses of IMP at weekly intervals during each dosing period as follows.

- Dosing Period 1 will be 4 weeks, with 2 parallel Treatment Groups (UCB7665 7mg/kg or placebo).
- Dosing Period 2 will be 2 weeks, with 2 parallel Treatment Groups (UCB7665 7mg/kg or UCB7665 4mg/kg).

# Change #14

5.1 Study description

**Óbservation Period:** All subjects must be followed for 8 weeks after the final dose of IMP is administered. Subjects will return to the clinic for Visits 15, 16, and 18 for efficacy and for safety assessments (see Section 5.2, Schedule of Assessments). Subjects will either return to the clinic/hospital, or, if possible and agreed by investigator and subject, have home visits conducted

by certified healthcare professionals, for Visits 17, 19, and 20. The Observation Period begins the day after the final dose of IMP (ie, Visit 13, Day 43); Visit 15 (Day 50) is the first visit in the Observation Period.

A DMC will be established to monitor mainly safety data during the study. In addition efficacy data will be assessed once during the study for futility. The DMC will be unblinded and details of the DMC composition, processes, and responsibilities will be documented in the DMC charter.

#### Has been changed to:

#### 5.1 Study description

**Observation Period:** All subjects must be followed for 8 weeks after the final dose of IMP is S, a., Subject, ha ... The Observat. ... 15 (Day 50) is the ... 15 ( administered. Subjects will return to the clinic for Visits 15, 16, 18, and 20 for efficacy and for safety assessments (see Section 5.2, Schedule of Assessments). Subjects will either return to the clinic/hospital, or, if possible and agreed by investigator and subject, have home visits conducted by certified healthcare professionals, for Visits 17 and 19. The Observation Period begins the day after the final dose of IMP (ie, Visit 13, Day 43); Visit 15 (Day 50) is the first visit in the


# Change #15

**Table 5.1:** Schedule of assessments

| UCB<br>Clinical Study Pr | otocol | | | | | | | | | UCB76 | 565 | | | | | | | | | | 15 Sep<br>Mo | p 201′<br>G000′ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Change #1 | | | | | | | | | | | | | | | | | | | | 13/18 | ijions | |
| Changes on the | e tables a Schedu | | | | ents | 5 | | | | | | | | | | | | SION | Sol | 7 | tions the | |
| Assessments | Screenin | ıg | Treati | nent l | Period | | | | | I | | | | | | Obs | | | eriod | | | UV |
| | | | Dosing | | | | | | I | | g Perio | | | I | | , King | | | I | l | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | 5b | 6 | 7b | 8 | 9 | 10b | 11 | 12b | 13 | 14b | 15 | 16 | 17 | 18 | 19 | 20 FV/PEOT<br>c | |
| | Day | -28 to<br>-1 | 1 | 2 | <b>8</b> (± 2 | 9 | 15<br>(± 2 | 16 | 22<br>(± 2 | 29<br>(± 2 | 30 | 36<br>(± 2 | 37 | 43)<br>(± 2 | 44 | 50 | 57 | 64 | 78 | 92 | 99<br>(± 2 days) | |
| | | | | | days) | | days) | | days) | days) | O <sub>X</sub> | days) | 366 <sub>111</sub> | days) | | | (± 2 | days) | 1 | | | |
| Written informed c | onsent | X | | | | | | | | ,Q` | , | 70, | 0 | | | | | | | | | |
| Written informed cogenomic substudy | onsent for | X | | | | | | | C | | 3112 | Y | | | | | | | | | | |
| Demographic data | | X | | | | | | ~ | Ò, | X | 300 | | | | | | | | | | | |
| Verification of inclexclusion criteria | usion | X | X | | | | | <b>/</b> - | | 100 | | | | | | | | | | | | |
| Call or enter IRT to | register | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Call to IRT / Rando | mization | | X | | | | a C | 7 | | X | | | | | | | | | | | | |
| Withdrawal criteria | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| General medical/pr<br>history | ocedures | X | | | O. | ,716 <sub>6,</sub> | | | | | | | | | | | | | | | | |
| Prior and concomit nedication | ant | X | X | X | × | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medicorocedures | al | | X | 72 | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Vital signs <sup>e</sup> | | X | X | | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |

Table 5.1: Schedule of assessments

| UCB<br>Clinical Study Pro | otocol | | | | | | | | - | UCB76 | 565 | | | | | | | | | | 15 Ser<br>MO | G0002 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | Schedu | le of | asse | ssm | ents | 6 | | | | | | | | | | | | | | | tions | |
| Assessments | Screenin | ıg | Treat | ment l | Period | | | | | | | | | | | Obs | ervat | tion P | eriod | Jaile | | UV |
| | | | Dosin | g Peri | od 1 | | | | | Dosin | g Perio | d 2 | | | | | | | c or | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | 5b | 6 | 7 <b>b</b> | 8 | 9 | 10b | 11 | 12b | 13 | 14b | 15 | 16 | .13 | 18 | 19 | 20 FV/PEOT | |
| | Day | -28 to<br>-1 | 1 | 2 | 8<br>(± 2<br>days) | 9 | 15<br>(± 2<br>days) | 16 | 22<br>(± 2<br>days) | 29<br>(± 2<br>days) | 30 | 36<br>(± 2<br>days) | 37 | 43<br>(± 2<br>days) | 44 | 50 | 57<br>(± 2 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| Body weight, heigh | f<br>nt | X | | | 3 / | | 3 / | | 3 / | X | | , | | | and | | | | | | X | |
| Recording of AEs | | X | X | X | X | X | X | X | X | X | X | X | X | X) | X | X | X | X | X | X | X | X |
| Full physical exami | ination | X | | | | | | | | | 5 | | dic | 300 | | | | | | | X | |
| Brief physical exan | nination | | X | | | | | | | X ( | 9 | | 3.66 | | | | | | | | | |
| Full neurological ex | xamination | X | | | | | | | Ć | (ED | :13 | ilon | | | | | | | | | X | |
| Brief neurological examination | | | X | | | | | OK. | OP. | X | not | | | | | | | | | | | |
| 12-lead ECG <sup>h</sup> | | X | X | | X | | X | | X | (X) | | X | | X | | X | | | X | | X | |
| Laboratory tests (he chemistry, urinalys | | X | X | | X | | X | ~3 | NAS. | X | | X | | X | | X | X | | X | | X | |
| Serology testing for<br>Hepatitis B, Hepati<br>active or latent TB | r HIV,<br>tis C, and | X | | | | | K al | 4 | | | | | | | | | | | | | | |
| Blood sampling for UCB7665 <sup>i</sup> | PK of | | X | | X | ilik | X | | X | X | | X | | X | | X | | | | | | |
| Blood sampling for analysis (optional) | DNA | | x <sup>j</sup> | 150 | | | | | $\mathbf{X}^{\mathrm{j}}$ | | | | | $X^{j}$ | | | | | | | | |
| Blood sampling for analysis (optional) | RNA | | X <sup>j</sup> | | X <sup>j</sup> | | | | $X^{j}$ | | | | | $X^{j}$ | | | | | | | X <sup>j</sup> | |
| Serum pregnancy to | est | X | U. | | | | | | | | | | | | | | | | | | | |

Table 5.1: Schedule of assessments

| Table 5.1: \$ | Schedu | le of | 2888 | sem | ente | | | | | | | | | | | | | | | | 15 September 15 September 15 Miles The Committee of the C | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screenin | | Treati | | | | | | | | | | | | | Obs | ervat | ion P | eriod | | | UV |
| | | | Dosing | g Peri | od 1 | | | | | Dosin | g Perio | d 2 | | | | | | | o's | 10 | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> b | 6 | 7 <b>b</b> | 8 | 9 | 10b | 11 | <b>12</b> b | 13 | <b>14</b> b | 15 | 16 | . <b>1</b> 30 | 18 | 19 | 20 FV/PEOT | |
| | Day | -28 to<br>-1 | 1 | 2 | 8<br>(± 2 | 9 | 15<br>(± 2 | 16 | 22<br>(± 2 | 29<br>(± 2 | 30 | 36<br>(± 2 | 37 | 43<br>(± 2 | 44 | 50 | 57 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| J | <u> </u><br>k | | X | | days)<br>X | | days)<br>X | | days)<br>X | days) | | days)<br>X | | days)<br>X | and | <b>X</b> | (± 2 | X | X | X | X | |
| Urine pregnancy test | | | | | X | | X | | Λ | X | | X | | - | <i>Q</i> , | Λ | Λ | Λ | A | Λ | A | |
| Administration of IM | IP | | X<br>X | | X | | X | | X | X | 7 | X | | XO. | | X | X | X | X | X | X | |
| Serum complement (<br>and plasma complem<br>(C3 <sub>A</sub> and C5a) | | | X | | X | | X | | X | X | 0 | X | 3/9 | X | | X | X | Λ | Λ | Λ | X | |
| Immunoglobulins (to<br>and IgG subclasses) | tal IgG | X | X | | X | | X | 1 | O.X.C | X | noill | X | | X | | X | X | X | X | X | X | |
| IgG depletion assay | | | X | | X | | X | 4 | X | X | | X | | X | | X | X | X | X | X | X | |
| IgA, IgM, IgE | | | X | | | | | | X | X | | X | | X | | X | X | | | | X | |
| MG-specific autoanti | ibodies | | X | | X | | | _0 | 1/2 | X | | X | | | | X | | | | | X | |
| Exploratory<br>biomarkers : includin | ng | | X | | Х | .05 | X | 7 | Х | X | | X | | X | | X | X | X | X | X | X | |
| BAFF analysis | | | X | | X c | 264 | X | | X | X | | X | | X | | | | X | | X | | |
| Cytokines <sup>m</sup> | | | X | 7 | X. | | X | | X | X | | X | | X | | X | X | X | X | X | X | Х |
| Vaccination-specific | antibody | Х | , /o <sup>©</sup> | 150 | | | | | | | | | | | | | | | | | X | |

Table 5.1: Schedule of assessments

| Assessments | Screenin | ıg | Treati | ment l | Period | | | | | | | | | | | Obs | ervat | ion P | eriod | Jail | 2 | UV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosing | g Peri | od 1 | | | | | Dosin | g Perio | d 2 | | | | | | | O | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | 5b | 6 | 7 <b>b</b> | 8 | 9 | 10b | 11 | 12b | 13 | 14b | 15 | 16 | .13°C | 18 | 19 | 20 FV/PEOT | |
| | Day | -28 to | 1 | 2 | 8 | 9 | 15 | 16 | 22 | 29 | 30 | 36 | 37 | 43 | 44 | 50 | 57 | 64 | 78 | 92 | 99 | |
| | | -1 | | | (± 2<br>days) | | (± 2<br>days) | | (± 2<br>days) | (± 2 days) | | (± 2<br>days) | | (± 2<br>days) | > 0 | Jiny. | (± 2 | days) | | | (± 2 days) | |
| QMG scale <sup>n</sup> | | X | X | | X | | X | | X | X | | X | | X | Silve | X | X | | X | | X | |
| Muscle weakness sev fatigability scale | verity and | | X | | X | | X | | X | X | 4 | X | | SHO | | X | X | X | X | X | X | |
| Fatigue scale | | | X | | X | | X | | X | X | OR | X | 30P1 | X | | X | X | X | X | X | X | |
| MGADL scale | | | X | | | | | | | X | ) | 5 | 0. | | | X | | X | | | X | |
| MGFA classification | | X | X | | | | | | ć | X | .13 | ), I | | | | | | | | | X | |
| SFEMG measuremen | nt <sup>o</sup> | | X | | | | | / | OR | X | COLL | | | | | | | | | | | |
| Headache questionna | ire <sup>p</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Stool sample assessm | nent <sup>q</sup> | | X | | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Subject exit interview | V | | | | | | | 2 | 3/1 | | | | | | | | | | | | X | |

AE=adverse event; BAFF=B-cell activating factor; BL=Baseline; BP=blood pressure; CSF=cerebrospinal fluid; CT=computed tomography; DNA=deoxyribonucleic acid; ECG=electrocardiogram; FV=Final Visit; GI=gastrointestinal; HIV=human immunodeficiency virus; IgA=immunoglobulin A; IgE=immunoglobulin E; IgG=immunoglobulin G; IgM=immunoglobulin M; IMP=investigational medicinal product; IRT=interactive response technology; LP=lumbar puncture; MG=myasthenia gravis; MGADL=myasthenia gravis-Activities of Daily Living; MGFA=Myasthenia Gravis Foundation of America; MRI=magnetic resonance imaging; PEOT=premature end of treatment;

PK=pharmacokinetics; PR=pulse rate; RNA=ribonucleic acid; QMG=Quantitative Myasthenia Gravis;

SFEMG=single fiber electromyogram; TB=tuberculosis; UV=Unscheduled Visit

a Subjects will return to the clinic for Visits 15, 16, and 18; for Visits 17, 19, and 20, subjects with either return to the clinic/hospital, or, if possible and agreed by the investigator and subject, have home visits conducted by certified healthcare professionals.

b This visit is a telephone contact 24 hours post-IMP dose start.

c Subjects who withdraw early will be encouraged to complete the PEOT Visit plus the FV (approximately 8 weeks after the final study drug administration).

e Includes consent for SFEMG for the subjects consenting to this measurement at the participating sites. Additional informed consent is needed for participation in the exploratory genomic substudy.


- f Systolic and diastolic BP, pulse rate, temperature, and respiratory rate. On dosing days, vital signs will be measured prior to IMP administration, 15 minutes after the start of the infusion, at the end of the infusion, 2 hours after the end of infusion and 4 hours after the end of the infusion. At nondosing visits, vital signs need only be taken once during the visit.
- g Body weight at Screening will be used for calculation of dose; height will be assessed only at Screening.
- h In addition to Screening and the FV, a full neurological examination should be performed for any subject who experiences severe headache.
- j ECGs will be read by a central reader.
- Pre- and postdose at Visits 2, 4, 6, 9, 11, and 13; postdose samples are to be taken 4 hours after the infusion has ended.
- <sup>j</sup> Blood sample to be taken prior to dosing of IMP.
- n Urine pregnancy test will be performed using a dipstick test; a positive urine pregnancy test must be confirmed using a serum pregnancy test.
- <sup>1</sup> Serum safety biomarkers levels measured at Baseline for all subjects and during follow up only in subjects with severe headache or moderate to severe GI disturbances.
- q At Baseline and subsequently only in subjects with infusion reaction.
- <sup>n</sup> Subjects must be off pyridostigmine (or any inhibitor medication) from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study.
- t For subjects consenting to this measurement at the participating sites; subjects should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study.
- u This assessment is applicable only to subjects experiencing severe headaches and will be performed daily until resolution (ie, if headache becomes moderate or mild, normal collection of AEs should apply); this assessment will be followed by a neurological assessment (including fundoscopy). Additionally, other diagnostic procedures including but not limited to CT scan, MRI and/or LP for CSF collection to be performed if indicated at the discretion of the investigator.
- v Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally.

# Has been changed to:

Table 5.1: Schedule of assessments

| Assessments | Screen | ning | Trea | tment I | Period | l | | | | | | | | | | Obs | serva | tion Ę | Period | ı <sup>a</sup> | | UV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ng Perio | od 1 | | | | | Dos | ing Per | riod 2 | | | | | | :101 | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 17 | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> (± 2 days) | 9 | 15 <sup>d</sup><br>(± 2<br>days) | 16 | 22 <sup>d</sup> (± 2 days) | 29 <sup>d</sup><br>(± 2<br>days) | 30 | 36 <sup>d</sup><br>(± 2<br>days) | 37 | 43 <sup>d</sup><br>(± 2<br>days) | 440 | 50 | 57<br>(± 2 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| Written informed | consent | X | | | days) | | uuy 5) | | | au y s ) | R7 | days) | Olics | | | | | | | | | |
| Written informed for genomic subs | | X | | | | | | | .45 | 5 | ( | 200 | R | | | | | | | | | |
| Demographic dat | a | X | | | | | | | ~C) * | | :12 | | | | | | | | | | | |
| Verification of in<br>/exclusion criteria | | X | X | | | | | 2 | Dr | Jilly | ), | | | | | | | | | | | |
| Call or enter IRT register the visit | to | X | | | X | | X | | eting | | | X | | X | | | | | | | X | |
| Call or enter IRT | / | | X | | | | | 7 | diff | X | | | | | | | | | | | | |
| Withdrawal criter | ria | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| General medical/<br>procedures histor | | X | | | | 100 | 300 | | | | | | | | | | | | | | | |
| Prior and concommedication | nitant | X | X | X | ÝQ c | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant med | lical | | X | SIZE | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Vital signs <sup>f</sup> | | X | X | | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Body weight, hei | ght <sup>g</sup> | X OF | | | | | | | | X | | | | | | | | | | | X | |

Table 5.1: Schedule of assessments

| Clinical Study P | rotocol | | | | | | | | UCF | 37665 | 5 | | | | | | | | DB nical Study Protocol UCB7665 UCB7665 UCB7665 UCB7665 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | Sche | nedule of assessments | | | | | | | | | | | | | | | | | | | | |
| Assessments | Screen | ning | Trea | Treatment Period | | | | | | | | | | | | | | tion F | eriod | l <sup>a</sup> | 7 | UV |
| | | | Dosing Period 1 | | | | | | | Dos | ing Pe | riod 2 | | | | | | | O | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 15 | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> | 9 | 15 <sup>d</sup> | 16 | 22 <sup>d</sup> | 29 <sup>d</sup> | 30 | 36 <sup>d</sup> | 37 | 43 <sup>d</sup> | 44 | 50 | 57 | 64 | 78 | 92 | 99 | |
| | | | | | (± 2 days) | | (± 2<br>days) | | (± 2 days) | (± 2<br>days) | ) | (± 2<br>days) | | (± 2<br>days) | 200 | | (± 2 | days) | | | (± 2 days) | |
| Recording of AEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Full physical examination | | X | | | | | | | | | 5 | | JICS. | 70. | | | | | | | X | |
| Brief physical examination | | | X | | | | | | .< | XC | ) , | 1000 | 56, | | | | | | | | | |
| Full neurological examination h | | X | | | | | | | ACTIO | | 1231 | | | | | | | | | | X | |
| Brief neurological examination | | | X | | | | | 4 | , | J.XC | | | | | | | | | | | | |
| Query for suicidal | ity <sup>i</sup> | X | X | | X | | X | | X ill | X | | X | | X | | X | X | X | X | X | X | X |
| 12-lead ECG <sup>j</sup> | | X | X | | X | | X | 2 | X | X | | X | | X | | X | | | X | | X | |
| Laboratory tests<br>(hematology, chen<br>urinalysis) | mistry, | X | X | | X | | X | 4 | X | X | | X | | X | | X | X | | X | | X | |
| Serology testing for Hepatitis B, and H | | X | | | ×0 | 7166 | | | | | | | | | | | | | | | | |
| IGRA tuberculosis | s test <sup>k</sup> | X | | 50 | ) | | | | | | | | | | | | | | | | | |
| Tuberculosis Sign<br>Symptoms question | s and<br>onnaire | X | 10 | S | | | | | | | | | | | | | | | | | X | |
| Blood sampling fo | or PK | car. | X | | X | | X | | X | X | | X | | X | | X | | | | | | |

Table 5.1: Schedule of assessments

| UCB<br>Clinical Study P | rotocol | | | | | | | | UCE | 3766 | 5 | | | | | | | | | | Neigh | Sep 20<br>MG00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | ole 5.1: Schedule of assessments | | | | | | | | | | | | | | ijons it. | | | | | | | |
| Assessments | Screen | Screening | | Treatment Period | | | | | | | | | | | | | | | Observation Period <sup>a</sup> | | | |
| | | | Dosing Period 1 | | | | | | | | ing Per | | | | | , or | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 15 | 18 | 19 | FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup><br>(± 2<br>days) | 9 | 15 <sup>d</sup><br>(± 2<br>days) | 16 | (± 2 days) | 29 <sup>d</sup><br>(± 2<br>days) | | 36 <sup>d</sup><br>(± 2<br>days) | | 43 <sup>d</sup><br>(± 2<br>days) | 44 | 50 | 57<br>(± 2 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| Blood sampling for DNA analysis sub-study <sup>m</sup> | | | X | | , , | | , | | X | , | | • / | | X | D. C. | | | | | | | |
| Blood sampling for RNA analysis sub-study | | | X | | X | | | | X | | RT | 3, | Splice | X | | | | | | | Х | |
| Serum pregnancy test | | X | | | | | | | | ) | J. | 50 | | | | | | | | | | |
| Urine pregnancy test <sup>n</sup> | | | X | | X | | X | | X | X | :130 | X | | X | | X | X | X | X | X | X | |
| Administration of | IMP | | Х | | X | | X | < | Ok | X | ), | X | | X | | | | | | | | |
| | | | X | | X | | X | 4 | X | X | | X | | X | | X | X | X | X | X | X | |
| Serum complement<br>(C3,C4) and plasma<br>complement levels (C3a<br>and C5a) | | | X | | X | | x | 40 | X.O. | X | | X | | Х | | X | X | | | | х | |
| Immunoglobulins (total<br>IgG and IgG subclasses) | | X | X | | X | ,O | X | | X | X | | X | | X | | X | X | X | X | X | X | |
| IgA, IgM, IgE | | | X | | C | 24 | | | X | X | | X | | X | | X | X | | | | X | |
| MG-specific autoantibodies | | | X | O. | X | | | | | X | | X | | | | X | | | | | X | |

Table 5.1: Schedule of assessments

| UCB<br>Clinical Study Pr | rotocol | | | | | | | | UCE | 3766 | 5 | | | | | | | | | | "Vell | Sep 201<br>MG000 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | 5.1: Schedule of assessments | | | | | | | | | | | | | | tions | | | | | | | |
| Assessments | Screen | ing | Treatment Period | | | | | | | | | | | | | | Observation Period <sup>a</sup> | | | | | |
| | | | Dosing Period 1 | | | | | | | Dosing Period 2 | | | | | | | | | O | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 15/6 | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup> | 9 | 15 <sup>d</sup> | 16 | 22 <sup>d</sup> | 29 <sup>d</sup> | 30 | 36 <sup>d</sup> | 37 | 43 <sup>d</sup> | 44 | 50 | 57 | 64 | 78 | 92 | 99 | |
| | | | | | (± 2<br>days) | | (± 2<br>days) | ) | (± 2 days) | (± 2<br>days) | | (± 2<br>days) | | (± 2<br>days) | 200 | | (± 2 days) | | | | (± 2 days) | |
| Blood sampling for<br>exploratory biomarker<br>analysis | | | X | | X | | X | | Х | X | 1 | X | Ö. | X | | | | X | | X | | |
| Blood sampling for<br>safety biomarker<br>analysis: may include but<br>not limited to | | | X | | X | | X | 2 | X | XC | )<br>3112 <sup>119</sup> | X | | X | | X | X | X | X | X | X | |
| BAFF analysis | | | X | | X | | X | | x iin | X | | X | | X | | | | X | | X | | |
| Cytokines <sup>p</sup> | | | X | | X | | X | | 3.3X | X | | X | | X | | X | X | X | X | X | X | X |
| Vaccination-specific antibody titers ( | | X | | | | | N. O. | 7 | | | | | | | | | | | | | X | |
| MG-composite scale | | X | X | | X | ,00 | X | | X | х | | X | | X | | X | X | X | X | х | Х | |
| QMG scale <sup>q</sup> | | X | Х | | XC | 5 | X | | X | Х | | X | | X | | X | X | | X | | X | |
| Muscle weakness<br>severity and fatigat<br>scale | bility | | X | eused | X | | X | | х | X | | X | | X | | X | X | X | X | X | X | |
| Fatigue scale | | | X. | | X | | X | | X | Х | | X | | X | | X | X | X | Х | X | Х | |
| MGADL scale | | 20 | X | | | | | | | Х | | | | | | X | | X | | | X | |
### **Table 5.1:** Schedule of assessments

| Assessments | Assessments Screening | | | | Period | | | | | | | | | | | Observation Period <sup>a</sup> | | | | | | UV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosing Period 1 | | | | | | | Dosing Period 2 | | | | | | O'S | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | Pa | 18 | 19 | 20<br>FV/PEOT | |
| Da | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> (± 2 days) | | 15 <sup>d</sup><br>(± 2<br>days) | | (± 2 days) | 29 <sup>d</sup> 3<br>(± 2<br>days) | 30 | 36 <sup>d</sup><br>(± 2<br>days) | , | 43 <sup>d</sup><br>(± 2<br>days) | 44 | 50 57 (± 2 | | 64 78 days) | | 92 | 99<br>(± 2 days) | |
| MGFA classificati | on | X | X | | | | | | | X | | | | 20 | 2, | | | | | | X | |
| SFEMG measuren | nent <sup>r</sup> | | X | | | | | | | X | 7 | | | 10 | | | | | | | | |
| Headache question | nnaire <sup>s</sup> | | X | X | X | X | X | X | X | XC | X | X | ZX/ | X | X | X | X | X | X | X | X | X |
| Stool sample asses | ssment <sup>t</sup> | | X | | X | | X | | X | X | .:.( | X. | | X | | X | X | X | X | X | X | X |
| Subject exit interv | iew | | | | | | | | G | | :120 | | | | | | | | | | X | |

AE=adverse event; BAFF=B-cell activating factor; BL=Baseline; BP=blood pressure; CSF=cerebrospinal fluid; CT=computed tomography; DNA=deoxyribonucleic acid; ECG=electrocardiogram; FV=Final Visit; GI=gastrointestinal; HIV=human immunodeficiency virus; IgA=immunoglobulin A; IgE=immunoglobulin E; IgG=immunoglobulin G; IGRA= interferon-gamma release assay; IgM=immunoglobulin M; IMP=investigational medicinal product; IRT=interactive response technology; LP=lumbar puncture; MG=myasthenia gravis; MGADL=myasthenia gravis-Activities of Daily Living; MGFA=Myasthenia Gravis Foundation of America; MRI=magnetic resonance imaging; PEOT=premature end of treatment; PK=pharmacokinetics; PR=pulse rate; RNA=ribonucleic acid; QMG=Quantitative Myasthenia Gravis;

SFEMG=single fiber electromyogram; TB=tuberculosis; UV=Unscheduled Visit

<sup>b</sup> This visit is a telephone contact 24 hours post-IMP dose start?


<sup>&</sup>lt;sup>a</sup> Subjects will return to the clinic/hospital for Visits 15, 16, 18, and 20; for Visits 17 and 19 subjects will either return to the clinic/hospital, or, if possible and agreed by both the investigator and subject, have home visits conducted by certified healthcare professionals.

<sup>&</sup>lt;sup>c</sup> Subjects who withdraw early will be encouraged to complete the PEOT Visit plus the FV (approximately 8 weeks after the final study drug administration).

d A visit window of ±2 days is allowed for the dosing visits. The visit window of ±2 days is relative to the first dosing visit date. However, there should be a minimum interval of 5 days and maximum interval of 9 days as compared to the previous dose.

e Includes consent for SFEMG for the subjects consenting to this measurement at the participating sites. Additional informed consent is needed for participation

in the exploratory genomic substudy.

f Systolic and diastolic BP, pulse rate, temperature, and respiratory rate. On dosing days, vital signs will be measured prior to IMP administration, 15 minutes after the start of the infusion, at the end of the infusion, 2 hours after the end of infusion and 4 hours after the end of the infusion. At nondosing visits, vital signs need only be taken once during the visit.

<sup>&</sup>lt;sup>g</sup> Body weight at Screening and at Visit 9 will be used for calculation of dose; height will be assessed only at Screening.

h In addition to Screening and the FV, a full neurological examination should be performed for any subject who experiences severe headache.

- Subjects must be off pyridostigmine (or any standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last any inhibitor dosing for each evaluation during the study.
- For subjects consenting to this measurement at the participating sites; subjects should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. If pyridostigmine is taken, the time must be documented.
- <sup>u</sup> This assessment is applicable only to subjects experiencing severe headaches and will be performed daily until resolution (ie, if headache becomes moderate or mild, normal collection of AEs should apply); this assessment will be followed by a neurological assessment (including fundoscopy). Additionally, other diagnostic procedures including but not limited to CT scan, MRI and/or LP for CSF collection to be performed if indicated at the discretion of the investigator.
- V Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally.

A query for suicidal ideation will be asked by Investigator at each clinical visit (including Visit 17 or Visit 19 when it is conducted at the clinic). A full C-SSRS assessment will be performed only when subject has a positive response to the suicidal ideation query. If a subject has active suicidal ideation as confirmed by the answer 'Yes' to Question 4 or Question 5 of the C-SSRS assessments, the subject will be excluded or withdrawn from the study and immediately referred to a Mental Healthcare Professional

<sup>&</sup>lt;sup>j</sup> ECGs will be read by a central reader.

k The IGRA test will be performed in a central laboratory. Subject should not be dosed until IGRA result is available and negative.

Pre- and postdose at Visits 2, 4, 6, 9, 11, and 13; postdose samples are to be taken 4 hours after the infusion has ended.

<sup>&</sup>lt;sup>m</sup> Blood sample to be taken prior to dosing of IMP.

<sup>&</sup>lt;sup>n</sup> Urine pregnancy test will be performed using a dipstick test; a positive urine pregnancy test must be confirmed using a serum pregnancy test.

<sup>&</sup>lt;sup>p</sup> Sampling for exploratory safety biomarkers at Baseline (Visit 2) and 4 hours post dosing (Visit 2) for all subjects. During follow up only in subjects with severe headache and/or moderate to severe GI disturbances.

<sup>&</sup>lt;sup>q</sup> Sampling at Baseline for all subjects and subsequently only in subjects with infusion reaction.

### 5.4.1 Choice of study design and endpoints

The primary objective of the study is to evaluate the clinical efficacy of UCB7665 as an ondemand treatment for subjects with moderate to severe generalized MG.

During the first Treatment Period a 2-arm parallel design study will allow comparison of the change from Baseline in QMG score to Visit 9 (Day 29) between IMP and placebo.

The choice of the primary outcome measures and the timing of approximately 4 weeks after the first dose of study drug are predicted to be the optimal approach to measure improvements based on effect seen in other therapies and recommendations of the Scientific Advisory Board of the MGFA (Barth 2013; Benatar 2012; Howard 2013). Then the second Dosing Period with a rerandomization allows for additional supportive data to be evaluated as well as minimizes the need for prolonged exposure of some subjects to placebo.

### Has been changed to:

### 5.4.1 Choice of study design and endpoints

The primary objective of the study is to evaluate the clinical efficacy of UCB7665 as a chronic-intermittent treatment for subjects with moderate to severe generalized MG. Additionally, this study will provide data for future study planning, whether for chronic-intermittent treatment or a longer therapy option by evaluating the general concept that UCB7665 has a clinical effect in patients with generalized MG.

During the first Treatment Period, a 2-arm parallel design study will allow comparison of the change from Baseline in QMG score to Visit 9 (Day 29) between UCB7665 7mg/kg and placebo.

The choice of the primary efficacy outcome measures and the timing of approximately 4 weeks after the first dose of study drug are predicted to be the optimal approach to measure improvements based on effect seen in other therapies and recommendations of the Scientific Advisory Board of the MGFA (Barth 2013; Benatar 2012; Howard 2013). Then the second Dosing Period with a rerandomization allows for additional supportive data to be evaluated as well as offering the placebo subjects a chance to receive UCB7665.

### Change #17

6.1 Inclusion criteria

The following inclusion criterion was amended.

6. Female subjects of child bearing potential must have a negative serum pregnancy test at the Screening Visit, which is confirmed to be negative by urine testing prior to the first dose of study drug at Week 1 (Visit 2) and prior to further dosing at each study visit thereafter.

Female subjects of childbearing potential must agree to use a highly effective method of birth control, during the study and for a period 2 months after their final dose of study drug. Highly effective forms of birth control are methods which achieve a failure rate of less than 1% per year when used consistently and correctly. Highly effective methods of birth control include:

- 6.1 Inclusion criteria
- 6. Female subjects of child bearing potential must have a negative serum pregnancy test at the Screening Visit, which is confirmed to be negative by urine testing prior to the first dose of study drug at Week 1 (Visit 2) and prior to further dosing at each study visit thereafter.

Female subjects of childbearing potential must agree to use a highly effective method of birth control, during the study and for a period 2 months after their final dose of study drug. According to the International Council for Harmonisation (ICH) M3 (R2), highly effective & forms of birth control are methods which achieve a failure rate of less than 1% per year when used consistently and correctly. Highly effective methods of birth control include:

### Change #18

The following exclusion criteria were amended.

- 6.2.1 Exclusion criteria related to health status
- 7. Subject has QMG score of <10.5 at Baseline.
- 12. Subject has 12-lead ECG with changes considered to be clinically significant upon medical review.
- 15. Subject has >1.5x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (>1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%).

For randomized subjects with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin but <1.5xULN, a Baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report form (eCRF).

If subject has >ULN, ALT, AST, or ALP that does not meet the exclusion limit at Screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the subject must be discussed with the medical monitor.

Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit (>1.5xULN) may be repeated once for confirmation. This includes rescreening.

- 21. Subject has a history of clinically relevant ongoing chronic infections including but not limited to human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C, active or latent 22. Subject has a family history of primary immunodeficiency. tuberculosis (TB) or who tests positive for HIV, Hepatitis B, or Hepatitis C at the Screening

- 6.2.1 Exclusion criteria related to health status
- 7. Subject has QMG score of <11 at Baseline.
- abnormality. The clinical significance of the findings needs to be assessed by the investigator to determine eligibility as defined by the protocol, and any queries regarding continuation of the subject must be addressed with the medical monitor.

  Subject has >2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALT) >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert) elevations only in total bilirubin that 12. Subject has 12-lead ECG with changes considered to be clinically significant upon medical
- 15. Subject has >2x upper limit of normal (ULN) of any of the following: alanine identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%)?

For randomized subjects with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin but <1.5xULN, a Baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report form (eCRF).

If subject has >ULN, ALT, AST, or ALP that does not meet the exclusion limit at Screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the subject must be discussed with the medical monitor.

Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit (>2xULN) may be repeated once for confirmation. This includes rescreening.

- 21. Subject has a history of clinically relevant ongoing chronic infections including but not limited to human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C, or who tests positive for HIV, Hepatitis B, or Hepatitis C at the Screening Visit.
- 22. Subject has a family history (immediate family member) of primary immunodeficiency.

### Change #19

The following exclusion criteria were amended. Exclusion criterion #29 was deleted.

- 6.2.2 Exclusion criteria related to concomitant medications/procedures
- 27. Subject has had prior treatment with rituximab in the 6 months prior to the Baseline Visit or subject has had prior treatment with rituximab in the 12 months prior to Baseline and B cells are not within the normal range.
- 28. Subject has not completed the washout period for the immunosuppressants, biologics, and other therapies as detailed in Table 6.1.
- 29. Subjects receiving immunoadsorption treatment.
- 30. Subject had a thymectomy in the past 6 months, a history of thymoma World Health Organization grade B2 or B3, or Masaoka grade III or IV, or thymoma requiring chemotherapy and/or radiotherapy.

- 6.2.2 Exclusion criteria related to concomitant medications/procedures
- 27. Subject has had prior treatment with rituximab in the 6 months prior to the Baseline Visit or

- Exclusion Criterion 29 was deleted per Protocol Amendment 1.

  30. Subject had a thymectomy in the past 6 months, a history of thymoma World Health Organization grade B2 or B3, or Masaoka grade III or IV, or history of a thymoma requirement and/or radiotherapy.

  Change #20

  [Table 6.1: Washout periods for insertion of the past of

| Generic name (commercial/trade names) | Washout Period relative to Baseline Visit (regardless of route) |
|---|---|
| Others | CO, SO |
| Intravenous immunoglobulin | |

### Has been changed to:

Table 6.1: No treatment periods for exclusionary immunosuppressants, biologics, and other therapies

| Generic name (commercial/trade names) | Period relative to Baseline Visit (regardless of route) |
|---|---|
| Others | |
| Intravenous or subcutaneous immunoglobulin | |

### Change #21

The below section was added:

- 6.2.3 Exclusion criteria related to other risks
- 31 Subject has a lifetime history of suicide attempt (including an or has suicidal ideation in the past 6 months as indicated by a positive response (Yes) to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening.
- Subjects with known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent tuberculosis infection (LTBI), or current/history of nontuberculous mycobacterial infection (NTMBI) are excluded.

- a. Known TB infection whether present or past is defined as:
- Active TB infection or clinical signs and symptoms suggestive of TB (pulmonary or extrapulmonary).
- History of active TB infection involving any organ system or findings in other organ systems consistent with TB infection.
- Any historical evidence by radiography or other imaging modalities consistent with previously active TB infection.
- b. High risk of acquiring TB infection is defined as:
- Known exposure to another person with active TB infection within the 3 months prior to Screening.
- Time spent in a healthcare delivery setting or institution where individuals infected with TB are housed and where the risk of transmission of infection is high.
- c. LTBI (see Section 12.3.1 for further details and instructions).
- d. NTMBI is defined as a group of lung infections caused by mycobacteria different from mycobacterium tuberculosis infections.

6.3 Rescreening and Rechecking

Subjects with isolated results that are outside the specified ranges and that are deemed potentially clinically nonsignificant will be allowed to rescreen at the discretion of the investigator, following discussion with the sponsor's medical monitor/study physician, if appropriate.

If a subject has 1 isolated test result outside the specific range which is deemed clinically significant, the abnormal value may be rechecked at the discretion of the investigator, following discussion with the sponsor's medical monitor/study physician. If the normalization of the test result occurs within the Screening Period, then no other Screening procedures need to be repeated.

## Has been changed to:

Subjects with isolated results that are outside the specified ranges and that are deemed potentially clinically significant will be allowed to rescreen at the discretion of the investigator, following discussion with the sponsor's medical monitor/study physician, if appropriate.

If a subject has 1 isolated test result outside the specific range which is deemed clinically nonsignificant, the abnormal value may be rechecked at the discretion of the investigator, following discussion with the sponsor's medical monitor/study physician. If the normalization of the test result occurs within the Screening Period, then no other Screening procedures need to be repeated.

6.4 Withdrawal criteria

Subjects MUST be withdrawn from IMP if any of the following events occur:

1. Subject develops an illness or has a change in health status that would interfere with his/her continued participation, including but not limited to:

The below was added:

- Subject has a TB test that is confirmed positive or any further evidence suggestive of potential TB infection (eg, exposure) and further examinations result in a diagnosis of active TB or LTBI (refer to Section 12.3.1) for further details and instructions.

  If an NTMBI is identified during a study, the same withdrawal for an active TB infection identified during a study, the below with the same withdrawal for an active TB infection identified during a study.
- If an NTMBI is identified during a study, the same withdrawal procedures as those used

Additionally, the below was added:

8. Subject has active suicidal ideation as indicated by a positive response (Yes) to either Question 4 or Question 5 of the "Since Last Visit" version of the C-SSRS. The subject should be referred immediately to a Mental Healthcare Professional.

### Change #24

Permitted concomitant medication 7.8.1

The following was added:

Subjects should not take pyridostigmine (or any inhibitor medication) from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last or any inhibitor medication inhibitor dosing for each evaluation during the study.

### Change #25

- 7.8.2 Prohibited concomitant treatments (medications and therapies)
- Dexamethasone

3<sup>rd</sup> paragraph:

If a subject needs or takes any prohibited medication or therapy (except IVIg, PLEX, dexamethasone or rituximab), the investigator will (where possible) discuss with the sponsor study physician and a decision will be made whether the subject can continue in the study or must be withdrawn. If the subject is treated with IVIg, rituximab, or PLEX, the subject must be withdrawn from the IMP, but should be encouraged to continue with Observation Period Visits.

## Has been changed to:

7.8.2 Prohibited concomitant treatments (medications and therapies)

Dexamethasone was removed from the bullet list and the following text.

### 3<sup>rd</sup> paragraph:

If a subject needs or takes any prohibited medication or therapy (except IVIg, PLEX, or rituximab), the investigator will (where possible) discuss with the sponsor study physician and a decision will be made whether the subject can continue in the study or must be withdrawn. If the subject is treated with IVIg, rituximab, or PLEX, the subject must be withdrawn from the IMP, but should be encouraged to continue with Observation Period Visits.

### Change #26

- 8.1.1 Visit 1 (Day -28 to -1) Screening Visit
- Blood sample for the following laboratory parameters:
  - Standard safety laboratory tests: hematology and clinical chemistry, plus serology testing for HIV. Hopetitis P. Harvetitis C. 1 for HIV, Hepatitis B, Hepatitis C, and active or latent TB

### Has been changed to:

- 8.1.1 Visit 1 (Day -28 to -1) Screening Visit
- Blood samples:
  - Standard safety laboratory tests: hematology and clinical chemistry, plus serology testing for HIV, Hepatitis B, and Hepatitis C

Additionally, the following were added:

- Query for suicidality (Screening) If positive response (Yes), a full C-SSRS will be performed.
- Tuberculosis assessments:
  - IGRA
  - Tuberculosis Sign and Symptoms questionnaire

### Change #27

The following laboratory parameters were updated.

- 8.2.1 Visit 2 (Day 1, Baseline)
- Blood sample for the following laboratory parameters:
  - IgG depletion assay
- only in subjects with severe headache and Cytokines (only in subjects with infusion reaction) only in subjects with severe headache and/or moderate to severe GI disturbance

- 8.2.1 Visit 2 (Day 1, Baseline)
- Blood samples:
  - Exploratory biomarker analysis
  - Exploratory safety biomarkers: may include but not limited to
  - Cytokines

In addition, the following were added:

- Tuberculosis Sign and Symptoms questionnaire
- Query for suicidality (Screening) If positive response (Yes), a full C-SSRS will be performed.

### Change #28

3 any extensions or variations thereof. The following changes were made in Section 8.2.3, 8.2.5, 8.2.7, 8.3.1, 8.3.3, 8.3.5, 8.4.3, and 8.4.5.

- Blood sample for the following laboratory parameters:
  - IgG depletion assay
  - Safety biomarkers: in subjects with severe headache and/or moderate to severe GI disturbance

### Has been changed to:

- Blood samples:
  - Exploratory biomarker analysis
  - Exploratory safety biomarkers: may include but not limited to

in subjects with

severe headache and/or moderate to severe GI disturbance

In addition, the following was added:

Query for suicidality (since last visit): If positive response (Yes), a full C-SSRS will be performed.

### Change #29

The following changes were made in Section 8.4.1, 8.4.2, 8.4.4, and 8.4.6.

- Blood sample for the following laboratory parameters:
  - IgG depletion assay
  - Exploratory safety biomarkers: only in subjects with severe headache and/or moderate to severe GI disturbance

Blood samples:

UCB

Exploratory safety biomarkers: may include but not limited to

extensions or variations thereof.

severe headache and/or moderate to severe GI disturbance

In addition, the following was added:

Query for suicidality (since last visit): If positive response (Yes), a full C-SSRS will be performed.

The following was added into Section 8.4.6 only:

Tuberculosis Sign and Symptoms questionnaire

### Change #30

The following sentence was deleted in Section 8.2.2, 8.2.4, 8.2.6, 8.3.2, 8.3.4, and 8.3.6.

The following item was deleted in Section 8.2.7 and 8.4.1 to 8.4.6.

• Call or enter IRT to register the visit

Change #32

8.4 Observation Period

During the Observation Period, visits will be part.

Visits 17, 18, and 19 urber. During the Observation Period, visits will be performed at weekly intervals, apart from between Visits 17, 18, and 19, when visits will be performed at 2 weekly intervals. Subjects will return to the clinic for Visits 15, 16, and 18 for efficacy and for safety assessments. Subjects will either return to the clinic, or, if possible and agreed by both the investigator and the subject, have home visits conducted by certified healthcare professionals, for Visits 17, 19, and 20. No IMP will be administered in the Observation Period.

### Has been changed to:

8.4 Observation Period

During the Observation Period, visits will be performed at weekly intervals, apart from between Visits 17, 18, and 19, when visits will be performed at 2 weekly intervals. Subjects will return to the clinic for Visits 15, 16, 18, and 20 for efficacy and for safety assessments. Subjects will either return to the clinic, or, if possible and agreed by both the investigator and the subject, have home visits conducted by certified healthcare professionals, for Visits 17 and 19. No IMP will be administered in the Observation Period.

8.6 Unscheduled Visit

The following was added:

Query for suicidality (since last visit): If positive response (Yes), a full C-SSRS will be performed.

### Change #34

9.5 Single Fiber EMG, 1<sup>st</sup> paragraph:

At participating sites, subjects consenting to SFEMG measurement should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. [...]

### Has been changed to:

9.5 Single Fiber EMG, 1<sup>st</sup> paragraph:

At participating sites, subjects consenting to SFEMG measurement should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing. but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. If pyridostigmine is taken, the time must be documented.

### Change #35

10.2 Pharmacodynamic variables

The following was deleted:

• IgG concentrations pre- and postdepletion

## Change #36

Immediate reporting of adverse events 12.1.1.5

The following AEs must be reported immediately using the Serious Adverse Event form:

- SAE: AE that the investigator classifies as serious by the above definitions regardless of causality
- Suspected transmission of an infectious agent via a medicinal product
- AE of special interest (see Section 12.1.1.3)
- AE of interest (see Section 12.1.1.4)

### Immediate reporting of adverse events 12.1.1.5

and any extensions or variations thereof. The following AEs must be reported immediately using the SAE Report Form according to the procedure in Section 12.1.2.3:

- SAE: AE that the investigator classifies as serious by the above definitions regardless of causality
- Suspected transmission of an infectious agent via a medicinal product
- AE of special interest (see Section 12.1.1.3)
- AE of interest (see Section 12.1.1.4)
- Confirmed LTBI, active TB, and NTMBI (see Section 12.3.1)

### Change #37

The following was added to clarify the suicidality assessment:

### 12.1.6 Suicidality

At screening, the Investigator will query each subject if he/she has a lifetime history of suicide or suicidal ideation attempt (including an in the past 6 months. A full C-SSRS "Lifetime recent" assessment will be performed only when the subject has a positive response to this query. This scale will be assessed by trained study personnel. When suicide attempt or suicidal ideation is confirmed by a positive response (Yes) to either Question 4 or Question 5 of the C-SSRS, the subject must be excluded and immediately referred to a Mental Healthcare Professional.

At each clinical visit, the investigator must query the suicidal ideation since the last visit. A full C-SSRS "Since last visit" assessment will be performed only when the subject has a positive response to this query. When suicide attempt or suicidal ideation is confirmed by a positive response (Yes) to either Question 4 or Question 5 of the C-SSRS, the subject must be withdrawn and immediately referred to a Mental Healthcare Professional. The details of C-SSRS will be provided in the Study Procedures Manual.

### Change #38

12.1.7 Safety signal detection, 1st paragraph

An unblinded DMC will oversee at least 1 interim analysis during the course of the study during which the safety and futility of UCB7665 will be assessed.

## Has been changed to:

12.1.7 Safety signal detection, 1<sup>st</sup> paragraph

which the safety of UCB7665 will be assessed. An unblinded DMC will oversee at least 1 interim analysis during the course of the study during

MG0002

### Change #39

Clinical Study Protocol

**UCB** 

Assessment of safety biomarkers was clarified.

12.1.10 Management of moderate or severe diarrhea (previous heading number), 2<sup>nd</sup> paragraph

ions of variations thereof. Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally. In addition, assessment of safety biomarkers is required for subjects with moderate to severe GI disturbances including

Management of moderate or severe diarrhea (new heading number), 2<sup>nd</sup> paragraph

moderate or severe diarrhea

alysis will be performed for subject aley of stool sampling will be as clinic, all be as clinic, along the samples will be performed to assment of exploratory safety biomarkers is redisturbances including diarrhea.

pe#40

Laboratory measurements, Table 12.2

Duplicate laboratory tests were removed and footnotes are updated. Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally. In addition, collection of blood samples for assessment of exploratory safety biomarkers is required for subjects with moderate

Table 12.2: Safety laboratory measurements

| Hematology | Chemistry | Urinalysis | Pregnancy test |
|---|---|---|---|
| Hematocrit | Calcium | Albumin | Urine HCG |
| Hemoglobin | Chloride | Protein | Serum HCG <sup>a</sup> |
| Platelet count | Magnesium | Nitrite | |
| RBC count | Electrolytes (calcium, | Glucose | |
| WBC count (including differential) | phosphate, sodium,<br>potassium, chloride, and<br>magnesium) | рН | Nextensions of vo |
| | Phosphate | Protein | ete |
| | ALP | Leukocytes | You. |
| HbA1c <sup>b</sup> | AST | Blood | |
| Hemoglobin (RBC and platelet count) | ALT | Bilirubin dilo | |
| Hematocrit | GGT | Urobilinogen | |
| Serology <sup>c</sup> | Total and direct bilirubin | Ketone | |
| HBsAg | LDH | Creatinine | |
| HCV Ab | Total cholesterol | Glucose | |
| HIV (anti-HIV1 or<br>anti-HIV2<br>antibodies) | LDL - cholesterol | Albumin | |
| Tuberculosis <sup>d</sup> | HDIO cholesterol, triglycerides | | |
| | Amylase | | |
| Serum biomarkers | Creatine kinase | | |
| | Creatinine | | |
| | Total protein | | |
| | Albumin | | |
| | alpha- and beta–<br>globulins | | |

### Table 12.2: Safety laboratory measurements

| Hematology | Chemistry | Urinalysis | Pregnancy test |
|------------|---------------|------------|----------------|
| | Urea-N | | |
| | Procalcitonin | | |
| | hsCRP | | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; FSH=follicle stimulating hormone; GGT=gamma glutamyltransferase; HbA1c=hemoglobin A1c; HBsAG=hepatitis B surface antigen; HCG=human chorionic gonadotropin; HCV Ab=hepatitis C virus antibody; HDL=high density lipoprotein; HIV=human immunodeficiency virus; hsCRP=high-sensitivity C-reactive protein; LDH=lactate dehydrogenase;

LDL=low density lipoprotein;

; RBC=red blood cell; WBC=white blood cell

Serum pregnancy testing is only performed at Visit 1 and, in the event of a positive pregnancy test to confirm the results of a urine test

HbA1c is performed at Screening only

and at each schedul a for moderate to severy the control of the co Serum biomarkers levels measured at Screening, Baseline, and at each scheduled assessment during Treatment and Observation Periods in subjects with severe headache and/or moderate to severe GI disturbance


| Hematology | Chemistry | Urinalysis | Pregnancy test |
|---|---|---|---|
| Hematocrit | Electrolytes (calcium, | Albumin | Urine HCG |
| Hemoglobin | phosphate, sodium, potassium, chloride, | Protein | Serum HCG <sup>a</sup> |
| Platelet count | and magnesium) | Nitrite | |
| RBC count | ALP | Glucose | |
| WBC count | AST | рН | 01/10 |
| (including differential) | ALT | Leukocytes | ansions of vall |
| HbA1c <sup>b</sup> | GGT | Blood | tiens |
| | Total and direct | Bilirubin | and of |
| <b>Serology</b> <sup>c</sup> | bilirubin | Urobilinogen | 8 |
| HBsAg | LDH | Ketone | |
| HCV Ab | Total cholesterol | Creatinine | |
| HIV (anti-HIV1 or | LDL - cholesterol | COX 359 | |
| anti-HIV2 antibodies) Tuberculosis <sup>d</sup> | HDL – cholesterol<br>triglycerides | orization | |
| | Amylase | JE! | |
| Exploratory Safety<br>Biomarkers <sup>e</sup> | Creatine kinase | | |
| | Creatinine | | |
| | Total protein | | |
| | Albumin | | |
| | alpha- and beta-<br>globulins | | |
| | Urea-N | | |
| CO. | Procalcitonin | | |
| CEIT. | hsCRP | | |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; GGT=gamma glutamyltransferase; HbA1c=hemoglobin A1c; HBsAG=hepatitis B surface antigen; HCG=human chorionic gonadotropin; HCV Ab=hepatitis C virus antibody; HDL=high density lipoprotein; HIV=human immunodeficiency virus; hsCRP=high-sensitivity C-reactive protein; LDH=lactate dehydrogenase; LDL=low density lipoprotein; RBC=red blood cell; WBC=white blood cell


b HbA1c is performed at Screening only

<sup>c</sup> This serology performed at Screening only

Interferon-gamma release assay by central laboratory.

### Change #41

### 12.2.1.1 Consultation with medical monitor and local hepatologist

Potential drug-induced liver injury events require notification of the medical monitor within 24 hours (eg. by laboratory alert), and the subject must be discussed with the medical monitor as soon as possible. If required, the subject must also be discussed with the local hepatologist.

### Has been changed to:

Potential drug-induced liver injury events require notification of the medical monitor within 24 hours (eg, by laboratory alert), and the subject must be discussed with the medical monitor as soon as possible. If required, the subject must also be discussed with the local hepatologist or gastroenterologist.

Change #42
The below was added:12.3.1 Assessment and management of TB and TB risk factors

With the currently available data, TB is not considered as an important potential or identified risk for treatment with UCB7665. As immunomodulation may carry risk of new or activation of LTBI, UCB has conservatively developed TB detection and management procedures taking into account the most current recommendations of international guidelines (2010 WHO) and most recent literature, covering any infection by the mycobacteria tuberculosis complex.

Appropriate rigorous precautions are being taken within this protocol to monitor the risk of TB infection in this study (see Section 6.3.2 [Exclusion Criterion 32] and Section 6.4 [Withdrawal Criteria 1]). Following are the key considerations of these procedures:

## TB Tests at Screening

IGRA and TB questionnaire are required as indicated in Schedule of Assessments (Table 5.1).

- TB screening is mandatory both before study entry and during the conduct of the study. The preferred screening test is IGRA performed at a Central Laboratory.
  - The IGRA result must be negative for subjects to enroll in this study
  - Subjects who test positive for IGRA test should be excluded from the study and referred for appropriate medical evaluation according to the local medical practice guidelines.
  - If the result of the IGRA test is indeterminate, the particular IGRA test previously performed may be repeated once; if positive or indeterminate on retest, the subject must not be randomized to study drug and, if already randomized, must undergo appropriate

<sup>&</sup>lt;sup>a</sup> Serum pregnancy testing is only performed at Visit 1 and, in the event of a positive pregnancy test, to confirm the results of a urine test

ions of variations thereof May include but not limited to the following biomarkers listed below. Samples collected for exploratory safety biomarkers at Baseline (Visit 2) and 4 hours post dosing (Visit 2) for all subjects and during follow up only in subjects with severe headache and/or moderate to severe GI disturbances. The Baseline samples will only be analysed in case the subject experienced a severe headache and/or moderate to severe GI disturbance.

15 Sep 2017

MG0002

study specified withdrawal procedures. The retest must be done during the protocol-defined Screening Period.

In addition to IGRA test, subjects will be evaluated for signs and symptoms of latent or active TB infection and for risk factors of exposure to TB, using the TB questionnaire, at Screening. See the 'TB signs and symptoms questionnaire' section for further instructions on using the questionnaire. Subjects with known TB, at a high risk of acquiring TB or with LTBI should be excluded from this study as described in Exclusion Criteria.

### Monitoring for TB during the study

Subjects will be monitored for signs/symptoms of TB using routine pharmacovigilance measures for Adverse Events. Subjects reporting AEs related to signs/symptoms of TB will be evaluated for LTBI and active TB according to the local medical practice guidelines.

Subjects with confirmed LTBI or active TB or NTMBI will be immediately withdrawn from the study as described in Withdrawal Criteria, Confirmed LTBI, active TB, and NTMBI must be reported to the Sponsor immediately regardless of seriousness using the SAE Report Form. Additional information received by the Investigator should be provided to the Sponsor within 24 hours of awareness.

Once withdrawn from study treatment, subjects should return for the PEOT, complete all early withdrawal assessments, and complete the follow-up visits.

### TB tests at Final/PEOT Visit

Subjects will be evaluated for signs and symptoms of latent or active TB infection and for risk factors of exposure to TB, using the TB questionnaire, at the Final/PEOT Visit. See the 'TB signs and symptoms questionnaire' section for further instructions on using the questionnaire

### Signs and symptoms of TB

The Investigator should consider all potential sites of infection when assessing for TB during the physical examination, and other evaluations, and based on the subject's history.

Common symptoms with which the subject may present with include cough, blood in sputum, night sweats, lymphadenitis, joint pain/swelling, spinal deformity, headache/confusion, abdominal pain mimicking inflammatory bowel disease, frequent or painful urination, scrotal mass in men and pelvic inflammatory disease in women as well as other symptoms, or nonspecific symptoms. This is not an exhaustive list and unusual presentations should always be considered.

### TB signs and symptoms questionnaire

The questionnaire "Evaluation of signs and symptoms of tuberculosis" should be used as a source document. The questionnaire will assist with the identification of subjects who may require therapy for TB. A subject who answers "Yes" to the question

at Screening is excluded. A "Yes" response to any of the other questions within the questionnaire at Screening should trigger further careful assessment to determine if subject has latent or active TB (see Section 6.2.3 [Exclusion Criterion 32]). A "Yes" response to any of the questions at the end of the study should trigger further assessments as per local medical guidelines to determine if the subject has either LTBI or active TB infection.

### LTBI, active TB or other NMTBI identified during study

During the study, subjects who develop evidence of LTBI or active TB or NMTBI must extensions of variations thereof. immediately stop further administration of study drug and will be referred to an appropriate medical specialist for further evaluation.

Confirmed LTBI or active TB or NTMBI must be reported to the Sponsor immediately as described above.

### Change #43

12.3.6 12-lead ECG

The heading numbering was changed as below:

12.3.7 12-lead ECG

In addition, the below was added:

The investigator may consult with the cardiologist at the central ECG laboratory to confirm the presence of a clinically significant ECG abnormality. It remains the responsibility of the investigator to decide whether an ECG finding is of clinical significance on the basis of the complete clinical picture and whether this finding influences the subject's participation in the study.

### Change #44

14.2

General statistical considerations, 5<sup>th</sup> paragraph stated otherwise 2<sup>11</sup> 5<sup>th</sup> . . . Unless stated otherwise, all statistical tests will be 1-sided and conducted at 0.05 alpha levels. For Dosing Period 2, only descriptive analyses will be performed.

### Has been changed to:

General statistical considerations, 5<sup>th</sup> paragraph 14.2

Unless stated otherwise, all statistical tests will be 1-sided and conducted at 0.05 alpha levels (due to the character of the study, no alpha adjustment for multiplicity will be done). For Dosing Period 2, only descriptive analyses will be performed.

### Change #45

14.3.1 Analysis of the primary efficacy variable, 2<sup>nd</sup> paragraph to the last paragraph

A 1-sided hypothesis test will be performed to test the primary hypothesis of superiority of UCB7665 7mg/kg vs placebo at Visit 9. The null hypothesis is that there is no difference in the change from Baseline between Treatment Groups. The alternative hypothesis is that the mean change from Baseline in QMG score is greater in the UCB7665 7mg/kg group than the placebo group.

The primary efficacy variable will be analyzed for the FAS using an analysis of covariance model with treatment as a factor and Baseline QMG as a covariate. Least Squares (LS) Means For changes from Baseline at Visit 9 for each treatment group will be presented together with LS mean differences (UCB7665 - 7mg/kg vs placebo) and 1-sided 95% confidence interval (CI). Last Observation Carried Forward (LOCF) imputation will be utilized to account for missing data at Visit 9.

The analysis of the primary efficacy variable will repeated for the PPS using the same methodology as described above.

### Has been changed to:

14.3.1 Analysis of the primary efficacy variable, 2<sup>nd</sup> paragraph to the last paragraph

A 1-sided hypothesis test will be performed to test the primary hypothesis of superiority of UCB7665 7mg/kg vs placebo at Visit 9. The null hypothesis is that there is no difference in the change from Baseline between Treatment Groups. The alternative hypothesis is that the mean change from Baseline in QMG score is smaller in the UCB7665 7mg/kg group than the placebo group.

The primary analysis of the primary variable will be based on a mixed model repeated measures (MMRM) analysis of covariance (ANCOVA) that includes terms for treatment group, the Baseline QMG score, and the interaction between treatment group and week. The model will define patient as a random effect and utilize an unstructured covariance pattern.

Least Squares (LS) Means for changes from Baseline at Visit 9 for each treatment group will be presented together with LS mean differences (UCB7665 - 7mg/kg vs placebo) and 1-sided 95% confidence interval (CI).

For subjects who prematurely withdraw for any reason before Visit 9 (Day 29), data collected during the PEOT Visit will be used to impute QMG scores at the next consecutive visit.

Different sensitivity analyses to evaluate the effect of missing observations on the primary analysis findings will be done. The first sensitivity analysis will be performed in the same way as the primary analysis for the PPS. A further analysis will utilize the Last Observation Carried Forward (LOCF) approach; missing values will be replaced by the last observed post-Baseline value of the variable and the analysis will be performed on the resulting dataset.

### Change #46

14.3.2 Other efficacy analyses, 1st to 4th paragraph

The change from Baseline in QMG score, MG-Composite score, muscle weakness severity and fatigability scale score and fatigue scale score, and MGADL score, at each assessed post-Randomization Visit (during Dosing Period 1 including Visit 9) will be analyzed similarly to the change from Baseline in QMG for the FAS as described in Section 14.3.1. However instead of LOCF, observed cases will be utilized.

QMG and MG-Composite responder rates at each assessed post-Randomization Visit (during Dosing Period 1) will be compared between the 2 Treatment Groups utilizing Fisher's exact test.

The percentage of subjects with each MGFA classification at each scheduled assessment during Treatment and Observation Periods will be calculated.

Psychometric analyses of the newly developed measures MG muscle weakness severity and fatigability and fatigue scales will be performed blinded from treatment arms. The association between PROs and clinical variables will also be explored, as well as the association between the various PROs. A psychometric analysis of the MG muscle weakness severity and Fatigue scale using Rasch analysis will be performed, but reported separately from the CSR.

14.3.2 Other efficacy analyses, 1st to 4th paragraph

The secondary variables and change from Baseline in QMG score, MG-Composite score, approach similarly to the change from Baseline in QMG for the use uescribed in Section 14.3.1.

QMG, MG-Composite, and MGADL responder rates at each assessed post-Randomization Visit (during Dosing Period 1) will be compared between the 2 Treatment Groups utilizing Fisher's exact test.

The percentage of subjects with each MGE.

Treatment and G.

Treatment and Observation Periods will be calculated.

Psychometric analyses of the newly developed measures MG muscle weakness severity and fatigability and fatigue scales will be performed blinded from treatment arms. The association between PROs and clinical variables will also be explored, as well as the association between the various PROs. A psychometric analysis of the MG muscle weakness severity and fatigability scale and fatigue scale using Rasch analysis will be performed, but reported separately from the CSR.

### Change #47

- Planned safety and other analyses
- 14.4.1 Safety analyses, 5<sup>th</sup> paragraph

Exploratory safety serum biomarkers will be summarized by treatment group and visit using descriptive statistics **Figures** of mean values over time and changes from Baseline may be presented.

### Has been changed to:

- Planned other and exploratory analyses 14.4
- 14.4.1 Safety analyses, 5<sup>th</sup> paragraph

Exploratory safety biomarkers will be summarized by treatment group and visit using descriptive statistics.

### Change #48

Pharmacodynamic analysis 2<sup>nd</sup> paragraph 14.4.2.2

The following was deleted:

Figures of mean values over time and changes from Baseline will be presented. The IgG concentrations pre- and postdepletion at each scheduled assessment will be listed and summarized by treatment group and visit.

### Planned interim analysis and data monitoring, 1st and 2nd paragraph 14.7

Two interim analyses will be performed. The first interim analysis will be conducted after 20 subjects (receiving 6 sc infusions) have attended the second visit of the observational period (ie, the visit 2 weeks after last dosing). Based on this unblinded analysis the safety of UCB7665 will be assessed by the DMC. The safety variables to be used and the decision rules to be applied will be specified in the DMC charter. The DMC can either recommend to continue the study as planned or to stop the study. In addition futility of UCB7665 will be assessed based on QMG score and MG-Composite score data. In case of futility, the study will be stopped. The decision rules for futility will be described in the DMC charter. During this review recruitment will not be stopped. The second interim analysis will be performed once all subjects have attended Visit 9. the first visit of the second Dosing Period (ie, Day 29). This interim analysis will provide the results for the primary variable 'change from Baseline to Visit 9 (Day 29) in the QMG score' and secondary variable 'change from Baseline to Visit 9 (Day 29) in MG-Composite score'. For the second interim analysis the DMC will not be utilized.

The analyses will be described in a separate Interim SAP. The first interim analysis will utilize all safety and efficacy data (as specified in the DMC charter), which will be available at the time the 20<sup>th</sup> subject attended Visit 16. For both interim analyses, the data subject to analysis should be as clean as possible; however, the database will not be locked and a snapshot will be taken.

### Has been changed to:

# Planned interim analysis and data monitoring, 1<sup>st</sup> and 2<sup>nd</sup> paragraph

At least three interim analyses will be performed. The first interim analysis for futility will be performed once approximately 20 subjects have attended Visit 9, the first visit of the second Dosing Period (ie, Day 29). Futility of UCB7665 will be assessed based on QMG score, MG-Composite score, and MGADL data. In case of futility, the study will be stopped or amended. The decision rules for futility will be described in the DMC charter. The second interim analysis will be conducted after approximately 20 subjects (receiving 6 sc infusions) have had Visit 16 (Day 57). Based on this unblinded analysis the safety of UCB7665 will be assessed by the DMC. The safety variables to be used and the potential outcomes of the analysis will be specified in the DMC charter. During this review recruitment will not be stopped. The third interim analysis will be performed once all subjects have attended Visit 9 (Day 29), the first visit of the second Dosing Period (ie, Day 29). This interim analysis will provide the results for the primary variable 'change from Baseline to Visit 9 (Day 29) in the QMG score', and secondary variables 'change from Baseline to Visit 9 (Day 29) in MG-Composite score' and 'change from Baseline to Visit 9 (Day 29) in the MGADL score'. For the third interim analysis the DMC will not be utilized.

The analyses will be described in a separate Interim SAP. The first interim analysis will utilize all efficacy data (as specified in the DMC charter), which will be available at the time the 20<sup>th</sup> subject attended Visit 9. The second interim analysis will utilize all safety data (as specified in the DMC charter), which will be available at the time the 20<sup>th</sup> subject attended Visit 16. For all interim analyses, the data subject to analysis should be as clean as possible; however, the database will not be locked and a snapshot will be taken.


### Determination of sample size, 3<sup>rd</sup> paragraph 14.8

Assuming a treatment difference of 3.4 points in the mean change from Baseline in QMG at Visit 9 between the placebo and UCB7665 treatment arm with SD equal to 3.4, a sample size of 40 subjects (20 for each treatment group) provides >90% power to detect a treatment Further it will be assumed that approximately 5% of the randomized for the FAS and, hence 42 subjects will be randomized. Assuming a treatment difference of 3.4 points in the mean change from Baseline in QMG at

JD equal to wer to detect a transmission and an analysis and an application and a subjects and analysis and a subject and an application and a subject a subject and a subject a subject a subject a subject a subject a subject as sub


### 18.13 **Protocol Amendment 2**

### Rationale for the amendment

The protocol has been amended to include an additional patient-reported outcome assessment, The printer of the pairs in jitter and state of the pairs in jitte

Administrative and stylistic changes may not be included in the summary of changes since they are considered minor.

The following shows the changes made in Amendment 2 compared to Protocol Amendment 1, dated 07 Feb 2017.

### Modifications and changes

### Global changes

The following changes were made throughout the protocol:

- Other efficacy and immunological variables were updated. Statistical analyses sections were updated accordingly.
- Additional term 'jitter' for the SFEMG performance for relevant sections. The term has been modified to be presented as 'jitter (SFEMG) measurement'.
- Instructions for subjects using pyridostigmine have been reworded to clarify the requisite for the QMG assessment. Subjects 'should not take' pyridostigmine.
- Study assessments and procedures for treatment visits only have been categorized as preduring- and postdose throughout Section 8 in line with the Schedule of Study Assessments.

### Specific changes

### Change #1

### Sponsor Study Physician

| Name: | |
|----------|---------------------------|
| Address: | UCB Biosciences, Inc. |
| SC | 8010 Arco Corporate Drive |
| | Raleigh, NC 27617 |
| | UNITED STATES |

| Phone: | |
|--------|---|
| Fax: | - |

| Name: | |
|----------|---------------------------|
| Address: | UCB Biosciences, Inc. |
| | 8010 Arco Corporate Drive |
| | Raleigh, NC 27617 |
| | UNITED STATES |
| Phone: | , Silot |
| Fax: | - exter |

### Change #2

List of Abbreviations – additional abbreviations

IPI interpotential interval

MCD mean consecutive difference

MGII Myasthenia Gravis Impairment Index

### Change #3

- 4.1.3 Other efficacy variables
- Change in mean jitter in SFEMG from Baseline to Visit 9 for the subjects consenting to this measurement at the participating sites

### Has been changed to:

- Change in the percentage of normal fiber pairs in jitter (SFEMG) studies from Baseline to Visit 9 for the subjects consenting to this measurement at the participating sites
- Change in MCD of the interpotential interval (IPI) in jitter (SFEMG) studies from Baseline to Visit 9 for the subjects consenting to this measurement at the participating sites
- A reduction in MCD of ≥9μs in jitter (SFEMG) studies will define clinical improvement

### Change #4

- 4.2.4 Immunological variables
- Charge from Baseline in serum complement levels (C3 and C4) and plasma complement levels (C3a and C5a) at each scheduled assessment during Treatment and Observation Periods
- status (negative/positive) and change from Baseline in relative mass units at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in serum BAFF levels

Change from Baseline in cytokines (in subjects experiencing infusion reactions) at assessments during Treatment and Observation Periods

### Has been changed to:

- (negative or confirmed positive) and either change confirmed positive and either change confirmed positive.

  Change from Baseline in serum BAFF levels.

  Change from Baseline in cytokines pre- and postdose (postdose in subjects experiencing infusion reactions) at assessments during Treatment and Observation Periods.
- Jose in subject Observation Period Observation Period Republication and and Republication application applicatio


Table 5.1: Schedule of assessments

| UCB<br>Clinical Study P | rotocol | | | | | | | | UCE | 37665 | 5 | | | | | | | | | | N) | ep 2017<br>4G0002 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Change #5 | | | | | | | | | | | | | | | | | | | | | tionsthe | |
| 5.2 Schedule | of stud | y assessn | nents | | | | | | | | | | | | | | | | | dis | illo | |
| Table 5.1: | Sche | edule of | ass | essm | ents | 5 | | | | | | | | | | | | | or | 70. | | |
| Assessments | Screen | ing | Trea | tment l | Period | | | | | | | | | | | Obs | servat | tion P | eriod | l <sup>a</sup> | | UV |
| | | | Dosi | ng Peri | od 1 | | | | | Dos | ing Per | riod 2 | | | | | Keil | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 150 | 16 | 17 | 18 | 19 | 20<br>FV/PEOT<br>c | |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup> (± 2 | 9 | 15 <sup>d</sup> (± 2 | 16 | 22 <sup>d</sup> (± 2 days) | 29 <sup>d</sup> (± 2 | 30 | 36 <sup>d</sup> (± 2 | 37 | <b>43<sup>d</sup></b> | 44 | 50 | 57 | 64 | 78 | 92 | 99<br>(± 2 days) | |
| | | | | | | days) | | | days) | | | | (± 2 days) | | | | ( = ==== | | | | | |
| Written informed | consent | X | | | | | | | | 5 | )× | | 56, | | | | | | | | | |
| Written informed for genomic subst | | X | | | | | | | 2010 | | 1230 | 9. | | | | | | | | | | |
| Demographic data | ı | X | | | | | | ~ | .O' | ill' | ) | | | | | | | | | | | |
| Verification of ind/exclusion criteria | | X | X | | | | | 4 | Politic | | | | | | | | | | | | | |
| Call or enter IRT register the visit | to | X | | | X | | X | 2 | dite | | | X | | X | | | | | | | X | |
| Call or enter IRT/<br>Randomization | | | X | | | | x ox | 7 | | X | | | | | | | | | | | | |
| Withdrawal criter | ia | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| General medical/<br>procedures history | <i>I</i> | X | | | ×0 | 74. | | | | | | | | | | | | | | | | |
| Prior and concom medication | itant | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant med procedures | ical | | X | S | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Vital signs <sup>f</sup> | | X S | X | | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |

Table 5.1: Schedule of assessments

| | rotocol | | | | | | | | 001 | 37665 | | | | | | | | | | B anical Study Protocol UCB7665 UCB7665 UCB7665 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5.1: | Sche | Schedule of assessments | | | | | | | | | | | | | | | HIONS | | | | | |
| Assessments | Screen | ning | Trea | reatment Period | | | | | | | | | | | | | | Observation Period <sup>a</sup> | | | | |
| | | | Dosing Period 1 | | | | | | | | Dosing Period 2 | | | | | | | o's | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | <b>10</b> <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | <b>14</b> <sup>b</sup> | 15 | 16 | P | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> | 9 | 15 <sup>d</sup> | 16 | 22 <sup>d</sup> | 29 <sup>d</sup> | 30 | 36 <sup>d</sup> | 37 | 43 <sup>d</sup> | 44 | 500 | 57 | 64 | 78 | 92 | 99 | |
| | | | | | (± 2 days) | | (± 2<br>days) | ı | (± 2 days) | (± 2<br>days) | | (± 2<br>days) | | (± 2<br>days) | 793 | | (± 2 c | days) | | | (± 2 days) | |
| Body weight, heig | ght <sup>g</sup> | X | | | | | | | | X | | | | S. | <i>D</i> . | | | | | | X | |
| Recording of AEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Full physical examination | | X | | | | | | | | C | 8 | 0 | Splin | | | | | | | | X | |
| Brief physical examination | | | X | | | | | | | $\mathcal{I}_{\mathrm{X}}$ | 1311 | 26 | | | | | | | | | | |
| Full neurological examination h | | X | | | | | | 2 | DR | Jilly | 3/11 | | | | | | | | | | X | |
| Brief neurological examination | | | X | | | | | | Ciling | X | | | | | | | | | | | | |
| Query for suicidal | ity <sup>i</sup> | X | X | | X | | X | 5 | X | X | | X | | X | | X | X | X | X | X | X | X |
| 12-lead ECG <sup>j</sup> | | X | X | | X | | X | 4 | X | X | | X | | X | | X | | | X | | X | |
| Laboratory tests (hematology, chenurinalysis) | mistry, | Х | X | | X | 11.P.P. | X | | X | X | | X | | X | | X | X | | X | | X | |
| Serology testing for Hepatitis B, and H | or HIV,<br>Iepatitis | X | | Se | ,0° | ) | | | | | | | | | | | | | | | | |
| IGRA tuberculosis | s test <sup>k</sup> | X | ~ | e | | | | | | | | | | | | | | | | | | |
| Tuberculosis Sign<br>Symptoms question | s and<br>onnaire | X | COL | | | | | | | | | | | | | | | | | | X | |

Table 5.1: Schedule of assessments

| Assessments | Screen | ning | Trea | tment P | eriod | l | | | | | | | | | | Obs | UV | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ng Perio | d 1 | | | | | Dos | ing Per | riod 2 | | | | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 15 | 18 | 19 | 20<br>FV/PEOT |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup><br>(± 2<br>days) | 9 | 15 <sup>d</sup><br>(± 2<br>days) | 16 | 22 <sup>d</sup><br>(± 2 days) | 29 <sup>d</sup><br>(± 2<br>days) | 30 | 36 <sup>d</sup><br>(± 2<br>days) | | 43 <sup>d</sup><br>(± 2<br>days) | 44 | 500 | 57<br>(± 2 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) |
| Blood sampling fo<br>of UCB7665 <sup>1</sup> | or PK | | X | | X | | Х | | X | X | 4 | X | | X | <i>D</i> . | X | | | | | |
| Blood sampling fo<br>analysis sub-study | | | X | | | | | | X | C) | RT | Ž | 8 blice | X | | | | | | | |
| Blood sampling for<br>analysis sub-study | | | X | | X | | | | X | ) | 1311 | 50 | | X | | | | | | | X |
| Serum pregnancy t | test | X | | | | | | | OR | . 20 | SUL | | | | | | | | | | |
| Urine pregnancy te | est <sup>n</sup> | | X | | X | | X | 4 | × ( | X | | X | | X | | X | X | X | X | X | X |
| Administration of | IMP | | X | | X | | X | | iilo | X | | X | | X | | | | | | | |
| | | | X | | X | | X | ζ | X | X | | X | | X | | X | X | X | X | X | X |
| Serum complemen<br>(C3,C4) and plasm<br>complement levels<br>and C5a) | na | | X | | X | .00 | X | 7 | X | X | | X | | х | | X | X | | | | х |
| Immunoglobulins<br>IgG and IgG subcl | | X | X | | X C | 7.4 | X | | X | X | | X | | X | | X | X | X | X | X | X |
| IgA, IgM, IgE | | | X | SO | | | | | X | X | | X | | X | | X | X | | | | X |
| MG-specific autoantibodies | | | X | S | X | | | | | X | | X | | | | X | | | | | X |

Table 5.1: Schedule of assessments

| Assessments | Screen | ing | Trea | ntment P | eriod | l | | | | | | | | | | Obs | serva | tion I | Period | Ig Oll | | UV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ing Perio | d 1 | | | | | Dos | ing Per | riod 2 | | | | | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | B | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup><br>(± 2 | 9 | 15 <sup>d</sup><br>(± 2 | 16 | 22 <sup>d</sup><br>(± 2 days) | 29 <sup>d</sup><br>(± 2 | 30 | 36 <sup>d</sup> (± 2 | 37 | 43 <sup>d</sup><br>(± 2 | 44 | 50 | 57 | 64 | 78 | 92 | 99<br>(± 2 days) | |
| | | | | | days) | | days) | | , | days) | | days) | | days) | 600 | | (± 2 | days) | | | | |
| Blood sampling for<br>exploratory biomark<br>analysis | | | X | | X | | X | | X | X | 7 | X | | X | <i>o</i> ` | | | X | | X | | |
| Blood sampling for<br>safety biomarker<br>analysis: may include<br>not limited to | | | X | | X | | X | P | X DACTE | XC | )<br>3112 <sup>11</sup> | X | | X | | X | X | X | X | X | X | |
| BAFF analysis | | | X | | X | | X | | X ill | X | | X | | X | | | | X | | X | | |
| Cytokines <sup>p</sup> | | | X | | X | | X | | N. T. | X | | X | | X | | X | X | X | X | X | X | X |
| Vaccination-specific antibody titers | c | X | | | | | N. O. | 7 | | | | | | | | | | | | | Х | |
| MG-composite scale | e | X | X | | X | ,00 | X | | X | X | | X | | X | | X | X | X | X | X | X | |
| QMG scale <sup>q</sup> | _ | X | X | | X | ), , | Х | | X | X | | X | | X | | X | Х | | X | | X | |
| Muscle weakness<br>severity and fatigab<br>scale | ility | | X | eused | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | |
| Fatigue scale | | | S. | | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | |
| MGADL scale | | 20 | X | | | | | | | X | | | | | | X | | X | | | X | |

### Table 5.1: Schedule of assessments

| Assessments | Screen | ing | Trea | tment F | Period | | | | | | | | | | | Obs | UV | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ng Perio | od 1 | | | | | Dos | Dosing Period 2 | | | | | | | O. | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | Pa | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> (± 2 days) | 9 | 15 <sup>d</sup><br>(± 2<br>days) | 16 | 22 <sup>d</sup> (± 2 days) | 29 <sup>d</sup><br>(± 2<br>days) | 30 | 36 <sup>d</sup><br>(± 2<br>days) | 37 | 43 <sup>d</sup><br>(± 2<br>days) | 44 | 50 | | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| MGFA classificati | on | X | X | | | | | | | X | | | | 0 | 9. | | | | | | X | |
| SFEMG measuren | nent <sup>r</sup> | | X | | | | | | | X | 7 | | ري. | 70. | | | | | | | | |
| Headache question | naire <sup>s</sup> | | X | X | X | X | X | X | X | XC | X | X | X | X | X | X | X | X | X | X | X | X |
| Stool sample asses | sment <sup>t</sup> | | X | | X | | X | | X | X | .:. | X. | | X | | X | X | X | X | X | X | X |
| Subject exit interv | iew | | | | | | | | G | | :130 | | | | | | | | | | X | |

AE=adverse event; BAFF=B-cell activating factor; BL=Baseline; BP=blood pressure; CSF=cerebrospinal fluid; CT=computed tomography; DNA=deoxyribonucleic acid; ECG=electrocardiogram; FV=Final Visit; GI=gastrointestinal; HIV=human immunodeficiency virus; IgA=immunoglobulin A; IgE=immunoglobulin E; IgG=immunoglobulin G; IGRA= interferon-gamma release assay; IgM=immunoglobulin M; IMP=investigational medicinal product; IRT=interactive response technology; LP=lumbar puncture; MG=myasthenia gravis; MGADL=myasthenia gravis-Activities of Daily Living; MGFA=Myasthenia Gravis Foundation of America; MRI=magnetic resonance imaging; PEOT=premature end of treatment; PK=pharmacokinetics; PR=pulse rate; RNA=ribonucleic acid; QMG=Quantitative Myasthenia Gravis;

SFEMG=single fiber electromyogram; TB=tuberculosis; UV=Unscheduled Visit


<sup>&</sup>lt;sup>a</sup> Subjects will return to the clinic/hospital for Visits 15, 16, 18, and 20; for Visits 17 and 19 subjects will either return to the clinic/hospital, or, if possible and agreed by both the investigator and subject, have home visits conducted by certified healthcare professionals.

b This visit is a telephone contact 24 hours post-IMP dose start.

<sup>&</sup>lt;sup>c</sup> Subjects who withdraw early will be encouraged to complete the PEOT Visit plus the FV (approximately 8 weeks after the final study drug administration).

<sup>&</sup>lt;sup>d</sup> A visit window of  $\pm 2$  days is allowed for the dosing visits. The visit window of  $\pm 2$  days is relative to the first dosing visit date. However, there should be a minimum interval of 5 days and maximum interval of 9 days as compared to the previous dose.

<sup>&</sup>lt;sup>e</sup> Includes consent for SFEMG for the subjects consenting to this measurement at the participating sites. Additional informed consent is needed for participation in the exploratory genomic substudy.

Systolic and diastolic BP, pulse rate, temperature, and respiratory rate. On dosing days, vital signs will be measured prior to IMP administration, 15 minutes after the start of the infusion, at the end of the infusion, 2 hours after the end of infusion and 4 hours after the end of the infusion. At nondosing visits, vital signs need only be taken once during the visit.

<sup>&</sup>lt;sup>g</sup> Body weight at Screening and at Visit 9 will be used for calculation of dose; height will be assessed only at Screening.

h In addition to Screening and the FV, a full neurological examination should be performed for any subject who experiences severe headache.

- Subjects must be off pyridostigmine (or any inhibitor medication) from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last any inhibitor dosing for each evaluation during the study.
- <sup>t</sup> For subjects consenting to this measurement at the participating sites; subjects should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. If pyridostigmine is taken, the time must be documented.
- <sup>u</sup> This assessment is applicable only to subjects experiencing severe headaches and will be performed daily until resolution (ie, if headache becomes moderate or mild, normal collection of AEs should apply); this assessment will be followed by a neurological assessment (including fundoscopy). Additionally, other diagnostic procedures including but not limited to CT scan, MRI and/or LP for CSF collection to be performed if indicated at the discretion of the investigator.
- <sup>v</sup> Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally.

<sup>&</sup>lt;sup>1</sup> A query for suicidal ideation will be asked by Investigator at each clinical visit (including Visit 17 or Visit 19 when it is conducted at the clinic). A full C SSRS assessment will be performed only when subject has a positive response to the suicidal ideation query. If a subject has active suicidal ideation as confirmed by the answer 'Yes' to Question 4 or Question 5 of the C SSRS assessments, the subject will be excluded or withdrawn from the study and immediately referred to a Mental Healthcare Professional

<sup>&</sup>lt;sup>j</sup> ECGs will be read by a central reader.

<sup>&</sup>lt;sup>k</sup> The IGRA test will be performed in a central laboratory. Subject should not be dosed until IGRA result is available and negative.

Pre- and postdose at Visits 2, 4, 6, 9, 11, and 13; postdose samples are to be taken 4 hours after the infusion has ended.

<sup>&</sup>lt;sup>m</sup> Blood sample to be taken prior to dosing of IMP.

<sup>&</sup>lt;sup>n</sup> Urine pregnancy test will be performed using a dipstick test; a positive urine pregnancy test must be confirmed using a serum pregnancy test.

<sup>&</sup>lt;sup>p</sup> Sampling for exploratory safety biomarkers at Baseline (Visit 2) and 4 hours post dosing (Visit 2) for all subjects. During follow up only in subjects with severe headache and/or moderate to severe GI disturbances.

<sup>&</sup>lt;sup>q</sup> Sampling at Baseline for all subjects and subsequently only in subjects with infusion reaction.

Table 18.1: Schedule of assessments

| Assessments | Screen | ning | Trea | Treatment Period Observation Period a | | | | | | | | | | | | | | | UV | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ng Perio | od 1 | | | | | Dos | ing Per | riod 2 | | | | | | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 17 | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> (± 2 days) | 9 | 15 <sup>d</sup><br>(± 2<br>days) | 16 | 22 <sup>d</sup> (± 2 days) | 29 <sup>d</sup><br>(± 2<br>days) | 30 | 36 <sup>d</sup><br>(± 2<br>days) | 37 | 43 <sup>d</sup><br>(± 2<br>days) | 81784 O | 50 | 57 (± 2 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| Written informed | consent | X | | | days) | | uuy 5) | | | days) | R7 | days) | Olics | | | | | | | | | |
| Written informed for genomic subst | | X | | | | | | | .45 | 0 | ( | 200 | R | | | | | | | | | |
| Demographic data | a | X | | | | | | | ~C) * | | :12 | | | | | | | | | | | |
| Verification of in-<br>/exclusion criteria | | X | X | | | | | 2 | Dr | Jilly | ), | | | | | | | | | | | |
| Call or enter IRT register the visit | to | X | | | X | | X | | eting | | | X | | X | | | | | | | X | |
| Call or enter IRT/<br>Randomization | / | | X | | | | | , ~ | diff | X | | | | | | | | | | | | |
| Withdrawal criter | ria | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| General medical/<br>procedures histor | | X | | | | 100 | 350 | | | | | | | | | | | | | | | |
| Prior and concommedication | nitant | X | X | X | ÝQ c | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant med procedures | lical | | X | SIZE | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Vital signs <sup>f</sup> | | X | X | | X | | X | | X | X | | X | | X | | X | X | X | X | X | X | X |
| Body weight, heigh | ght <sup>g</sup> | X OF | | | | | | | | X | | | | | | | | | | | X | |
Table 18.1: Schedule of assessments

| | rotocol | | | | | | | | | 37665 | , | | | | | | | | | | ille | ep 201′<br>4G000′ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 18.1: | Sche | edule of | ass | essm | ents | 6 | | | | | | | | | | | | | | | tions | |
| Assessments | Screen | ning | Trea | tment ] | Period | | | | | | | | | | | Observation Period <sup>a</sup> | | | | | | |
| | | | | | | | | | Dosing Period 2 | | | | | | o d | | | | | | | |
| Vi | Visit | t 1 | 2<br>BL | | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | <b>10</b> <sup>b</sup> | 11 | <b>12</b> <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | P | 18 | 19 | 20<br>FV/PEOT |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> | 9 | 15 <sup>d</sup> | 16 | 22 <sup>d</sup> | 29 <sup>d</sup> | 30 | 36 <sup>d</sup> | 37 | 43 <sup>d</sup> | 44 | 500 | 57 | 64 | 78 | 92 | 99 | |
| | | | | | (± 2 days) | | (± 2<br>days) | | (± 2 days) | (± 2<br>days) | | (± 2<br>days) | | (± 2<br>days) | 79.00 | | (± 2 | days) | | | (± 2 days) | |
| Recording of AEs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Full physical examination | | X | | | | | | | | | 5 | | Jics | | | | | | | | X | |
| Brief physical examination | | | X | | | | | | .< | X <sub>C</sub> | )` | 100 | 54 | | | | | | | | | |
| Full neurological examination h | | X | | | | | | | ACIE! | | 1230 | ) | | | | | | | | | X | |
| Brief neurological examination | | | X | | | | | 4 | , | J.X | , | | | | | | | | | | | |
| Query for suicidali | ity <sup>i</sup> | X | X | | X | | X | | X till | X | | X | | X | | X | X | X | X | X | X | X |
| 12-lead ECG <sup>j</sup> | | X | X | | X | | X | 2 | X | X | | X | | X | | X | | | X | | X | |
| Laboratory tests<br>(hematology, chen<br>urinalysis) | nistry, | X | X | | X | | X | 70 | X | X | | X | | X | | X | X | | X | | X | |
| Serology testing for Hepatitis B, and H C | | X | | | ×0 | 716.6 | | | | | | | | | | | | | | | | |
| IGRA tuberculosis | s test <sup>k</sup> | X | | SO | > | | | | | | | | | | | | | | | | | |
| Tuberculosis Signs<br>Symptoms questio | s and<br>nnaire | X | , 'C | 2 | | | | | | | | | | | | | | | | | X | |
| Blood sampling fo of UCB7665 <sup>l</sup> | r PK | call' | X | | X | | X | | X | X | | X | | X | | X | | | | | | |

Table 18.1: Schedule of assessments

| Assessments | Screen | ing | Trea | ntment I | Period | l | | | | | | | | | | Obs | UV | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ing Perio | od 1 | | | | | Dos | ing Per | riod 2 | | | | O'S | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 15 | 18 | 19 | FV/PEOT |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup> (± 2 | | 15 <sup>d</sup> (± 2 | 16 | 22 <sup>d</sup><br>(± 2 days) | 29 <sup>d</sup><br>(± 2 | 30 | 36 <sup>d</sup> (± 2 | 37 | 43 <sup>d</sup> (± 2 | 44 | 500 | 57 | 64<br>days) | 78 | 92 | 99<br>(± 2 days) |
| Blood sampling for<br>analysis sub-study | | | X | | days) | | days) | | Х | days) | | days) | | days) | 3,0 | | (+2 | (lays) | | | |
| Blood sampling for<br>analysis sub-study | r RNA<br>m | | X | | X | | | | X | () | RT | ~ | 29lice | X | | | | | | | X |
| Serum pregnancy t | est | X | | | | | | | | | .:.( | 200 | | | | | | | | | |
| Urine pregnancy te | est <sup>n</sup> | | X | | X | | X | | X | X | :1200 | X | | X | | X | X | X | X | X | X |
| Administration of | IMP | | X | | X | | Х | | OR. | X | 2. | X | | X | | | | | | | |
| | | | X | | X | | X | 4 | X | X | | X | | X | | X | X | X | X | X | X |
| Serum complemen<br>(C3,C4) and plasm<br>complement levels<br>and C5a) <sup>0</sup> | ıa | | Х | | Х | | X | 400 | diket | X | | Х | | Х | | | | | | | X |
| Immunoglobulins (<br>IgG and IgG subcl | | X | X | | X | 90. | X | | X | Х | | Х | | X | | Х | Х | Х | Х | X | X |
| IgA, IgM, IgE | | | X | | Ç. | 24 | | | X | X | | X | | X | | X | X | | | | X |
| MG-specific autoantibodies | | | X | Sec | X | | | | | X | | X | | | | X | | | | | Х |
| Blood sampling for<br>exploratory biomar<br>analysis | | _4 | X | 8 | X | | X | | Х | Х | | Х | | X | | | | Х | | Х | |
| Blood sampling for | r | Cal | Х | | X | | X | | X | Х | | X | | X | | X | Х | X | X | X | X |

Table 18.1: Schedule of assessments

| Assessments | Screen | ning | Trea | tment F | Period | l | | | | | | | | | | Ob | UV | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ng Perio | od 1 | | | | | Dos | ing Per | riod 2 | | | | | | | O. | 1 | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | 5 <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | 15 | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | 8 <sup>d</sup> (± 2 | | 15 <sup>d</sup> (± 2 | 16 | 22 <sup>d</sup><br>(± 2 days) | 29 <sup>d</sup><br>(± 2 | 30 | 36 <sup>d</sup> (± 2 | 37 | 43 <sup>d</sup><br>(± 2 | 44 | 500 | 57 | 64 | 78 | 92 | 99<br>(± 2 days) | |
| | | | | | (= 2<br>days) | | days) | | (- 2 days) | days) | | days) | | (= 2<br>days) | | | (± 2 | days) | | | | |
| safety biomarker<br>analysis: may | F | | | | | | | | | C | R <sup>7</sup> | or of | Plica | lor, | <i>S</i> * | | | | | | | |
| BAFF analysis | | | X | | X | | X | | X | X | :13 | Х | | X | | | | X | | X | | |
| Cytokines <sup>q</sup> | | | X | | | | X | _< | Ök | X | 5 | | | X | | | | | | | X | X |
| Vaccination-specifi<br>antibody titers | ic | х | | | | | | <b>*</b> | leting? | 2 | | | | | | | | | | | X | |
| MG-composite sca | le <sup>r</sup> | X | X | | X | | X | 2 | ⊗x | X | | X | | X | | X | X | X | X | X | X | |
| QMG scale <sup>s</sup> | | X | X | | X | | X | 9 | X | X | | X | | X | | X | X | | X | | X | |
| Muscle weakness<br>severity and fatigat<br>scale | bility | | X | | X | J.P.P. | X | | х | X | | X | | X | | X | Х | X | X | X | X | |
| Fatigue scale | | | X | | X | | X | | X | Х | | Х | | Х | | X | х | X | х | X | X | |
| MGADL scale | | | X | Sec | | | | | | X | | | | | | X | | X | | | X | |
| MGII | | | X | S | | | X | | | X | | | | X | | | X | | X | | X | |
| MGFA classification | on | X | , X | | | | | | | X | | | | | | | | | | | X | |
| Jitter (SFEMG) | | (31) | X | | | | | | | X | | | | | | | | | | | | |

### Table 18.1: Schedule of assessments

| Assessments | Screen | ing | Trea | atment l | Period | l | | | | | | | | | | Obs | UV | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dosi | ing Peri | od 1 | | | | | Dosing Period 2 | | | | | | | o <sup>x</sup> | | | | | |
| | Visit | 1 | 2<br>BL | 3 <sup>b</sup> | 4 | <b>5</b> <sup>b</sup> | 6 | 7 <sup>b</sup> | 8 | 9 | 10 <sup>b</sup> | 11 | 12 <sup>b</sup> | 13 | 14 <sup>b</sup> | 15 | 16 | PX | 18 | 19 | 20<br>FV/PEOT | |
| | Day | -28 to -1 | 1 | 2 | <b>8</b> <sup>d</sup> (± 2 days) | 9 | 15 <sup>d</sup><br>(± 2<br>days) | 16 | 22 <sup>d</sup> (± 2 days) | 29 <sup>d</sup><br>(± 2<br>days) | 30 | 36 <sup>d</sup><br>(± 2<br>days) | | 43 <sup>d</sup><br>(± 2<br>days) | ्रं | 500 | | 64<br>days) | 78 | 92 | 99<br>(± 2 days) | |
| measurement <sup>t</sup> | | | | | | | | | | | | | | 0 | <i>S</i> ` | | | | | | | |
| Headache question | nnaire <sup>u</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Stool sample asses | ssment | | X | | X | | X | | X | X | R | X | 26/10 | X | | X | X | X | X | X | X | X |
| Subject exit interv | iew | | | | | | | | _< | | | 10.0 | | | | | | | | | X | |

AE=adverse event; BAFF=B-cell activating factor; BL=Baseline; BP=blood pressure; CSF=cerebrospinal fluid; CT=computed tomography; DNA=deoxyribonucleic acid; ECG=electrocardiogram; FV=Final Visit; GI=gastrointestinal; HIV=human immunodeficiency virus; IgA=immunoglobulin A; IgE=immunoglobulin E; IgG=immunoglobulin G; IGRA= interferon-gamma release assay; IgM=immunoglobulin M; IMP=investigational medicinal product; IRT=interactive response technology; LP=lumbar puncture; MG=myasthenia gravis; MGADL=myasthenia gravis-Activities of Daily Living; MGFA=Myasthenia Gravis Foundation of America; MRI=magnetic resonance imaging; PEOT=premature end of treatment; PK=pharmacokinetics; PR=pulse rate; RNA=ribonucleic acid; QMG=Quantitative Myasthenia Gravis;

SFEMG=single fiber electromyogram; TB=tuberculosis; UV=Unscheduled Visit


<sup>&</sup>lt;sup>a</sup> Subjects will return to the clinic/hospital for Visits 15, 16, 18, and 20; for Visits 17 and 19 subjects will either return to the clinic/hospital, or, if possible and agreed by both the investigator and subject, have home visits conducted by certified healthcare professionals.

b This visit is a telephone contact 24 hours post-IMP dose start.

<sup>&</sup>lt;sup>c</sup> Subjects who withdraw early will be encouraged to complete the PEOT Visit plus the FV (approximately 8 weeks after the final study drug administration).

d A visit window of ±2 days is allowed for the dosing visits. The visit window of ±2 days is relative to the first dosing visit date. However, there should be a minimum interval of 5 days and maximum interval of 9 days as compared to the previous dose.

<sup>&</sup>lt;sup>e</sup> Includes consent for jitter (SFEMG) for the subjects consenting to this measurement at the participating sites. Additional informed consent is needed for participation in the exploratory genomic substudy.

f Systolic and diastolic BP, pulse rate, temperature, and respiratory rate. On dosing days, vital signs will be measured prior to IMP administration, 15 minutes after the start of the infusion, at the end of the infusion, 2 hours after the end of infusion and 4 hours after the end of the infusion. At nondosing visits, vital signs need only be taken once during the visit.

<sup>&</sup>lt;sup>g</sup> Body weight at Screening and at Visit 9 will be used for calculation of dose; height will be assessed only at Screening.

h In addition to Screening and the FV, a full neurological examination should be performed for any subject who experiences severe headache.

- A query for suicidal ideation will be asked by Investigator at each clinical visit (including Visit 17 or Visit 19 when it is conducted at the clinic). A full Columbia Suicide Severity Rating Scale (C-SSRS) assessment will be performed only when subject has a positive response to the suicidal ideation query. If a subject has active suicidal ideation as confirmed by the answer 'Yes' to Question 4 or Question 5 of the C-SSRS assessments, the subject will be excluded or withdrawn from the study and immediately referred to a Mental Healthcare Professional.
- <sup>j</sup> ECGs will be read by a central reader.
- k The IGRA test will be performed in a central laboratory. Subject should not be dosed until IGRA result is available and negative.
- Pre- and postdose at Visits 2, 4, 6, 9, 11, and 13; postdose samples are to be taken 4 hours after the infusion has ended.
- <sup>m</sup>Blood sample to be taken prior to dosing of IMP.
- <sup>n</sup> Urine pregnancy test will be performed using a dipstick test; a positive urine pregnancy test must be confirmed using a serum pregnancy test.
- <sup>o</sup> Sampling will be performed predose at Visit 2 and 4 hours postdose at Visits 2, 4, 6, 9, 11 and 13. A sample will be obtained at Visit 20.
- <sup>p</sup> Sampling for exploratory safety biomarkers at Baseline (Visit 2) and 4 hours post dosing (Visit 2) for all subjects. During follow up only in subjects with severe headache and/or moderate to severe GI disturbances.
- <sup>q</sup> Sampling will be performed pre- and 4 hours postdose at Visits 2, 6, 9 and 13. A sample will be obtained at Visit 20. Samples will be obtained at Visits 4 and 11 for subjects with an infusion reaction.
- This assessment will be performed at the clinic/hospital. If the subject has a home visit with certified health professionals at Visit 17 and Visit 19, this assessment will not be performed.
- Subjects should not take pyridostigmine (or any medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last any inhibitor dosing for each evaluation during the study.
- <sup>u</sup> This assessment is applicable only to subjects experiencing severe headaches and will be performed daily until resolution (ie, if headache becomes moderate or mild, normal collection of AEs should apply); this assessment will be followed by a neurological assessment (including fundoscopy). Additionally, other diagnostic procedures including but not limited to CT scan, MRI and/or LP for CSF collection to be performed if indicated at the discretion of the investigator.
- <sup>v</sup> Stool collection and analysis will be performed for subjects reporting moderate or severe diarrhea. The frequency of stool sampling will be as clinically indicated in the opinion of the investigator. Analysis of stool samples will be performed locally.

# Change #6

- Jessence (current or historical) evidence in his/her medical higher medical highe

- 6.2.2 Exclusion criteria related to concomitant medications/procedures
- 30. Subject had a thymectomy in the past 6 months, a history of thymoma World Health Organization grade B2 or B3, or Masaoka grade III or IV, or history of a thymoma requiring chemotherapy and/or radiotherapy.

# Has been changed to:

30. Subject had a thymectomy in the past 6 month or a thymoma at any time that required chemotherapy and/or radiotherapy.

# Change #8

6.4 Withdrawal Criteria

Changes to criterions #1 and #5.

Subjects MUST be withdrawn from IMP if any of the following events occur:

- 1. Subject develops an illness or has a change in health status that would interfere with his/her continued participation, including but not limited to:
  - Subject has a serious infective episode requiring hospitalization or iv antibiotic therapy (including but not limited to bacteremia or sepsis, bacterial meningitis, osteomyelitis or septic arthritis, bacterial pneumonia, or visceral abscess).
  - Subject experiences a severe adverse event (AE) of GI disturbance or headache which is considered related to the IMP in the opinion of the investigator.
- 5. Subject received IVIg or PLEX during the Treatment Period.

# Has been changed to:

Subjects MUST discontinue IMP if any of the following events occur:

- 1. Subject develops an illness or has a change in health status that would interfere with his/her continued participation, including but not limited to:
  - Subject has a serious infective episode requiring hospitalization or iv antibiotic therapy (including but not limited to bacteremia or sepsis, bacterial meningitis, osteomyelitis or septic arthritis, bacterial pneumonia, or visceral abscess).
  - Subject experiences a severe adverse event (AE) of GI disturbance or severe headache
    which is considered related to the IMP in the opinion of the investigator.
- 5. Subject received prohibited concomitant medications (as defined in Section 7.8.2 of this protocol) during the Treatment Period.

# Change #9

7.8.1 Permitted concomitant medications

Table 7.1 lists the concomitant medications that are permitted during the course of the study at a stable dose.

Table 7.1: Permitted concomitant treatments

| Permitted<br>Medications | Dose | Comment | iication |
|---|---|---|---|
| Oral Corticosteroids (eg, prednisolone) | - | | |
| Methotrexate | ≤30mg/week | | |
| Mycophenolate mofetil | ≤3g/day | | |
| Cyclosporin | ≤5mg/day | | |
| Azathioprine | ≤3mg/kg/day | | |
| Cholinesterase inhibitors | ≤600mg<br>Pyridostigmine/day | | |
| Tacrolimus | 3mg/day | | |

# Has been changed to:

Table 7.1 lists the concomitant medications that are permitted during the course of the study at a stable dose.

**Table 7.1:** Permitted concomitant treatments

| Permitted<br>Medications | Dose | Comment | ions |
|---|---|---|---|
| Oral Corticosteroids (eg, prednisolone) | - | | Valialle |
| Methotrexate | ≤30mg/week | | ensions of variations in |
| Mycophenolate<br>mofetil | ≤3g/day | | <u></u> Z` |
| Cyclosporin <sup>a</sup> | ≤5mg/kg/day for<br>unmodified<br>≤4mg/kg/day for modified<br>(microemulsion) | | |
| Azathioprine | ≤3mg/kg/day | | |
| Cholinesterase inhibitors | ≤600mg<br>Pyridostigmine/day<br>≤5mg/day | | |
| Tacrolimus <sup>b</sup> | ≤5mg/day | | |

<sup>&</sup>lt;sup>a</sup> Doses higher than listed are permissible if trough level is ≤300ng/L.

# Change #10

- 7.8.2 Prohibited concomitant treatments (medications and therapies)
- Medications which could interfere with the function of the NMJ (and which therefore could impair subjects with MG), such as, but not limited to, the following medications. For a more detailed list please refer to the Study Procedures Manual.

# Has been changed to:

Medications which could interfere with the function of the NMJ (and which therefore could impair subjects with MG), such as, but not limited to, the following medications. For a more detailed list please refer to the MGFA medication list (http://www.myasthenia.org/LivingwithMG/DrugstoAvoid.aspx).

<sup>&</sup>lt;sup>b</sup> If the total daily weight-based dose is >5mg, then a plasma trough level should be checked to ensure subject is not above the recommended therapeutic range.

# Change #11

### 9.3 Patient-reported outcomes

Subjects will complete 3 patient-reported outcomes (PROs) and participate in 1 subject exit

The PROs and the subject exit interview should be completed in the following order: MG muscle weakness and fatigability, Fatigue, and MGADL, followed by the subject exit interview (which will be performed only at the FV). The PROs should only be chester 1.2 dosing days, the PROs will be completed.

### Has been changed to:

Subjects will complete 4 patient-reported outcomes (PROs) and participate in 1 subject exit interview as per time points mentioned in the schedule of study assessments in Section 5.2. Study personnel other than the treating physician should administer the PROs. The PROs should be completed by the subject themselves in a quiet place.

The PROs and the subject exit interview should be completed in the following order: MG muscle weakness and fatigability, Fatigue, MGADL and MGH, followed by the subject exit interview (which will be performed only at the FV). The PROs should only be checked for completeness. On dosing days, the PROs will be completed prior to dosing.

# Change #12

Additional subsection:

### 9.3.4 Myasthenia Gravis Index Impairment

The MGII is a measure of disease severity based on the signs and symptoms of Myasthenia Gravis patients (Appendix 18.6). It was developed using a patient-centered approach and following current guidelines for outcome measure development, incorporating patient input throughout the different development phases (Barnett et al, 2014, Barnett et al, 2016). The MGII has 22 patient-reported and 6 examination items, and scores are presented as a sum of all items for a total score but also as an ocular and generalized sub-score.

The MGII has shown construct validity and reliability in an outpatient setting. It has less floor effect compared to other commonly used outcome measures, and it can effectively discriminate among patients with different degrees of severity (Barnett et al. 2016). Finally, the MGII is sensitive to detect clinical change after interventions, and most importantly it can detect patientmeaningful change. Additionally, the MGII showed more relative efficiency than the QMGS, MGC and MG-ADL to detect change in short-term interventions for Myasthenia. Estimates for the minimal important difference were developed.

# Change #13

### Single Fiber Electromyography

At participating sites, subjects consenting to SFEMG measurement should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be

performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. If pyridostigmine is taken, the time must be documented. This measurement will be performed by adequately trained and equipped investigators. Via a single isions or variations thereof. fiber needle inserted into a muscle, this investigation permits the recording of the action potentials in individual muscle fibers. This enables the measurement of fiber density and neuromuscular jitter which is a sensitive measurement of transmission across the NMJ) (Sanders, 2014). Jitter can assist in demonstrating MG-associated abnormalities. In well treated MG, the SFEMG displays a more normal profile.

Details of the SFEMG performance will be described in the SFEMG manual.

# Has been changed to:

9.5 Jitter (Single Fiber Electromyography)

At participating sites, subjects consenting to jitter (SFEMG) measurement should not take pyridostigmine from midnight before testing when medically safe to do so to standardize testing, but if not medically appropriate, then the treatment can be continued but the testing should be performed as best as possible at the same timeframe post last inhibitor dosing for each evaluation during the study. If pyridostigmine is taken, the time must be documented. This measurement will be performed by adequately trained and equipped investigators. Jitter measurements may be performed with a single-fiber EMG (SFEMG) electrode having a sideported recording surface with a 25µm diameter, or a disposable concentric needle electrode. This enables the measurement of fiber density and neuromuscular litter (SFEMG) (which is a sensitive measurement of transmission across the NMJ) (Sanders, 2014). Jitter (SFEMG) can assist in demonstrating MG-associated abnormalities. In well treated MG, the jitter (SFEMG) displays a more normal profile.

Details of the jitter (SFEMG) performance will be described in the SFEMG manual Subjects.

# Change #14

- Assessment of other immunological variables
- Plasma ADA ( status (negative/positive) and changes in relative mass units

# Has been changed to

Plasma ADA ( status (negative or confirmed positive) and changes in relative mass units for all scheduled assessments or titre for those confirmed positive

# Change #15

14.3.2 Other efficacy analyses

The secondary variables and change from Baseline in QMG score, MG-Composite score, MGADL score, muscle weakness severity and fatigability scale score and fatigue scale score, at each assessed post Randomization Visit (during Dosing Period 1 including Visit 9) will also be analyzed utilizing the MMRM approach similarly to the change from Baseline in QMG for the FAS as described in Section 14.3.1.

QMG, MG-Composite, and MGADL responder rates at each assessed post-Randomization Visit (during Dosing Period 1) will be compared between the 2 Treatment Groups utilizing Fisher's exact test.

The percentage of subjects with each MGFA classification at each scheduled assessment during

raugability and fatigue scales will be performed blinded from treatment arms. The association between PROs and clinical variables will also be explored, as well as the association between the various PROs. A psychometric analysis of the MG muscle weakness severity and fatigability scale and fatigue scale using Rasch analysis will be performed but reconstruction.

Changes in SFEMG will be summarized using descriptive statistics, by treatment group and time point, including changes from Baseline

### Has been changed to:

The secondary variables and change from Baseline in QMG score, MG-Composite score, MGADL score, MGII score, muscle weakness severity and fatigability scale score and fatigue scale score, at each assessed post Randomization Visit (during Dosing Period 1 including Visit 9) will also be analyzed utilizing the MMRM approach similarly to the change from Baseline in QMG for the FAS as described in Section 14.3.1.

QMG, MG-Composite, and MGADL responder rates at each assessed post-Randomization Visit (during Dosing Period 1) will be compared between the 2 Treatment Groups utilizing Fisher's exact test.

The percentage of subjects with each MGFA classification at each scheduled assessment during Treatment and Observation Periods will be calculated.

Psychometric analyses of the newly developed measures MG muscle weakness severity and fatigability and fatigue scales will be performed blinded from treatment arms. The association between PROs and clinical variables will also be explored, as well as the association between the various PROs. A psychometric analysis of the MG muscle weakness severity and fatigability scale and fatigue scale using Rasch analysis will be performed, but reported separately from the CSR.

Changes in MCD of the IPI, and normal fiber pairs in jitter (SFEMG) will be summarized using descriptive statistics, by treatment group and time point, including changes from Baseline. A reduction in MCD of ≥9µs in jitter (SFEMG) studies will also be summarized using descriptive statistics, by treatment group and time point, including changes from Baseline.

# Change #16

14.4.4 Immunological variables

All immunological variables including concentrations of Igs (IgA, IgE, and IgM), serum complement levels (C3 and C4) and plasma complement levels (C3a and C5a), and serum BAFF will be listed and summarized, using descriptive statistics, by Treatment Group and visit including changes from Baseline. Concentrations of cytokines will be listed and summarized if

15 Sep 2017 MG0002

there are sufficient data. Figures of mean values and changes from Baseline of immunological variables may be presented, and will be described in the SAP.

The status (negative/positive) and changes in relative mass units from Baseline will be listed and summarized by treatment group.

The antibodies will be listed and summarized by treatment group.

# Has been changed to:

All immunological variables including concentrations of Igs (IgA, IgE, and IgM), serum complement levels (C3 and C4) and plasma complement levels (C3a and C5a), and serum BAFF will be listed and summarized, using descriptive statistics, by Treatment Group and visit including changes from Baseline. Concentrations of cytokines will be listed and summarized if there are sufficient data. Figures of mean values and changes from Baseline of immunological variables may be presented, and will be described in the SAP.

The status (negative or confirmed positive) and either changes in relative mass units from Baseline for all scheduled assessments or titres for those confirmed positive will be listed and summarized by treatment group.

The antibodies will be listed and summarized by treatment group.

# Change #17

Additional in-text references:

### 17 References

Barnett C, Bril V, Kapral M, Kulkarni A, Davis AM. A conceptual framework for evaluating impairments in myasthenia gravis. PLos One. 2014;9(5).

Barnett C, Bril V, Kapral M, Kulkarni A, Davis AM Development and validation of the Myasthenia Gravis Impairment Index. Neurology. 2016; 87(9): 879–886.

### 19 DECLARATION AND SIGNATURE OF INVESTIGATOR

I confirm that I have carefully read and understood this protocol and agree to conduct this clinical study as outlined in this protocol, according to current Good Clinical Practice and local

The objectives and content of this protocol as well as the results deriving from it will be treated confidentially, and will not be made available to third parties without prior authorization by UCB.

All rights of publication of the results reside will as separate contract.

| Investigator: | and an arrangement of the second |
|---------------|----------------------------------|
| | - d :: calill |
| Printed name | Date/Signature |

# 20

SPONSOR DECLARATION Have carefully rout and col and col and market I confirm that I have carefully read and understand this protocol and agree to conduct this clinical study as outlined in this protocol and according to current Good Clinical Practice.

# $mg0002\hbox{-protocol-amend-}\#2$

# **ELECTRONIC SIGNATURES**

| E | LECTRONIC SIGNATURES | Server Approval Date | ationstheres |
|---|---|---|---|
| Signed by | Meaning of Signature | Server Approval Date<br>(dd-mon-yyyy<br>(HH:mm)) | |
| | Clinical Approval | 20-Sep-2017 10:00 GMT+02<br>20-Sep-2017 14:01 GMT+02 | |
| A PORT | Meaning of Signature Clinical Approval Clinical Approval Clinical Approval Clinical Approval | 21-Sep-2017 05:27 GMT+02 | |
| 3 document cannot be used to supt | | | |